CLINICAL TRIAL: NCT02173379
Title: A Clinical Evaluation of Absorb™ BVS, the Everolimus Eluting Bioresorbable Vascular Scaffold in the Treatment of Subjects With de Novo Native Coronary Artery Lesions
Brief Title: Absorb IV Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10-392 C
Record Dates: First submitted 2014-06-09; First posted 2014-06-25 (Estimated); Results first posted 2018-07-24 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Coronary Artery Disease; Coronary Artery Stenosis; Coronary Disease; Coronary Stenosis
Keywords: Absorb™ BVS; Angioplasty; Bioabsorbable; BVS; Coronary Artery Disease; Coronary Artery Endothelial Responsiveness; Coronary artery restenosis; Coronary artery stenosis; Coronary scaffold; Coronary Stent; Drug eluting stents; Everolimus; Myocardial ischemia; Stent thrombosis; Stents
MeSH Terms: conditions — Coronary Artery Disease; Coronary Stenosis; Coronary Disease; Coronary Restenosis; Myocardial Ischemia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Absorb BVS (Experimental): Subjects receiving Absorb Bioresorbable Vascular Scaffold (BVS) System, and the Absorb GT1™ BVS System
  Interventions: Device: Absorb BVS
- XIENCE (Active Comparator): Subjects receiving XIENCE V, XIENCE PRIME, or XIENCE Xpedition, XIENCE Alpine, XIENCE Pro (outside of the US only) and XIENCE ProX (outside of the US only)
  Interventions: Device: XIENCE

INTERVENTIONS:
Device: Absorb BVS — * Scaffold diameters: 2.5, 3.0 and 3.5 mm
  * Scaffold lengths: 8, 12, 18, and 28 mm. Both the 8 mm and 12 mm lengths will be available for the 2.5/3.0 mm diameter Absorb BVS. Only the 12 mm length will be available for the 3.5 mm diameter.
  * Once Absorb GT1™ BVS System is commercially available, it can also be used in the ABSORB IV trial. Scaffold diameters: 2.5, 3.0 and 3.5 mm of and scaffold lengths: 8, 12, 18, 23, and 28 mm.
  * The commercially approved CE marked device will be used in geographies where it is commercially available. The commercially approved CE marked 23mm Absorb BVS device will not be used in this study.
  Bioabsorbable drug eluting stent implantation for improving coronary luminal diameter in patients, including those with diabetes mellitus, with ischemic heart disease due to de novo native coronary artery lesions (length ≤ 24 mm) with a reference vessel diameter of ≥ 2.5 mm and ≤ 3.75 mm.
  Arms: Absorb BVS
Device: XIENCE — Commercially approved XIENCE Family Stent System, inclusive of XIENCE V, XIENCE PRIME, XIENCE Xpedition, XIENCE Alpine, XIENCE Pro (OUS only), and XIENCE ProX (OUS only).
  * Stent diameters: 2.5, 2.75, 3.0, 3.25, 3.5 and 4.0 mm. The 3.25 mm is only available for XIENCE Xpedition
  * Stent lengths: 8, 12, 15, 18, 23, and 28 mm
  * For geographies where these devices are commercially available, the investigational sties may use only their locally approved devices
  To improve coronary luminal diameter in patients, including those with diabetes mellitus, with ischemic heart disease due to de novo native coronary artery lesions (length ≤ 24 mm) with a reference vessel diameter of ≥ 2.5 mm and ≤ 3.75 mm.
  Arms: XIENCE

SUMMARY:
ABSORB IV is a prospective, randomized (1:1, Absorb BVS to XIENCE), single-blind, multi-center study, registering approximately 2610 subjects from approximately 140 sites in the United States and outside the United States. ABSORB IV is a continuation of ABSORB III (NCT01751906) trial which are maintained under one protocol because both trial designs are related. The data from ABSORB III and ABSORB IV will be pooled to support the ABSORB IV primary endpoint. Both the trials will evaluate the safety and effectiveness of Absorb BVS.

The ABSORB IV Randomized Controlled Trial (RCT) is designed to continue to evaluate the safety and effectiveness as well as the potential short and long-term benefits of Abbott Vascular Absorb™ Bioresorbable Vascular Scaffold (BVS) System, and the Absorb GT1™ BVS System (once commercially available), as compared to the commercially approved, control stent XIENCE.

DETAILED DESCRIPTION:
ABSORB IV:

A. Primary Objective:

* To evaluate 30-day clinical outcomes of the Absorb BVS compared to XIENCE in the treatment of subjects with ischemic heart disease caused by up to three de novo native coronary artery lesions in a maximum of two epicardial vessels, with a maximum of two lesions per epicardial vessel.
* To evaluate long-term clinical outcomes of Absorb BVS compared to XIENCE in the treatment of subjects with ischemic heart disease caused by up to three denovo native coronary artery lesions in a maximum of two epicardial vessels, with a maximum of two lesions per epicardial vessel.

B. Secondary Objectives:

* To evaluate 1-year clinical outcomes of the Absorb BVS compared to XIENCE in the treatment of subjects with ischemic heart disease caused by up to three de novo native coronary artery lesions in a maximum of two epicardial vessels, with a maximum of two lesions per epicardial vessel.
* To evaluate the incidence of angina occurring within 1 year, with treatment of Absorb BVS compared to XIENCE.

The enrollment of the 2610 subjects in ABSORB IV will start after enrollment completion of the 2000 primary analysis subjects in ABSORB III. All registered subjects will have clinical follow-up at 30, 90, 180, 270 days and 1, 2, 3, 4 and 5 years.

Note: All registered subjects in ABSORB IV will be followed up to 5 years via telephone contact/office visit if it is necessary as determined by the Sponsor.

In addition, all 2610 subjects in ABSORB IV will complete patient-reported outcome (PRO) self-administered questionnaires at baseline, 30 days,180 days, 1 year, 3 years and 5 years.

ELIGIBILITY:
General Inclusion Criteria:

1. Subject must be at least 18 years of age.
2. Subject or a legally authorized representative must provide written Informed Consent prior to any study related procedure, per site requirements.
3. Subject must have evidence of myocardial ischemia (e.g., silent ischemia, stable or unstable angina, non-ST-segment elevation MI (NSTEMI), OR recent ST-segment elevation MI (STEMI). Patients with stable coronary syndromes can be enrolled any time after symptom onset if eligibility criteria are otherwise met. Patients with acute coronary syndrome can be enrolled under the following conditions:

   1. Unstable angina or NSTEMI within 2 weeks of the index procedure.
   2. STEMI > 72 hours ≤ 2 weeks prior to the index procedure.

   Note: Subjects with Unstable angina (UA) or NSTEMI or STEMI occurring > 2 weeks of the index procedure can be included in the trial but should be categorized based on their current angina class.
4. Subjects must be suitable for PCI. Subjects with stable angina or silent ischemia and < 70% diameter stenosis must have objective signs of ischemia as determined by one of the following: abnormal stress echocardiogram, nuclear scan, electrocardiogram (ECG), positron emission tomography (PET), magnetic resonance imaging (MRI), and/or fractional flow reserve (FFR).

   (Note: subject with silent ischemia must have a prior history of typical angina, angina-equivalent symptoms, or atypical angina within the past year to be included in the trial.)
5. Subject must be an acceptable candidate for coronary artery bypass graft (CABG) surgery.
6. Female subject of childbearing potential who does not plan pregnancy for up to 1 year following the index procedure. For a female subject of childbearing potential a pregnancy test must be performed with negative results known within 7 days prior to the index procedure per site standard.
7. Female subject is not breast-feeding at the time of the screening visit and will not be breast-feeding for at least 1 year following the index procedure.
8. Subject agrees to not participate in any other investigational or invasive clinical study for a period of 5 years following the index procedure.

Angiographic Inclusion Criteria:

Treatment of up to three de novo lesions in a maximum of two epicardial vessels, with a maximum of two lesions per epicardial vessel. If only a single lesion is to be treated, it must be a target lesion. Up to one non-target lesion can be treated. Non-target lesion treatment can occur only in a non-target vessel.

If there are two target lesions within the same epicardial vessel, the two target lesions must be at least 15 mm apart per visual estimation; otherwise this is considered as a single target lesion for lesion (and stent) length determination and must be treated with a single study device.

1. Target lesion(s) must be located in a native coronary artery with a visually estimated or quantitatively assessed %DS of ≥50% and < 100%, with a thrombolysis in myocardial infarction (TIMI) flow of ≥ 1, and one of the following: stenosis ≥ 70%, an abnormal functional test (e.g., fractional flow reserve ≤0.80 AND/OR a positive stress test), or presentation with an acute coronary syndrome (unstable angina or NSTEMI within 2 weeks of index procedure, or STEMI >72 hours but ≤ 2 weeks prior to the index procedure).

1. Target lesion(s) must be located in a native coronary artery with reference vessel diameter (RVD) by visual estimation of ≥ 2.50 mm and ≤ 3.75 mm.
2. Target lesion(s) must be located in a native coronary artery with length by visual estimation of ≤ 24 mm.

Note: Subjects with Unstable angina (UA) or NSTEMI or STEMI occurring > 2 weeks of the index procedure can be included in the trial but should be categorized based on their current angina class.

Note: To exclude enrollment of excessively small vessels, if the operator believes that based on visual angiographic assessments, the distal reference vessel diameter is ≤ 2.75 mm such that the plan is to implant a 2.5 mm device (stent or scaffold) in a target lesion, it is strongly recommended that either on-line QCA or intravascular imaging (ultrasound or optical coherence tomography) is used and demonstrates that the measured distal RVD for this target lesion is ≥ 2.50 mm (by at least one of these imaging modalities). This measurement may be performed before or after pre-dilatation, but before randomization. If the distal RVD measures <2.5 mm, that lesion IS NOT ELIGIBLE for randomization. Such a lesion may be treated as a non-target lesion.

General Exclusion Criteria:

1. Any surgery requiring general anesthesia or discontinuation of aspirin and/or a P2Y12 receptor inhibitor is planned within 12 months after the procedure.
2. Subject has known hypersensitivity or contraindication to device material and its degradants (everolimus, poly (L-lactide), poly (DL-lactide), lactide, lactic acid) and cobalt, chromium, nickel, platinum, tungsten, acrylic and fluoro polymers that cannot be adequately pre-medicated. Subject has a known contrast sensitivity that cannot be adequately pre-medicated.
3. Subject has known allergic reaction, hypersensitivity or contraindication to any of the following: aspirin; or clopidogrel and prasugrel and ticagrelor; or heparin and bivalirudin, and therefore cannot be adequately treated with study medications.
4. Subject had an acute STEMI (appropriate clinical syndrome with ≥1 mm of ST-segment elevation in ≥2 contiguous leads) within 72 hours of the index procedure.
5. Subject has a cardiac arrhythmia identified at the time of screening for which at least one of the following criteria is met:

   1. Subject requires coumadin or any other agent for chronic oral anticoagulation.
   2. Subject is likely to become hemodynamically unstable due to their arrhythmia.
   3. Subject has poor survival prognosis due to their arrhythmia.
6. Subject has a left ventricular ejection fraction (LVEF) < 30% assessed by any quantitative method, including but not limited to echocardiography, MRI, multiple-gated acquisition (MUGA) scan, contrast left ventriculography, PET scan, etc. LVEF may be obtained within 6 months prior to the procedure for subjects with stable CAD. For subjects presenting with acute coronary syndrome (ACS), LVEF must be assessed within 1 week of the index procedure and after ACS presentation, which may include contrast left ventriculography during the index procedure but prior to randomization in order to confirm the subject's eligibility.
7. Subject has undergone prior PCI within the target vessel during the last 12 months. Prior PCI within the non-target vessel or any peripheral intervention is acceptable if performed anytime >30 days before the index procedure, or between a minimum of 24 hours and 30 days before the index procedure if successful and uncomplicated.
8. Subject requires future staged PCI of any lesion other than a target lesion identified at the time of index procedure; or subject requires future peripheral vascular interventions < 30 days after the index procedure.
9. Subject has received any solid organ transplants or is on a waiting list for any solid organ transplants.
10. At the time of screening, the subject has a malignancy that is not in remission.
11. Subject is receiving immunosuppressant therapy or has known immunosuppressive or severe autoimmune disease that requires chronic immunosuppressive therapy (e.g., human immunodeficiency virus, systemic lupus erythematosus, etc.). Note: corticosteroids are not included as immunosuppressant therapy.
12. Subject has previously received or is scheduled to receive radiotherapy to a coronary artery (vascular brachytherapy), or the chest/mediastinum.
13. Subject is receiving or will require chronic anticoagulation therapy (e.g., coumadin, dabigatran, apixaban, rivaroxaban, edoxaban or any other related agent for any reason).
14. Subject has a platelet count < 100,000 cells/mm3 or > 700,000 cells/mm3.
15. Subject has a documented or suspected hepatic disorder as defined as cirrhosis or Child-Pugh ≥ Class B.
16. Subject has renal insufficiency as defined as an estimated glomerular filtration rate (GFR) < 30 ml/min/1.73m2 or dialysis at the time of screening.
17. Subject is high risk of bleeding for any reason; has a history of bleeding diathesis or coagulopathy; has had a significant gastrointestinal or significant urinary bleed within the past six months.
18. Subject has had a cerebrovascular accident or transient ischemic neurological attack (TIA) within the past six months, or any prior intracranial bleed, or any permanent neurologic defect, or any known intracranial pathology (e.g. aneurysm, arteriovenous malformation, etc.).
19. Subject has extensive peripheral vascular disease that precludes safe 6 French sheath insertion. Note: femoral arterial disease does not exclude the patient if radial access may be used.
20. Subject has a life expectancy <5 years for any non-cardiac or cardiac cause.
21. Subject is in the opinion of the Investigator or designee, unable to comply with the requirements of the study protocol or is unsuitable for the study for any reason. This includes completion of Patient Reported Outcome instruments.
22. Subject is currently participating in another clinical trial that has not yet completed its primary endpoint.
23. Subject is part of a vulnerable population who, in the judgment of the investigator, is unable to give Informed Consent for reasons of incapacity, immaturity, adverse personal circumstances or lack of autonomy. This may include: Individuals with a mental disability, persons in nursing homes, children, impoverished persons, persons in emergency situations, homeless persons, nomads, refugees, and those incapable of giving informed consent. Vulnerable populations also may include members of a group with a hierarchical structure such as university students, subordinate hospital and laboratory personnel, employees of the Sponsor, members of the armed forces, and persons kept in detention.

Angiographic Exclusion Criteria:

All exclusion criteria apply to the target lesion(s) or target vessel(s).

1. Unsuccessful pre-dilatation, defined as the presence of one or more of the following (note: successful pre-dilatation of at least one target lesion is required prior to randomization):

   1. Residual %diameter stenosis (DS) after pre-dilatation is ≥ 40% (per visual estimation). Note: achieving a %DS ≤ 20% prior to randomization is strongly recommended.
   2. TIMI flow grade <3 (per visual estimation).
   3. Any angiographic complication (e.g. distal embolization, side branch closure).
   4. Any dissection NHLBI grade D-F.
   5. Any chest pain lasting > 5 minutes.
   6. Any ST-segment depression or elevation lasting > 5 minutes.
2. Lesion is located in left main or there is a ≥30% diameter stenosis in the left main (unless the left main lesion is a protected left main (i.e. a patent bypass graft to the LAD and/or LCX arteries is present), and there is no intention to treat the protected left main lesion).
3. Aorto-ostial right coronary artery (RCA) lesion (within 3 mm of the ostium).
4. Lesion located within 3 mm of the origin of the left anterior descending artery (LAD) or left circumflex artery (LCX).
5. Lesion involving a bifurcation with a:

   1. side branch ≥ 2 mm in diameter, or
   2. side branch with either an ostial or non-ostial lesion with diameter stenosis >50%, or
   3. side branch requiring dilatation
6. Anatomy proximal to or within the lesion that may impair delivery of the Absorb BVS or XIENCE stent:

   1. Extreme angulation (≥ 90°) proximal to or within the target lesion.
   2. Excessive tortuosity (≥ two 45° angles) proximal to or within the target lesion.
   3. Moderate or heavy calcification proximal to or within the target lesion. If intravascular ultrasound (IVUS) used, subject must be excluded if calcium arc in the vessel prior to the lesion or within the lesion is ≥ 180°.
7. Lesion or vessel involves a myocardial bridge.
8. Vessel has been previously treated with a stent and the target lesion is within 5 mm proximal or distal to a previously stented lesion.
9. Target lesion located within an arterial or saphenous vein graft or distal to any arterial or saphenous vein graft.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2604 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2022-04-06 (Actual); Study Completion 2022-04-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregg W Stone, MD, Study Chair — Columbia University Medical Center, New York, NY; Gregg W Stone, MD, Principal Investigator — Columbia University Medical Center, New York, NY; Stephen G Ellis, MD, Principal Investigator — Cleveland Clinic, Cleveland OH; Dean J Kereiakes, MD, Principal Investigator — The Christ Hospital, Cincinnati, OH
Locations (120):
- United States (98):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Chandler Regional Medical Center, Chandler, Arizona
  - Mercy Gilbert Medical Center, Gilbert, Arizona
  - Scottsdale Healthcare, Scottsdale, Arizona
  - Arkansas Heart Hospital, Little Rock, Arkansas
  - John Muir Health Concord, Concord, California
  - Washington Hospital, Fremont, California
  - Scripps Memorial Hospital La Jolla, La Jolla, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Univ Of California Davis Med Ctr, Sacramento, California
  - Sharp Memorial Hospital, San Diego, California
  - Stanford Hospital and Clinics, Stanford, California
  - Little Company Of Mary Hospital, Torrance, California
  - Medical Center of the Rockies, Loveland, Colorado
  - Yale-New Haven Hospital, New Haven, Connecticut
  - Morton Plant Hospital, Clearwater, Florida
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Baptist Medical Center Jacksonville, Jacksonville, Florida
  - UF Health Jacksonville, Jacksonville, Florida
  - Tallahassee Memorial Hospital, Tallahassee, Florida
  - Tampa General Hospital, Tampa, Florida
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - St. John's Hospital, Springfield, Illinois
  - Elkhart General Hospital, Elkhart, Indiana
  - Franciscan St Francis Health, Indianapolis, Indiana
  - Baptist Health Lexington, Lexington, Kentucky
  - University Of Kentucky Hospital, Lexington, Kentucky
  - Jewish Hospital, Louisville, Kentucky
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - MedStar Union Memorial Hospital, Baltimore, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - St. Joseph Mercy Hospital, Ann Arbor, Michigan
  - Harper University Hospital, Detroit, Michigan
  - St John Hospital & Medical Center, Detroit, Michigan
  - Northern Michigan Hospital, Petoskey, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - North Mississippi Medical Center, Tupelo, Mississippi
  - Boone Hospital Center/ Missouri Cardiovascular Specialists, LLP, Columbia, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - Barnes Jewish Hospital, St Louis, Missouri
  - St. Patrick Hospital, Missoula, Montana
  - Nebraska Heart Institute Heart Hosp., Lincoln, Nebraska
  - CHI Health Bergan Mercy, Omaha, Nebraska
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Cooper University Hospital, Camden, New Jersey
  - Our Lady of Lourdes Medical Center, Camden, New Jersey
  - Englewood Hospital and Medical Center, Englewood, New Jersey
  - NewYork-Presbyterian/Queens, Flushing, New York
  - NYP Weill Cornell Medical Center, New York, New York
  - Mount Sinai Medical Center, New York, New York
  - Columbia University Medical Center, New York, New York
  - Rochester General Hospital, Rochester, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - St. Joseph's Hospital Health Center, Syracuse, New York
  - Montefiore Medical Center, The Bronx, New York
  - Carolinas Medical Center-Northeast, Charlotte, North Carolina
  - Carolinas Medical Center, Charlotte, North Carolina
  - Novant Health Heart & Vascular Institute/Presbyterian Hospital, Charlotte, North Carolina
  - Carolinas Medical Center-Pineville, Charlotte, North Carolina
  - Rex Hospital, Inc., Raleigh, North Carolina
  - WakeMed, Raleigh, North Carolina
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - Aultman Hospital, Canton, Ohio
  - The Christ Hospital, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio State University Medical Center, Columbus, Ohio
  - Mercy St. Vincent Medical Center, Toledo, Ohio
  - Genesis Hospital, Zanesville, Ohio
  - Integris Baptist Medical Center, Inc., Oklahoma City, Oklahoma
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Holy Spirit Hospital, Camp Hill, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Doylestown Hospital, Doylestown, Pennsylvania
  - Pinnacle Health Hospitals, Harrisburg, Pennsylvania
  - Forbes Hospital, Monroeville, Pennsylvania
  - Penn Presbyterian Medical Center, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Upmc Presbyterian, Pittsburgh, Pennsylvania
  - St. Joseph Medical Center, Reading, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - The Miriam Hospital, Providence, Rhode Island
  - Anmed Health Medical Center, Anderson, South Carolina
  - Providence Hospital, Columbia, South Carolina
  - Wellmont Holston Valley Medical Center, Kingsport, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Northwest Texas Healthcare System, Amarillo, Texas
  - Seton Medical Center, Austin, Texas
  - Baylor Heart and Vascular Hospital, Dallas, Texas
  - Houston Methodist Hospital, Houston, Texas
  - East Texas Medical Center, Tyler, Texas
  - Carilion Roanoke Memorial Hospital, Roanoke, Virginia
  - Winchester Medical Center, Winchester, Virginia
  - Providence Reg Med Ctr Everett, Everett, Washington
  - Medstar Health Research Institute/ Medstar Washington Hospital Center, Northwest, Washington
- Australia (6):
  - Liverpool Hospital, Liverpool, New South Wales
  - The Prince Charles Hospital, Brisbane, Queensland
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - St Vincent's Hospital Melbourne, Fitzroy, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia
  - Royal Perth Hospital, Perth, Western Australia
- Canada (4):
  - St. Michael's Hospital, Toronto, Ontario
  - Montreal Heart Institute, Montreal, Quebec
  - Hopital du Sacre-Coeur de Montreal, Montreal, Quebec
  - CHUM-Hotel Dieu, Montreal, Quebec
- Germany (11):
  - Universitatsklinikum Freiburg, Freiburg im Breisgau, Baden-Wurttemberg
  - Universitätsklinikum Ulm, Ulm, Baden-Wurttemberg
  - Kliniken Oberallgau gGmbH, Immenstadt im Allgäu, Bavaria
  - Klinikum Kempten, Klinikverbund Kempten-Oberallgaeu gGmbH, Kempten (Allgäu), Bavaria
  - University Giessen, Giessen, Hesse
  - Klinikum Oldenburg, Oldenburg, Lower Saxony
  - Universitatsklinikum Bonn, Bonn, North Rhine-Westphalia
  - Elisabeth-Krankenhaus, Essen, North Rhine-Westphalia
  - Johannes Gutenberg-Universitaet, Mainz, Rhineland-Palatinate
  - Segeberger Kliniken GmbH - Herzzentrum, Bad Segeberg, Schleswig-Holstein
  - Immanuel Klinikum Bernau Herzzentrum Brandenburg, Bernau, State of Berlin
- National Heart Centre, Singapore, Pte, Ltd., Singapore, Singapore

REFERENCES:
- [Derived] Power DA, Camaj A, Kereiakes DJ, Ellis SG, Gao R, Kimura T, Ali ZA, Stockelman KA, Dressler O, Onuma Y, Serruys PW, Stone GW; ABSORB Investigators. Early and Late Outcomes With the Absorb Bioresorbable Vascular Scaffold: Final Report From the ABSORB Clinical Trial Program. JACC Cardiovasc Interv. 2025 Jan 13;18(1):1-11. doi: 10.1016/j.jcin.2024.08.050. PMID 39814482
- [Derived] Stone GW, Kereiakes DJ, Gori T, Metzger DC, Stein B, Erickson M, Torzewski J, Kabour A, Piegari G, Cavendish J, Bertolet B, Stockelman KA, West NEJ, Ben-Yehuda O, Choi JW, Marx SO, Spertus JA, Ellis SG; ABSORB IV Investigators. 5-Year Outcomes After Bioresorbable Coronary Scaffolds Implanted With Improved Technique. J Am Coll Cardiol. 2023 Jul 18;82(3):183-195. doi: 10.1016/j.jacc.2023.05.003. Epub 2023 May 17. PMID 37207924
- [Derived] Stone GW, Ellis SG, Gori T, Metzger DC, Stein B, Erickson M, Torzewski J, Williams J Jr, Lawson W, Broderick TM, Kabour A, Piegari G, Cavendish J, Bertolet B, Choi JW, Marx SO, Genereux P, Kereiakes DJ; ABSORB IV Investigators. Blinded outcomes and angina assessment of coronary bioresorbable scaffolds: 30-day and 1-year results from the ABSORB IV randomised trial. Lancet. 2018 Oct 27;392(10157):1530-1540. doi: 10.1016/S0140-6736(18)32283-9. Epub 2018 Sep 25. PMID 30266412

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 2604 subjects were randomized at 147 sites between August 15, 2014 and March 31, 2017. The last 5-year follow-up visit occurred on April 06, 2022. The database was then cleaned, and data extraction for the 5-year analysis occurred on July 29, 2022.
Pre-assignment Details: The number of All-Cause Mortality will differ from that reported in the Participant Flow module. This is due to the follow-up window 'treatment' of the data. Only deaths that occurred prior to the beginning of the 5-year visit window (Day 1797=1825-28) are counted in the Participant Flow; whereas in the AE table, participants who died within the follow-up window are counted.
Groups:
- Absorb BVS: Subjects receiving Absorb Bioresorbable Vascular Scaffold (BVS), and the Absorb GT1™ BVS System
- XIENCE: Subjects receiving XIENCE V, XIENCE PRIME, XIENCE Xpedition, XIENCE Alpine, XIENCE Pro (outside of the US only) or XIENCE ProX (outside of the US only)
Period: Overall Study
Arm/Group | Absorb BVS | XIENCE
Started | 1296 | 1308
Completed | 1099 | 1118
Not Completed | 197 | 190
Not completed — Lost to Follow-up | 89 | 81
Not completed — Withdrawal by Subject | 24 | 29
Not completed — Physician Decision | 8 | 8
Not completed — Death | 75 | 72
Not completed — Other Reason | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Absorb BVS: Subjects receiving public) Absorb Bioresorbable Vascular Scaffold (BVS), and the Absorb GT1™ BVS System
- Total: Total of all reporting groups
Arm/Group | Absorb BVS | XIENCE | Total
Number analyzed (Participants) | 1296 | 1308 | 2604
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.1 (10.1) | 62.2 (10.3) | 62.65 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 369 | 361 | 730
  Male | 927 | 947 | 1874
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 40 | 29 | 69
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 1256 | 1279 | 2535
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 8 | 12
  Asian | 30 | 36 | 66
  Native Hawaiian or Other Pacific Islander | 11 | 4 | 15
  Black or African American | 71 | 61 | 132
  White | 1135 | 1160 | 2295
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 45 | 39 | 84
Region of Enrollment [Number; unit: participants]
  Canada | 28 | 26 | 54
  United States | 1021 | 1041 | 2062
  Australia | 80 | 68 | 148
  Germany | 164 | 171 | 335
  Singapore | 3 | 2 | 5
Prior Coronary Intervention [Count of Participants; unit: Participants] — Population: The number of participants analyzed includes subjects who were available at that time of analysis
  Participants
    number analyzed (Participants) | 1294 | 1307 | 2601
    (all) | 390 | 435 | 825

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Target Lesion Failure (TLF)
Description: Target lesion failure (TLF) composite of Cardiac Death, Myocardial Infarction attributable to Target Vessel (TV-MI), or Ischemia-Driven Target Lesion Revascularization (ID-TLR))
Time Frame: 30 days
Population: ITT population.The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1288 | 1303
Participants | 64 | 48
Statistical Analysis 1: Comparison: Absorb BVS vs XIENCE; The hypothesis test is designed to show non-inferiority of Absorb BVS to XIENCE for the primary endpoint with a one-sided alpha of 0.025. The null (H0) and alternative (HA) hypotheses are: H0: TLFAbsorb - TLFXIENCE ≥ ∆TLF HA: TLFAbsorb - TLFXIENCE < ∆TLF; Test type: Non-Inferiority — One-sided p-value by using Farrington-Manning non-inferiority test statistic with non-inferiority margin of 2.9%, to be compared with a one-sided significance level of 0.025; p = 0.0244, Farrington-Manning

2. Secondary Outcome: TLF at 1-year, Non-inferiority Against the Control
Description: One-sided p-value by using Farrington-Manning non-inferiority test will be used with non-inferiority margin of 4.8%, to be compared with a one-sided significance level of 0.025.
Time Frame: 1 year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1254 | 1272
Participants | 98 | 82
Statistical Analysis 1: Comparison: Absorb BVS vs XIENCE; Test type: Non-Inferiority — One-sided p-value by using Farrington-Manning non-inferiority test statistic with non-inferiority margin of 4.8%, to be compared with a one-sided significance level of 0.025; p = 0.0006, Farrington-Manning

3. Secondary Outcome: Angina at 1-year, Non-inferiority Against the Control
Description: * Angina is defined as any angina or angina equivalent symptoms determined by the physician and/or research coordinator after interview of the patient, and as adjudicated by a clinical events committee (CEC).
  * This analysis will exclude angina or angina equivalent symptoms that occurred following the index procedure through hospital discharge or 7 days, whichever occurs first.
Time Frame: 1 year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1248 | 1265
Participants | 459 | 494

4. Secondary Outcome: Percentage of Target Lesion With Acute Success- Device Success (Lesion Level Analysis)
Description: Successful delivery and deployment of the study scaffold/stent at the intended target lesion and successful withdrawal of the delivery system with attainment of final in-scaffold/stent residual stenosis of less than 30% by quantitative coronary angiography (QCA) (by visual estimation if QCA unavailable). When bailout scaffold/stent is used, the success or failure of the bailout scaffold/stent delivery and deployment is not one of the criteria for device success.
Time Frame: In-hospital (≤ 7days)
Population: as for outcome 1
Measure: Number; unit: Percentage of target lesions
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1282 | 1303
Number analyzed (Target lesions) | 1424 | 1450
Percentage of target lesions | 94.6 | 99.0

5. Secondary Outcome: Number of Participants With Acute Success- Procedural Success (Subject Level Analysis)
Description: Achievement of final in-scaffold/stent residual stenosis of less than 30% by QCA (by visual estimation if QCA unavailable) with successful delivery and deployment of at least one study scaffold/stent at the intended target lesion and successful withdrawal of the delivery system for all target lesions without the occurrence of cardiac death, target vessel MI or repeat TLR during the hospital stay (maximum of 7 days).
Time Frame: In-hospital (≤ 7days)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1282 | 1303
Participants | 1194 | 1246

6. Secondary Outcome: Number of Death (Cardiac, Vascular, Non-cardiovascular)
Description: Cardiac death: Any death due to proximate cardiac cause (e.g. MI, low-output failure, fatal arrhythmia), unwitnessed death and death of unknown cause, all procedure related deaths including those related to concomitant treatment.
  Non-cardiovascular death: Any death not covered by the above definitions such as death caused by infection, malignancy, sepsis, pulmonary causes, accident, suicide or trauma.
Time Frame: In-hospital (≤ 7 days post index procedure)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1291 | 1304
Participants | 1 | 0

7. Secondary Outcome: Number of Death (Cardiac, Vascular, Non-cardiovascular)
Description: Cardiac death (CD): Any death due to proximate cardiac cause (e.g. MI, low-output failure, fatal arrhythmia), unwitnessed death and death of unknown cause, all procedure related deaths including those related to concomitant treatment.
  Non-cardiovascular death: Any death not covered by the above definitions such as death caused by infection, malignancy, sepsis, pulmonary causes, accident, suicide or trauma.
Time Frame: 30 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1288 | 1303
Participants | 1 | 1

8. Secondary Outcome: Number of Death (Cardiac, Vascular, Non-cardiovascular)
Description: as for outcome 7
Time Frame: 90 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1286 | 1300
Participants | 5 | 5

9. Secondary Outcome: Number of Death (Cardiac, Vascular, Non-cardiovascular)
Description: as for outcome 7
Time Frame: 180 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1282 | 1291
Participants | 7 | 8

10. Secondary Outcome: Number of Death (Cardiac, Vascular, Non-cardiovascular)
Description: as for outcome 7
Time Frame: 270 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1264 | 1279
Participants | 10 | 11

11. Secondary Outcome: Number of Death (Cardiac, Vascular, Non-cardiovascular)
Description: as for outcome 7
Time Frame: 1 year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1255 | 1273
Participants | 16 | 15

12. Secondary Outcome: Number of Death (Cardiac, Vascular, Non-cardiovascular)
Description: as for outcome 7
Time Frame: 2 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1236 | 1255
Participants | 22 | 22

13. Secondary Outcome: Number of Death (Cardiac, Vascular, Non-cardiovascular)
Description: as for outcome 7
Time Frame: 3 years
Population: ITT population. The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1219 | 1241
Participants | 39 | 32

14. Secondary Outcome: Number of Death (Cardiac, Vascular, Non-cardiovascular)
Description: as for outcome 7
Time Frame: 4 years
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1206 | 1220
Participants | 54 | 49

15. Secondary Outcome: Number of Death (Cardiac, Vascular, Non-cardiovascular)
Description: Cardiac death (CD): Any death due to proximate cardiac cause (e.g. MI, low-output failure, fatal arrhythmia), unwitnessed death and death of unknown cause, all procedure related deaths including those related to concomitant treatment. Non-cardiovascular death: Any death not covered by the above definitions such as death caused by infection, malignancy, sepsis, pulmonary causes, accident, suicide or trauma.
  For the All-Cause Mortality data, the denominator excludes participants who are lost-to-follow-up or withdrawn (by subject or physician) through a given timepoint without any DMR event (all death, MI and revascularization, respectively). If these participants were included in the denominator in each arm, that would equate to assuming that these participants are alive, potentially underestimating the death rate by inflating the denominator.
Time Frame: 5 years
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1189 | 1200
Participants | 77 | 72

16. Secondary Outcome: Number of Participants With Myocardial Infarction (MI)
Description: * Attributable to target vessel (TV-MI)
  * Not attributable to target vessel (NTV-MI)
Time Frame: In-hospital (≤ 7 days post index procedure)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1291 | 1304
Participants | 50 | 43

17. Secondary Outcome: Number of Participants With Myocardial Infarction (MI)
Description: * Attributable to target vessel (TV-MI)
  * Not attributable to target vessel (NTV-MI)
Time Frame: 30 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1288 | 1303
Participants | 58 | 47

18. Secondary Outcome: Number of Participants With Myocardial Infarction (MI)
Description: * Attributable to target vessel (TV-MI)
  * Not attributable to target vessel (NTV-MI)
Time Frame: 90 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1286 | 1300
Participants | 66 | 50

19. Secondary Outcome: Number of Participants With Myocardial Infarction (MI)
Description: * Attributable to target vessel (TV-MI)
  * Not attributable to target vessel (NTV-MI)
Time Frame: 180 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1282 | 1291
Participants | 70 | 56

20. Secondary Outcome: Number of Participants With Myocardial Infarction (MI)
Description: * Attributable to target vessel (TV-MI)
  * Not attributable to target vessel (NTV-MI)
Time Frame: 270 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1264 | 1279
Participants | 75 | 62

21. Secondary Outcome: Number of Participants With Myocardial Infarction (MI)
Description: * Attributable to target vessel (TV-MI)
  * Not attributable to target vessel (NTV-MI)
Time Frame: 1 year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1255 | 1273
Participants | 80 | 65

22. Secondary Outcome: Number of Participants With Myocardial Infarction (MI)
Description: * Attributable to target vessel (TV-MI)
  * Not attributable to target vessel (NTV-MI)
Time Frame: 2 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1236 | 1255
Participants | 104 | 86

23. Secondary Outcome: Number of Participants With Myocardial Infarction (MI)
Description: * Attributable to target vessel (TV-MI)
  * Not attributable to target vessel (NTV-MI)
Time Frame: 3 years
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1219 | 1241
Participants | 126 | 104

24. Secondary Outcome: Number of Participants With Myocardial Infarction (MI)
Description: * Attributable to target vessel (TV-MI)
  * Not attributable to target vessel (NTV-MI)
Time Frame: 4 years
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1206 | 1220
Participants | 145 | 119

25. Secondary Outcome: Number of Participants With Myocardial Infarction (MI)
Description: * Attributable to target vessel (TV-MI)
  * Not attributable to target vessel (NTV-MI)
Time Frame: 5 years
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1189 | 1200
Participants | 154 | 134

26. Secondary Outcome: Number of Participants With Target Vessel Myocardial Infarction (TV-MI)
Description: Myocardial infarction attributed to target vessel myocardial infarction (TV-MI)
Time Frame: In-hospital (≤ 7 days post index procedure)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1291 | 1304
Participants | 50 | 43

27. Secondary Outcome: Number of Participants With Target Vessel Myocardial Infarction (TV-MI)
Description: Myocardial infarction attributed to target vessel myocardial infarction (TV-MI)
Time Frame: 30 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1288 | 1303
Participants | 57 | 47

28. Secondary Outcome: Number of Participants With Target Vessel Myocardial Infarction (TV-MI)
Description: Myocardial infarction attributed to target vessel myocardial infarction (TV-MI)
Time Frame: 90 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1286 | 1300
Participants | 63 | 48

29. Secondary Outcome: Number of Participants With Target Vessel Myocardial Infarction (TV-MI)
Description: Myocardial infarction attributed to target vessel myocardial infarction (TV-MI)
Time Frame: 180 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1282 | 1291
Participants | 67 | 53

30. Secondary Outcome: Number of Participants With Target Vessel Myocardial Infarction (TV-MI)
Description: Myocardial infarction attributed to target vessel myocardial infarction (TV-MI)
Time Frame: 270 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1264 | 1279
Participants | 71 | 56

31. Secondary Outcome: Number of Participants With Target Vessel Myocardial Infarction (TV-MI)
Description: Myocardial infarction attributed to target vessel myocardial infarction (TV-MI)
Time Frame: 1 year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1255 | 1273
Participants | 75 | 58

32. Secondary Outcome: Number of Participants With Target Vessel Myocardial Infarction (TV-MI)
Description: Myocardial infarction attributed to target vessel myocardial infarction (TV-MI)
Time Frame: 2 year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1236 | 1255
Participants | 94 | 72

33. Secondary Outcome: Number of Participants With Target Vessel Myocardial Infarction (TV-MI)
Description: Myocardial infarction attributed to target vessel myocardial infarction (TV-MI)
Time Frame: 3 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1219 | 1241
Participants | 112 | 86

34. Secondary Outcome: Number of Participants With Target Vessel Myocardial Infarction (TV-MI)
Description: Myocardial infarction attributed to target vessel myocardial infarction (TV-MI)
Time Frame: 4 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1206 | 1220
Participants | 126 | 94

35. Secondary Outcome: Number of Participants With Target Vessel Myocardial Infarction (TV-MI)
Description: Myocardial infarction attributed to target vessel myocardial infarction (TV-MI)
Time Frame: 5 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1189 | 1200
Participants | 134 | 106

36. Secondary Outcome: Number of Participants With Target Lesion Revascularization (TLR)
Description: TLR is defined as any repeat percutaneous intervention of the target lesion or bypass surgery of the target vessel performed for restenosis or other complication of the target lesion. All TLR should be classified prospectively as ischemia driven or not ischemia driven by the investigator prior to repeat angiography.
Time Frame: In-hospital (≤ 7 days post index procedure)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1291 | 1304
Participants | 8 | 1

37. Secondary Outcome: Number of Participants With Target Lesion Revascularization (TLR)
Description: as for outcome 36
Time Frame: 30 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1288 | 1303
Participants | 14 | 3

38. Secondary Outcome: Number of Participants withTarget Lesion Revascularization (TLR)
Description: as for outcome 36
Time Frame: 90 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1286 | 1300
Participants | 16 | 4

39. Secondary Outcome: Number of Participants With Target Lesion Revascularization (TLR)
Description: as for outcome 36
Time Frame: 180 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1282 | 1291
Participants | 23 | 11

40. Secondary Outcome: Number of Participants With Target Lesion Revascularization (TLR)
Description: as for outcome 36
Time Frame: 270 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1264 | 1279
Participants | 33 | 15

41. Secondary Outcome: Number of Participants With Target Lesion Revascularization (TLR)
Description: as for outcome 36
Time Frame: 1 year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1255 | 1273
Participants | 38 | 24

42. Secondary Outcome: Number of Participants With Target Lesion Revascularization (TLR)
Description: as for outcome 36
Time Frame: 2 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1236 | 1255
Participants | 70 | 38

43. Secondary Outcome: Number of Participants With Target Lesion Revascularization (TLR)
Description: as for outcome 36
Time Frame: 3 years
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1219 | 1241
Participants | 90 | 50

44. Secondary Outcome: Number of Participants With Target Lesion Revascularization (TLR)
Description: as for outcome 36
Time Frame: 4 years
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1206 | 1220
Participants | 107 | 65

45. Secondary Outcome: Number of Participants With Target Lesion Revascularization (TLR)
Description: as for outcome 36
Time Frame: 5 years
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1189 | 1200
Participants | 114 | 82

46. Secondary Outcome: Number of Participants With Ischemia Driven TLR (ID-TLR)
Description: as for outcome 36
Time Frame: In-hospital (≤ 7 days post index procedure)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1291 | 1304
Participants | 8 | 1

47. Secondary Outcome: Number of Participants With Ischemia Driven TLR (ID-TLR)
Description: as for outcome 36
Time Frame: 30 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1288 | 1303
Participants | 13 | 3

48. Secondary Outcome: Number of Participants With Ischemia Driven TLR (ID-TLR)
Description: as for outcome 36
Time Frame: 90 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1286 | 1300
Participants | 15 | 4

49. Secondary Outcome: Number of Participants With Ischemia Driven TLR (ID-TLR)
Description: as for outcome 36
Time Frame: 180 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1282 | 1291
Participants | 22 | 11

50. Secondary Outcome: Number of Participants With Ischemia Driven TLR (ID-TLR)
Description: as for outcome 36
Time Frame: 270 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1264 | 1279
Participants | 32 | 15

51. Secondary Outcome: Number of Participants With Ischemia Driven TLR (ID-TLR)
Description: as for outcome 36
Time Frame: 1 year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1255 | 1273
Participants | 37 | 24

52. Secondary Outcome: Number of Participants With Ischemia Driven TLR (ID-TLR)
Description: as for outcome 36
Time Frame: 2 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1236 | 1255
Participants | 67 | 38

53. Secondary Outcome: Number of Participants With Ischemia Driven TLR (ID-TLR)
Description: as for outcome 36
Time Frame: 3 years
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1219 | 1241
Participants | 87 | 50

54. Secondary Outcome: Number of Participants With Ischemia Driven TLR (ID-TLR)
Description: as for outcome 36
Time Frame: 4 years
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1206 | 1220
Participants | 104 | 65

55. Secondary Outcome: Number of Participants With Ischemia Driven TLR (ID-TLR)
Description: as for outcome 36
Time Frame: 5 years
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1189 | 1200
Participants | 111 | 82

56. Secondary Outcome: Number of Participants With Target Vessel Revascularization (TVR)
Description: TVR is defined as any repeat percutaneous intervention or surgical bypass of any segment of the target vessel. The target vessel is defined as the entire major coronary vessel proximal and distal to the target lesion which includes upstream and downstream branches and the target lesion itself.
  * TVR includes both Ischemic driven TVR and Non-ischemic driven TVR.
  * TVR includes all TVR, excluding TLR
Time Frame: In-hospital (≤ 7 days post index procedure)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1291 | 1304
Participants | 3 | 0

57. Secondary Outcome: Number of Participants With Target Vessel Revascularization (TVR)
Description: as for outcome 56
Time Frame: 30 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1288 | 1303
Participants | 5 | 1

58. Secondary Outcome: Number of Participants With Target Vessel Revascularization (TVR)
Description: as for outcome 56
Time Frame: 90 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1286 | 1300
Participants | 10 | 6

59. Secondary Outcome: Number of Participants With Target Vessel Revascularization (TVR)
Description: TVR is defined as any repeat percutaneous intervention or surgical bypass of any segment of the target vessel. The target vessel is defined as the entire major coronary vessel proximal and distal to the target lesion which includes upstream and downstream branches and the target lesion itself. classified as: Ischemic driven TVR and Non-ischemic driven TVR.
  -TVR includes all TVR, excluding TLR
Time Frame: 180 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1282 | 1291
Participants | 14 | 14

60. Secondary Outcome: Number of Participants With Target Vessel Revascularization (TVR)
Description: as for outcome 56
Time Frame: 270 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1264 | 1279
Participants | 19 | 16

61. Secondary Outcome: Number of Participants With Target Vessel Revascularization (TVR)
Description: as for outcome 56
Time Frame: 1 year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1255 | 1273
Participants | 22 | 20

62. Secondary Outcome: Number of Participants With Target Vessel Revascularization (TVR)
Description: as for outcome 56
Time Frame: 2 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1236 | 1255
Participants | 44 | 39

63. Secondary Outcome: Number of Participants With Target Vessel Revascularization (TVR)
Description: as for outcome 56
Time Frame: 3 years
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1219 | 1241
Participants | 67 | 49

64. Secondary Outcome: Number of Participants With Target Vessel Revascularization (TVR)
Description: as for outcome 56
Time Frame: 4 years
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1206 | 1220
Participants | 82 | 66

65. Secondary Outcome: Number of Participants With Target Vessel Revascularization (TVR)
Description: as for outcome 56
Time Frame: 5 years
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1189 | 1200
Participants | 91 | 81

66. Secondary Outcome: Number of Participants With ID-TVR Excluding TLR
Description: as for outcome 56
Time Frame: In-hospital (≤ 7 days post index procedure)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1291 | 1304
Participants | 3 | 0

67. Secondary Outcome: Number of Participants With ID-TVR Excluding TLR
Description: as for outcome 56
Time Frame: 30 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1288 | 1303
Participants | 5 | 1

68. Secondary Outcome: Number of Participants With ID-TVR Excluding TLR
Description: as for outcome 56
Time Frame: 90 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1286 | 1300
Participants | 10 | 6

69. Secondary Outcome: Number of Participants With ID-TVR Excluding TLR
Description: as for outcome 56
Time Frame: 180 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1282 | 1291
Participants | 14 | 14

70. Secondary Outcome: Number of Participants With ID-TVR Excluding TLR
Description: as for outcome 56
Time Frame: 270 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1264 | 1279
Participants | 19 | 16

71. Secondary Outcome: Number of Participants With ID-TVR Excluding TLR
Description: as for outcome 56
Time Frame: 1 year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1255 | 1273
Participants | 22 | 20

72. Secondary Outcome: Number of Participants With ID-TVR Excluding TLR
Description: as for outcome 56
Time Frame: 2 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1236 | 1255
Participants | 42 | 38

73. Secondary Outcome: Number of Participants With ID-TVR Excluding TLR
Description: as for outcome 56
Time Frame: 3 years
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1219 | 1241
Participants | 65 | 48

74. Secondary Outcome: Number of Participants With ID-TVR Excluding TLR
Description: as for outcome 56
Time Frame: 4 years
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1206 | 1220
Participants | 80 | 65

75. Secondary Outcome: Number of Participants With ID-TVR Excluding TLR
Description: as for outcome 56
Time Frame: 5 years
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1189 | 1200
Participants | 89 | 80

76. Secondary Outcome: Number of Participants With All Coronary Revascularization
Description: Revascularization includes TLR, TVR excluding TLR, and non TVR.
Time Frame: In-hospital (≤ 7 days post index procedure)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1291 | 1304
Participants | 10 | 4

77. Secondary Outcome: Number of Participants With All Coronary Revascularization
Description: Revascularization includes TLR, TVR excluding TLR, and non TVR.
Time Frame: 30 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1288 | 1303
Participants | 19 | 8

78. Secondary Outcome: Number of Participants With All Coronary Revascularization
Description: Revascularization includes TLR, TVR excluding TLR, and non TVR.
Time Frame: 90 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1286 | 1300
Participants | 28 | 15

79. Secondary Outcome: Number of Participants With All Coronary Revascularization
Description: Revascularization includes TLR, TVR excluding TLR, and non TVR.
Time Frame: 180 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1282 | 1291
Participants | 41 | 30

80. Secondary Outcome: Number of Participants With All Coronary Revascularization
Description: Revascularization includes TLR, TVR excluding TLR, and non TVR.
Time Frame: 270 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1264 | 1279
Participants | 54 | 39

81. Secondary Outcome: Number of Participants With All Coronary Revascularization
Description: Revascularization includes TLR, TVR excluding TLR, and non TVR.
Time Frame: 1 year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1255 | 1273
Participants | 64 | 51

82. Secondary Outcome: Number of Participants With All Coronary Revascularization
Description: Revascularization includes TLR, TVR excluding TLR, and non TVR.
Time Frame: 2 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1236 | 1255
Participants | 117 | 89

83. Secondary Outcome: Number of Participants With All Coronary Revascularization
Description: Revascularization includes TLR, TVR excluding TLR, and non TVR.
Time Frame: 3 years
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1219 | 1241
Participants | 157 | 113

84. Secondary Outcome: Number of Participants With All Coronary Revascularization
Description: Revascularization includes TLR, TVR excluding TLR, and non TVR.
Time Frame: 4 years
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1206 | 1220
Participants | 185 | 141

85. Secondary Outcome: Number of Participants With All Coronary Revascularization
Description: Revascularization includes TLR, TVR excluding TLR, and non TVR.
Time Frame: 5 years
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1189 | 1200
Participants | 198 | 167

86. Secondary Outcome: Number of Participants Experienced All Death/All MI
Description: All deaths includes
  * Cardiac death: Any death due to proximate cardiac cause (e.g. MI, low-output failure, fatal arrhythmia), unwitnessed death and death of unknown cause, all procedure related deaths including those related to concomitant treatment.
  * Vascular death: Death due to non-coronary vascular causes such as cerebrovascular disease, pulmonary embolism, ruptured aortic aneurysm, dissecting aneurysm, or other vascular cause.
  * Non-cardiovascular death: Any death not covered by the above definitions such as death caused by infection, malignancy, sepsis, pulmonary causes, accident, suicide or trauma.
  Myocardial Infarction (MI) - Q wave MI: Development of new, pathological Q wave on the ECG.
  -Non-Q wave MI: Those MIs which are not Q-wave MI
Time Frame: In-hospital (≤ 7 days post index procedure)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1291 | 1304
Participants | 51 | 43

87. Secondary Outcome: Number of Participants Experienced All Death/All MI
Description: as for outcome 86
Time Frame: 30 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1288 | 1303
Participants | 59 | 48

88. Secondary Outcome: Number of Participants Experienced All Death/All MI
Description: as for outcome 86
Time Frame: 90 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1286 | 1300
Participants | 69 | 55

89. Secondary Outcome: Number of Participants Experienced All Death/All MI
Description: as for outcome 86
Time Frame: 180 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1282 | 1291
Participants | 74 | 64

90. Secondary Outcome: Number of Participants Experienced All Death/All MI
Description: as for outcome 86
Time Frame: 270 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1264 | 1279
Participants | 80 | 72

91. Secondary Outcome: Number of Participants Experienced All Death/All MI
Description: as for outcome 86
Time Frame: 1 year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1255 | 1273
Participants | 89 | 79

92. Secondary Outcome: Number of Participants Experienced All Death/All MI
Description: as for outcome 86
Time Frame: 2 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1236 | 1255
Participants | 116 | 106

93. Secondary Outcome: Number of Participants Experienced All Death/All MI
Description: as for outcome 86
Time Frame: 3 years
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1219 | 1241
Participants | 150 | 132

94. Secondary Outcome: Number of Participants Experienced All Death/All MI
Description: as for outcome 86
Time Frame: 4 years
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1206 | 1220
Participants | 181 | 159

95. Secondary Outcome: Number of Participants Experienced All Death/All MI
Description: as for outcome 86
Time Frame: 5 years
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1189 | 1200
Participants | 209 | 188

96. Secondary Outcome: Number of Participants Experienced Cardiac Death/All MI
Description: Cardiac death (CD): Any death due to proximate cardiac cause (e.g. MI, low-output failure, fatal arrhythmia), unwitnessed death and death of unknown cause, all procedure related deaths including those related to concomitant treatment.
Time Frame: In-hospital (≤ 7 days post index procedure)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1291 | 1304
Participants | 51 | 43

97. Secondary Outcome: Number of Participants Experienced Cardiac Death/All MI
Description: as for outcome 96
Time Frame: 30 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1288 | 1303
Participants | 59 | 47

98. Secondary Outcome: Number of Participants Experienced Cardiac Death/All MI
Description: as for outcome 96
Time Frame: 90 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1286 | 1300
Participants | 67 | 53

99. Secondary Outcome: Number of Participants Experienced Cardiac Death/All MI
Description: as for outcome 96
Time Frame: 180 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1282 | 1291
Participants | 71 | 61

100. Secondary Outcome: Number of Participants Experienced Cardiac Death/All MI
Description: as for outcome 96
Time Frame: 270 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1264 | 1279
Participants | 77 | 68

101. Secondary Outcome: Number of Participants Experienced Cardiac Death/All MI
Description: as for outcome 96
Time Frame: 1 year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1255 | 1273
Participants | 83 | 73

102. Secondary Outcome: Number of Participants Experienced Cardiac Death/All MI
Description: as for outcome 96
Time Frame: 2 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1236 | 1255
Participants | 107 | 96

103. Secondary Outcome: Number of Participants Experienced Cardiac Death/All MI
Description: as for outcome 96
Time Frame: 3 years
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1219 | 1241
Participants | 133 | 118

104. Secondary Outcome: Number of Participants Experienced Cardiac Death/All MI
Description: as for outcome 96
Time Frame: 4 years
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1206 | 1220
Participants | 157 | 137

105. Secondary Outcome: Number of Participants Experienced Cardiac Death/All MI
Description: as for outcome 96
Time Frame: 5 years
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1189 | 1200
Participants | 171 | 155

106. Secondary Outcome: Number of Participants Experienced Cardiac Death/TV-MI/ID-TLR (TLF)
Description: Target Lesion Failure is composite of Cardiac death/ Target Vessel Myocardial Infarction (TV-MI)/ Ischemic-Driven Target Lesion Revascularization (ID-TLR).
Time Frame: In-hospital (≤ 7 days post index procedure)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1291 | 1304
Participants | 57 | 44

107. Secondary Outcome: Number of Participants Experienced Cardiac Death/TV-MI/ID-TLR (TLF)
Description: as for outcome 106
Time Frame: 30 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1288 | 1303
Participants | 64 | 48

108. Secondary Outcome: Number of Participants Experienced Cardiac Death/TV-MI/ID-TLR (TLF)
Description: as for outcome 106
Time Frame: 90 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1286 | 1300
Participants | 71 | 53

109. Secondary Outcome: Number of Participants Experienced Cardiac Death/TV-MI/ID-TLR (TLF)
Description: as for outcome 106
Time Frame: 180 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1282 | 1291
Participants | 77 | 64

110. Secondary Outcome: Number of Participants Experienced Cardiac Death/TV-MI/ID-TLR (TLF)
Description: as for outcome 106
Time Frame: 270 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1264 | 1279
Participants | 90 | 71

111. Secondary Outcome: Number of Participants Experienced Cardiac Death/TV-MI/ID-TLR (TLF)
Description: as for outcome 106
Time Frame: 1 year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1255 | 1273
Participants | 98 | 83

112. Secondary Outcome: Number of Participants Experienced Cardiac Death/TV-MI/ID-TLR (TLF)
Description: as for outcome 106
Time Frame: 2 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1236 | 1255
Participants | 138 | 107

113. Secondary Outcome: Number of Participants Experienced Cardiac Death/TV-MI/ID-TLR (TLF)
Description: as for outcome 106
Time Frame: 3 years
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1219 | 1241
Participants | 171 | 134

114. Secondary Outcome: Number of Participants Experienced Cardiac Death/TV-MI/ID-TLR (TLF)
Description: as for outcome 106
Time Frame: 4 years
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1206 | 1220
Participants | 200 | 153

115. Secondary Outcome: Number of Participants Experienced Cardiac Death/TV-MI/ID-TLR (TLF)
Description: as for outcome 106
Time Frame: 5 years
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1189 | 1200
Participants | 216 | 180

116. Secondary Outcome: Number of Participants Experienced Cardiac Death/All MI/ID-TLR (Major Adverse Cardiac Events-MACE)
Description: Major adverse cardiac events (MACE) is defined as the composite of cardiac death, all myocardial infarction, and ischemic driven target lesion revascularization (ID-TLR).
Time Frame: In-hospital (≤ 7 days post index procedure)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1291 | 1304
Participants | 57 | 44

117. Secondary Outcome: Number of Participants Experienced With Cardiac Death/All MI/ID-TLR (MACE)
Description: as for outcome 116
Time Frame: 30 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1288 | 1303
Participants | 65 | 48

118. Secondary Outcome: Number of Participants Experienced Cardiac Death/All MI/ID-TLR (MACE)
Description: as for outcome 116
Time Frame: 90 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1286 | 1300
Participants | 74 | 55

119. Secondary Outcome: Number of Participants Experienced Cardiac Death/All MI/ID-TLR (MACE)
Description: as for outcome 116
Time Frame: 180 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1282 | 1291
Participants | 80 | 67

120. Secondary Outcome: Number of Participants Experienced Cardiac Death/All MI/ID-TLR (MACE)
Description: as for outcome 116
Time Frame: 270 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1264 | 1279
Participants | 93 | 77

121. Secondary Outcome: Number of Participants Experienced Cardiac Death/All MI/ID-TLR (MACE)
Description: as for outcome 116
Time Frame: 1 year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1255 | 1273
Participants | 102 | 89

122. Secondary Outcome: Number of Participants Experienced Cardiac Death/All MI/ID-TLR (MACE)
Description: as for outcome 116
Time Frame: 2 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1236 | 1255
Participants | 146 | 121

123. Secondary Outcome: Number of Participants Experienced Cardiac Death/All MI/ID-TLR (MACE)
Description: as for outcome 116
Time Frame: 3 years
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1219 | 1241
Participants | 183 | 152

124. Secondary Outcome: Number of Participants Experienced Cardiac Death/All MI/ID-TLR (MACE)
Description: as for outcome 116
Time Frame: 4 years
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1206 | 1220
Participants | 217 | 178

125. Secondary Outcome: Number of Participants Experienced Cardiac Death/All MI/ID-TLR (MACE)
Description: as for outcome 116
Time Frame: 5 years
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1189 | 1200
Participants | 233 | 207

126. Secondary Outcome: Number of Participants Experienced Cardiac Death/All MI/ID-TLR/ID-TVR, Non TL (Target Vessel Failure, TVF)
Description: Target Vessel Failure (TVF) is the composite of Cardiac Death, Myocardial infarction (MI) or Ischemic-Driven Target Vessel Revascularization (ID-TVR).
Time Frame: In-hospital (≤ 7 days post index procedure)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1291 | 1304
Participants | 57 | 44

127. Secondary Outcome: Number of Participants Experienced Cardiac Death/All MI/ID-TLR/ID-TVR, Non TL (TVF)
Description: as for outcome 126
Time Frame: 30 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1288 | 1303
Participants | 66 | 48

128. Secondary Outcome: Number of Participants Experienced Cardiac Death/All MI/ID-TLR/ID-TVR, Non TL (TVF)
Description: as for outcome 126
Time Frame: 90 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1286 | 1300
Participants | 77 | 59

129. Secondary Outcome: Number of Participants Experienced Cardiac Death/All MI/ID-TLR/ID-TVR, Non TL (TVF)
Description: as for outcome 126
Time Frame: 180 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1282 | 1291
Participants | 86 | 75

130. Secondary Outcome: Number of Participants Experienced Cardiac Death/All MI/ID-TLR/ID-TVR, Non TL (TVF)
Description: as for outcome 126
Time Frame: 270 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1264 | 1279
Participants | 101 | 86

131. Secondary Outcome: Number of Participants Experienced Cardiac Death/All MI/ID-TLR/ID-TVR, Non TL (TVF)
Description: as for outcome 126
Time Frame: 1 year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1255 | 1273
Participants | 111 | 101

132. Secondary Outcome: Number of Participants Experienced Cardiac Death/All MI/ID-TLR/ID-TVR, Non TL (TVF)
Description: as for outcome 126
Time Frame: 2 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1236 | 1255
Participants | 163 | 139

133. Secondary Outcome: Number of Participants Experienced Cardiac Death/All MI/ID-TLR/ID-TVR, Non TL (TVF)
Description: as for outcome 126
Time Frame: 3 years
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1219 | 1241
Participants | 211 | 171

134. Secondary Outcome: Number of Participants Experienced Cardiac Death/All MI/ID-TLR/ID-TVR, Non TL (TVF)
Description: as for outcome 126
Time Frame: 4 years
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1206 | 1220
Participants | 246 | 203

135. Secondary Outcome: Number of Participants Experienced Cardiac Death/All MI/ID-TLR/ID-TVR, Non TL (TVF)
Description: as for outcome 126
Time Frame: 5 years
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1189 | 1200
Participants | 262 | 240

136. Secondary Outcome: Number of Participants Experienced Death/All MI/All Revascularization (DMR)
Description: DMR is the composite of All Death, All Myocardial infarction (MI) and All Revascularization.
Time Frame: In-hospital (≤ 7 days post index procedure)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1291 | 1304
Participants | 57 | 46

137. Secondary Outcome: Number of Participants Experienced Death/All MI/All Revascularization (DMR)
Description: DMR is the composite of All Death, All Myocardial infarction (MI) and All Revascularization.
Time Frame: 30 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1288 | 1303
Participants | 67 | 53

138. Secondary Outcome: Number of Participants Experienced Death/All MI/All Revascularization (DMR)
Description: DMR is the composite of All Death, All Myocardial infarction (MI) and All Revascularization.
Time Frame: 90 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1286 | 1300
Participants | 81 | 65

139. Secondary Outcome: Number of Participants Experienced Death/All MI/All Revascularization (DMR)
Description: DMR is the composite of All Death, All Myocardial infarction (MI) and All Revascularization.
Time Frame: 180 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1282 | 1291
Participants | 94 | 82

140. Secondary Outcome: Number of Participants Experienced Death/All MI/All Revascularization (DMR)
Description: DMR is the composite of All Death, All Myocardial infarction (MI) and All Revascularization.
Time Frame: 270 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1264 | 1279
Participants | 110 | 97

141. Secondary Outcome: Number of Participants Experienced Death/All MI/All Revascularization (DMR)
Description: DMR is the composite of All Death, All Myocardial infarction (MI) and All Revascularization.
Time Frame: 1 year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1255 | 1273
Participants | 125 | 114

142. Secondary Outcome: Number of Participants Experienced Death/All MI/All Revascularization (DMR)
Description: DMR is the composite of All Death, All Myocardial infarction (MI) and All Revascularization.
Time Frame: 2 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1236 | 1255
Participants | 185 | 161

143. Secondary Outcome: Number of Participants Experienced Death/All MI/All Revascularization (DMR)
Description: DMR is the composite of All Death, All Myocardial infarction (MI) and All Revascularization.
Time Frame: 3 years
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1219 | 1241
Participants | 241 | 198

144. Secondary Outcome: Number of Participants Experienced Death/All MI/All Revascularization (DMR)
Description: DMR is the composite of All Death, All Myocardial infarction (MI) and All Revascularization.
Time Frame: 4 years
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1206 | 1220
Participants | 281 | 239

145. Secondary Outcome: Number of Participants Experienced Death/All MI/All Revascularization (DMR)
Description: DMR is the composite of All Death, All Myocardial infarction (MI) and All Revascularization.
Time Frame: 5 years
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1189 | 1200
Participants | 310 | 284

146. Secondary Outcome: Number of Participants With Acute Scaffold/Stent Thrombosis (Per Academic Research Consortium (ARC) Definition)
Description: Stent thrombosis was defined by Academic Research Consortium (ARC) criteria as definite (angiographic confirmation with at least one of the following: acute onset of ischemic symptoms at rest, new ischemic ECG changes that suggest acute ischemia or typical rise and fall of cardiac biomarkers OR pathological confirmation at autopsy or via examination of tissue retrieved following thrombectomy), probable (any unexplained death within the first 30 days or, regardless of the time after the index procedure, any Myocardial infarction (MI) related to documented acute ischemia in the territory of the implanted stent without angiographic confirmation and in the absence of any other obvious cause), and possible (any unexplained death from 30 days after intracoronary stenting until end of trial follow-up). Stent thrombosis was categorized as acute (0-24 hours post stent implantation), Subacute (>24 hours to 30 days post stent implantation), late (>30 days to 1 year post stent implantation).
Time Frame: 0 - 24 hours post stent implantation
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1291 | 1305
Participants
  Definite | 3 | 0
  Definite/Probable | 4 | 0
  Probable | 1 | 0

147. Secondary Outcome: Number of Participants With Subacute Scaffold/Stent Thrombosis (Per ARC Definition)
Description: as for outcome 146
Time Frame: >24 hours - 30 days post stent implantation
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1287 | 1301
Participants
  Definite | 4 | 2
  Definite/Probable | 4 | 2
  Probable | 0 | 0

148. Secondary Outcome: Number of Participants With Late Scaffold/Stent Thrombosis (Per ARC Definition)
Description: as for outcome 146
Time Frame: 30 days - 1 year post stent implantation
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1239 | 1259
Participants
  Definite | 1 | 2
  Definite/Probable | 1 | 2
  Probable | 0 | 0

149. Secondary Outcome: Number of Participants With Cumulative Scaffold/Stent Thrombosis (Per ARC Definition)
Description: Stent thrombosis was defined by Academic Research Consortium (ARC) criteria as definite (angiographic confirmation with at least one of the following: acute onset of ischemic symptoms at rest, new ischemic ECG changes that suggest acute ischemia or typical rise and fall of cardiac biomarkers OR pathological confirmation at autopsy or via examination of tissue retrieved following thrombectomy), probable (any unexplained death within the first 30 days or, regardless of the time after the index procedure, any Myocardial infarction (MI) related to documented acute ischemia in the territory of the implanted stent without angiographic confirmation and in the absence of any other obvious cause), and possible (any unexplained
Time Frame: 0 to 730 Days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1214 | 1232
Participants
  Definite | 11 | 6
  Definite/Probable | 12 | 6
  Probable | 1 | 0

150. Secondary Outcome: Number of Participants With Rehospitalization
Description: * Coronary artery disease (CAD) related
  * Cardiovascular, non-CAD related
  * Non-cardiovascular related
Time Frame: 30 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1288 | 1302
Participants | 66 | 59

151. Secondary Outcome: Number of Participants With Rehospitalization
Description: * CAD related
  * Cardiovascular, non-CAD related
  * Non-cardiovascular related
Time Frame: 90 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1285 | 1298
Participants | 111 | 122

152. Secondary Outcome: Number of Participants With Rehospitalization
Description: * CAD related
  * Cardiovascular, non-CAD related
  * Non-cardiovascular related
Time Frame: 180 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1282 | 1291
Participants | 178 | 178

153. Secondary Outcome: Number of Participants With Rehospitalization
Description: * CAD related
  * Cardiovascular, non-CAD related
  * Non-cardiovascular related
Time Frame: 270 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1265 | 1278
Participants | 227 | 237

154. Secondary Outcome: Number of Participants With Rehospitalization
Description: * CAD related
  * Cardiovascular, non-CAD related
  * Non-cardiovascular related
Time Frame: 1 year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1254 | 1271
Participants | 277 | 289

155. Secondary Outcome: Number of Participants With Rehospitalization
Description: * CAD related
  * Cardiovascular, non-CAD related
  * Non-cardiovascular related
Time Frame: 2 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1238 | 1254
Participants | 443 | 446

156. Secondary Outcome: Number of Participants With Rehospitalization
Description: * CAD related
  * Cardiovascular, non-CAD related
  * Non-cardiovascular related
Time Frame: 3 years
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1226 | 1242
Participants | 544 | 525

157. Secondary Outcome: Number of Participants With Rehospitalization
Description: * CAD related
  * Cardiovascular, non-CAD related
  * Non-cardiovascular related
Time Frame: 4 years
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1215 | 1226
Participants | 612 | 578

158. Secondary Outcome: Number of Participants With Rehospitalization
Description: * CAD related
  * Cardiovascular, non-CAD related
  * Non-cardiovascular related
Time Frame: 5 years
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1205 | 1210
Participants | 654 | 621

159. Secondary Outcome: Number of Participants With Repeat Coronary Arteriography
Time Frame: In-hospital (≤ 7 days post index procedure)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1290 | 1304
Participants | 4 | 7

160. Secondary Outcome: Number of Participants With Repeat Coronary Arteriography
Time Frame: 30 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1288 | 1301
Participants | 18 | 21

161. Secondary Outcome: Number of Participants With Repeat Coronary Arteriography
Time Frame: 90 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1282 | 1295
Participants | 33 | 40

162. Secondary Outcome: Number of Participants With Repeat Coronary Arteriography
Time Frame: 180 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1278 | 1284
Participants | 57 | 64

163. Secondary Outcome: Number of Participants With Repeat Coronary Arteriography
Time Frame: 270 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1259 | 1270
Participants | 71 | 87

164. Secondary Outcome: Number of Participants With Repeat Coronary Arteriography
Time Frame: 1 year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1242 | 1260
Participants | 84 | 103

165. Secondary Outcome: Number of Participants With Repeat Coronary Arteriography
Time Frame: 2 years
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1218 | 1237
Participants | 140 | 161

166. Secondary Outcome: Number of Participants With Repeat Coronary Arteriography
Time Frame: 3 years
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1186 | 1212
Participants | 186 | 188

167. Secondary Outcome: Number of Participants With Repeat Coronary Arteriography
Time Frame: 4 years
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1157 | 1178
Participants | 209 | 220

168. Secondary Outcome: Number of Participants With Repeat Coronary Arteriography
Time Frame: 5 years
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1125 | 1144
Participants | 225 | 237

169. Secondary Outcome: Number of Participants With Target Lesion Failure (TLF)
Description: The analysis will be based on 4610 subjects (2000 primary analysis subjects of ABSORB III and 2610 subjects of ABSORB IV)
Time Frame: 1 year
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Groups:
- Absorb BVS: Subjects receiving Absorb Bioresorbable Vascular Scaffold (BVS) System, and the Absorb GT1™ BVS System
  Absorb BVS: -Scaffold diameters: 2.5, 3.0 and 3.5 mm
  * Scaffold lengths: 8, 12, 18, and 28 mm. Both the 8 mm and 12 mm lengths will be available for the 2.5/3.0 mm diameter Absorb BVS. Only the 12 mm length will be available for the 3.5 mm diameter.
  * Once Absorb GT1™ BVS System is commercially available, it can also be used in the ABSORB IV trial. Scaffold diameters: 2.5, 3.0 and 3.5 mm of and scaffold lengths: 8, 12, 18, 23, and 28 mm.
  * The commercially approved CE marked device will be used in geographies where it is commercially available. The commercially approved CE marked 23mm Absorb BVS device will not be used in this study.
  Bioabsorbable drug eluting stent implantation for improving coronary luminal diameter in patients, including those with diabetes mellitus, with ischemic heart disease due to de novo native coronary artery lesions (length ≤ 24 mm) with a reference vessel diameter of ≥ 2.5 mm and ≤ 3.75 mm.
- XIENCE: Subjects receiving XIENCE V, XIENCE PRIME, or XIENCE Xpedition, XIENCE Alpine, XIENCE Pro (outside of the US only) and XIENCE ProX (outside of the US only)
  XIENCE: Commercially approved XIENCE Family Stent System, inclusive of XIENCE V, XIENCE PRIME, XIENCE Xpedition, XIENCE Alpine, XIENCE Pro (OUS only), and XIENCE ProX (OUS only).
  * Stent diameters: 2.5, 2.75, 3.0, 3.25, 3.5 and 4.0 mm. The 3.25 mm is only available for XIENCE Xpedition
  * Stent lengths: 8, 12, 15, 18, 23, and 28 mm
  * For geographies where these devices are commercially available, the investigational sties may use only their locally approved devices
  To improve coronary luminal diameter in patients, including those with diabetes mellitus, with ischemic heart disease due to de novo native coronary artery lesions (length ≤ 24 mm) with a reference vessel diameter of ≥ 2.5 mm and ≤ 3.75 mm.
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1255 | 1273
Participants | 98 | 83

ADVERSE EVENTS:
Time Frame: 5 years
Groups:
- Absorb BVS: Subjects receiving Absorb Bioresorbable Vascular Scaffold (BVS)
- XIENCE: Subjects receiving XIENCE V, XIENCE PRIME, or XIENCE Xpedition
Arm/Group | Absorb BVS | XIENCE
All-Cause Mortality (participants affected / at risk) | 77/1296 | 72/1308
Serious Adverse Events (participants affected / at risk) | 827/1296 | 774/1308
Other Adverse Events (participants affected / at risk) | 1012/1296 | 1034/1308
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Absorb BVS (N=1296) | XIENCE (N=1308)
ANAEMIA (Blood and lymphatic system disorders) | 11 | 17
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 0 | 1
HAEMORRHAGIC ANAEMIA (Blood and lymphatic system disorders) | 3 | 2
IRON DEFICIENCY ANAEMIA (Blood and lymphatic system disorders) | 4 | 4
NORMOCHROMIC NORMOCYTIC ANAEMIA (Blood and lymphatic system disorders) | 2 | 0
PANCYTOPENIA (Blood and lymphatic system disorders) | 0 | 1
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1 | 0
ACUTE CORONARY SYNDROME (Cardiac disorders) | 10 | 7
ACUTE LEFT VENTRICULAR FAILURE (Cardiac disorders) | 1 | 1
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 23 | 26
ANGINA PECTORIS (Cardiac disorders) | 135 | 113
ANGINA UNSTABLE (Cardiac disorders) | 53 | 57
AORTIC VALVE INCOMPETENCE (Cardiac disorders) | 1 | 0
AORTIC VALVE STENOSIS (Cardiac disorders) | 2 | 3
ARRHYTHMIA (Cardiac disorders) | 1 | 2
ARTERIOSCLEROSIS CORONARY ARTERY (Cardiac disorders) | 4 | 2
ARTERIOSPASM CORONARY (Cardiac disorders) | 0 | 1
ATRIAL FIBRILLATION (Cardiac disorders) | 45 | 32
ATRIAL FLUTTER (Cardiac disorders) | 3 | 2
ATRIAL TACHYCARDIA (Cardiac disorders) | 1 | 0
ATRIAL THROMBOSIS (Cardiac disorders) | 0 | 1
ATRIOVENTRICULAR BLOCK (Cardiac disorders) | 0 | 1
ATRIOVENTRICULAR BLOCK COMPLETE (Cardiac disorders) | 2 | 3
ATRIOVENTRICULAR BLOCK SECOND DEGREE (Cardiac disorders) | 1 | 0
BRADYCARDIA (Cardiac disorders) | 4 | 4
BUNDLE BRANCH BLOCK LEFT (Cardiac disorders) | 0 | 1
CARDIAC ARREST (Cardiac disorders) | 10 | 4
CARDIAC FAILURE (Cardiac disorders) | 13 | 3
CARDIAC FAILURE ACUTE (Cardiac disorders) | 4 | 5
CARDIAC FAILURE CHRONIC (Cardiac disorders) | 4 | 2
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 24 | 23
CARDIAC PERFORATION (Cardiac disorders) | 1 | 0
CARDIAC TAMPONADE (Cardiac disorders) | 1 | 0
CARDIAC VALVE DISEASE (Cardiac disorders) | 0 | 1
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 0 | 2
CARDIOGENIC SHOCK (Cardiac disorders) | 5 | 0
CARDIOMYOPATHY (Cardiac disorders) | 3 | 1
CARDIOPULMONARY FAILURE (Cardiac disorders) | 0 | 1
CHRONOTROPIC INCOMPETENCE (Cardiac disorders) | 1 | 1
CONGESTIVE CARDIOMYOPATHY (Cardiac disorders) | 0 | 1
COR PULMONALE (Cardiac disorders) | 1 | 0
CORONARY ARTERY DISEASE (Cardiac disorders) | 45 | 39
CORONARY ARTERY DISSECTION (Cardiac disorders) | 41 | 17
CORONARY ARTERY EMBOLISM (Cardiac disorders) | 1 | 0
CORONARY ARTERY OCCLUSION (Cardiac disorders) | 3 | 4
CORONARY ARTERY PERFORATION (Cardiac disorders) | 1 | 1
CORONARY ARTERY STENOSIS (Cardiac disorders) | 14 | 15
HYPERTENSIVE HEART DISEASE (Cardiac disorders) | 0 | 1
HYPERTROPHIC CARDIOMYOPATHY (Cardiac disorders) | 1 | 0
IN-STENT CORONARY ARTERY RESTENOSIS (Cardiac disorders) | 1 | 0
INTRACARDIAC THROMBUS (Cardiac disorders) | 1 | 0
INTRAPERICARDIAL THROMBOSIS (Cardiac disorders) | 1 | 0
ISCHAEMIC CARDIOMYOPATHY (Cardiac disorders) | 3 | 5
MITRAL VALVE INCOMPETENCE (Cardiac disorders) | 3 | 2
MITRAL VALVE PROLAPSE (Cardiac disorders) | 1 | 0
MITRAL VALVE STENOSIS (Cardiac disorders) | 1 | 0
MYOCARDIAL INFARCTION (Cardiac disorders) | 67 | 54
MYOCARDIAL ISCHAEMIA (Cardiac disorders) | 5 | 5
MYOCARDITIS (Cardiac disorders) | 0 | 1
MYOPERICARDITIS (Cardiac disorders) | 0 | 1
PALPITATIONS (Cardiac disorders) | 1 | 2
PERICARDIAL EFFUSION (Cardiac disorders) | 2 | 0
PERICARDIAL HAEMORRHAGE (Cardiac disorders) | 0 | 1
PERICARDITIS (Cardiac disorders) | 2 | 2
PRINZMETAL ANGINA (Cardiac disorders) | 2 | 1
PULSELESS ELECTRICAL ACTIVITY (Cardiac disorders) | 0 | 1
SICK SINUS SYNDROME (Cardiac disorders) | 5 | 4
STRESS CARDIOMYOPATHY (Cardiac disorders) | 2 | 0
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 3 | 5
TACHYCARDIA (Cardiac disorders) | 2 | 1
TRICUSPID VALVE INCOMPETENCE (Cardiac disorders) | 1 | 0
VENTRICULAR EXTRASYSTOLES (Cardiac disorders) | 1 | 0
VENTRICULAR FIBRILLATION (Cardiac disorders) | 5 | 0
VENTRICULAR TACHYCARDIA (Cardiac disorders) | 3 | 6
ARTERIOVENOUS MALFORMATION (Congenital, familial and genetic disorders) | 1 | 0
ATRIAL SEPTAL DEFECT (Congenital, familial and genetic disorders) | 1 | 0
CORNEAL DYSTROPHY (Congenital, familial and genetic disorders) | 1 | 0
GASTROINTESTINAL ARTERIOVENOUS MALFORMATION (Congenital, familial and genetic disorders) | 0 | 1
HYDROCELE (Congenital, familial and genetic disorders) | 1 | 0
PERONEAL MUSCULAR ATROPHY (Congenital, familial and genetic disorders) | 0 | 1
PHIMOSIS (Congenital, familial and genetic disorders) | 0 | 2
URACHAL ABNORMALITY (Congenital, familial and genetic disorders) | 0 | 1
VERTIGO (Ear and labyrinth disorders) | 2 | 4
VERTIGO POSITIONAL (Ear and labyrinth disorders) | 0 | 2
ADRENAL INSUFFICIENCY (Endocrine disorders) | 1 | 0
CARCINOID SYNDROME (Endocrine disorders) | 0 | 1
GOITRE (Endocrine disorders) | 0 | 1
HYPERPARATHYROIDISM (Endocrine disorders) | 0 | 1
HYPOTHYROIDIC GOITRE (Endocrine disorders) | 0 | 1
THYROID MASS (Endocrine disorders) | 0 | 1
AMAUROSIS FUGAX (Eye disorders) | 0 | 2
CATARACT (Eye disorders) | 4 | 5
DIPLOPIA (Eye disorders) | 1 | 1
GLAUCOMA (Eye disorders) | 1 | 0
MACULAR FIBROSIS (Eye disorders) | 0 | 1
RETINAL ARTERY EMBOLISM (Eye disorders) | 0 | 1
RETINAL DETACHMENT (Eye disorders) | 0 | 1
RETINAL DISORDER (Eye disorders) | 0 | 1
TOLOSA-HUNT SYNDROME (Eye disorders) | 0 | 1
VITREOUS HAEMORRHAGE (Eye disorders) | 0 | 2
ABDOMINAL HERNIA (Gastrointestinal disorders) | 1 | 0
ABDOMINAL MASS (Gastrointestinal disorders) | 1 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 7 | 5
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 0 | 1
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1 | 1
ANAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1
ASCITES (Gastrointestinal disorders) | 1 | 1
BARRETT'S OESOPHAGUS (Gastrointestinal disorders) | 0 | 1
CHRONIC GASTROINTESTINAL BLEEDING (Gastrointestinal disorders) | 1 | 0
COLITIS (Gastrointestinal disorders) | 7 | 4
COLITIS ISCHAEMIC (Gastrointestinal disorders) | 0 | 2
COLITIS ULCERATIVE (Gastrointestinal disorders) | 1 | 0
COLONIC POLYP (Gastrointestinal disorders) | 4 | 4
CONSTIPATION (Gastrointestinal disorders) | 1 | 3
CROHN'S DISEASE (Gastrointestinal disorders) | 1 | 0
DENTAL CARIES (Gastrointestinal disorders) | 1 | 0
DIARRHOEA (Gastrointestinal disorders) | 1 | 4
DIVERTICULAR PERFORATION (Gastrointestinal disorders) | 0 | 1
DIVERTICULITIS INTESTINAL HAEMORRHAGIC (Gastrointestinal disorders) | 0 | 2
DIVERTICULUM (Gastrointestinal disorders) | 2 | 2
DIVERTICULUM INTESTINAL (Gastrointestinal disorders) | 0 | 4
DIVERTICULUM INTESTINAL HAEMORRHAGIC (Gastrointestinal disorders) | 1 | 0
DUODENAL PERFORATION (Gastrointestinal disorders) | 1 | 0
DUODENAL ULCER (Gastrointestinal disorders) | 0 | 1
DUODENAL ULCER PERFORATION (Gastrointestinal disorders) | 1 | 0
DYSPEPSIA (Gastrointestinal disorders) | 2 | 0
DYSPHAGIA (Gastrointestinal disorders) | 1 | 1
ENTERITIS (Gastrointestinal disorders) | 1 | 0
ENTEROCOLITIS HAEMORRHAGIC (Gastrointestinal disorders) | 1 | 0
ENTEROVESICAL FISTULA (Gastrointestinal disorders) | 0 | 1
FAECALOMA (Gastrointestinal disorders) | 1 | 1
GASTRIC DISORDER (Gastrointestinal disorders) | 0 | 1
GASTRIC ULCER (Gastrointestinal disorders) | 1 | 1
GASTRIC ULCER HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1
GASTRITIS (Gastrointestinal disorders) | 3 | 5
GASTRITIS EROSIVE (Gastrointestinal disorders) | 0 | 1
GASTRITIS HAEMORRHAGIC (Gastrointestinal disorders) | 1 | 0
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 14 | 13
GASTROINTESTINAL MUCOSAL EXFOLIATION (Gastrointestinal disorders) | 1 | 0
GASTROINTESTINAL ULCER HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 3 | 4
GINGIVAL BLEEDING (Gastrointestinal disorders) | 1 | 0
HAEMATEMESIS (Gastrointestinal disorders) | 0 | 1
HAEMATOCHEZIA (Gastrointestinal disorders) | 1 | 1
HAEMORRHOIDAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1
HAEMORRHOIDS (Gastrointestinal disorders) | 1 | 0
HIATUS HERNIA (Gastrointestinal disorders) | 3 | 0
ILEUS (Gastrointestinal disorders) | 1 | 2
IMPAIRED GASTRIC EMPTYING (Gastrointestinal disorders) | 1 | 1
INGUINAL HERNIA (Gastrointestinal disorders) | 13 | 4
INGUINAL HERNIA, OBSTRUCTIVE (Gastrointestinal disorders) | 1 | 0
INTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1
INTESTINAL ISCHAEMIA (Gastrointestinal disorders) | 1 | 1
INTESTINAL MASS (Gastrointestinal disorders) | 1 | 0
LARGE INTESTINE PERFORATION (Gastrointestinal disorders) | 0 | 1
LOWER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 2 | 1
MALLORY-WEISS SYNDROME (Gastrointestinal disorders) | 0 | 1
MELAENA (Gastrointestinal disorders) | 1 | 1
MESENTERIC HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0
NAUSEA (Gastrointestinal disorders) | 2 | 2
OBSTRUCTION GASTRIC (Gastrointestinal disorders) | 0 | 1
OESOPHAGEAL STENOSIS (Gastrointestinal disorders) | 1 | 0
OESOPHAGITIS (Gastrointestinal disorders) | 0 | 2
PANCREATIC MASS (Gastrointestinal disorders) | 1 | 0
PANCREATITIS (Gastrointestinal disorders) | 1 | 6
PANCREATITIS ACUTE (Gastrointestinal disorders) | 1 | 5
PANCREATITIS CHRONIC (Gastrointestinal disorders) | 0 | 2
PROCTALGIA (Gastrointestinal disorders) | 0 | 1
PROCTITIS ULCERATIVE (Gastrointestinal disorders) | 1 | 0
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 6
RECTAL POLYP (Gastrointestinal disorders) | 0 | 2
RETROPERITONEAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 1
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 10 | 6
SPIGELIAN HERNIA (Gastrointestinal disorders) | 0 | 1
STOMATITIS (Gastrointestinal disorders) | 1 | 0
UMBILICAL HERNIA (Gastrointestinal disorders) | 2 | 2
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 7 | 1
VOLVULUS (Gastrointestinal disorders) | 1 | 0
VOMITING (Gastrointestinal disorders) | 1 | 2
ADVERSE DRUG REACTION (General disorders) | 3 | 7
ASTHENIA (General disorders) | 3 | 4
CARDIAC COMPLICATION ASSOCIATED WITH DEVICE (General disorders) | 1 | 0
CARDIAC DEATH (General disorders) | 1 | 0
CATHETER SITE HAEMATOMA (General disorders) | 4 | 1
CATHETER SITE NECROSIS (General disorders) | 0 | 1
CHEST DISCOMFORT (General disorders) | 8 | 7
CHEST PAIN (General disorders) | 36 | 29
CHILLS (General disorders) | 0 | 1
COMPLICATION OF DEVICE REMOVAL (General disorders) | 1 | 0
DEATH (General disorders) | 7 | 11
DEVICE BREAKAGE (General disorders) | 1 | 1
DEVICE FAILURE (General disorders) | 0 | 1
DEVICE ISSUE (General disorders) | 1 | 1
DEVICE MALFUNCTION (General disorders) | 1 | 0
DEVICE MATERIAL ISSUE (General disorders) | 0 | 1
DISEASE PROGRESSION (General disorders) | 0 | 1
EARLY SATIETY (General disorders) | 0 | 1
FACIAL PAIN (General disorders) | 0 | 1
FATIGUE (General disorders) | 2 | 0
GAIT DISTURBANCE (General disorders) | 1 | 1
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 0 | 2
HERNIA (General disorders) | 1 | 2
HYPERTHERMIA (General disorders) | 1 | 0
IMPAIRED HEALING (General disorders) | 0 | 2
MALAISE (General disorders) | 0 | 1
MEDICAL DEVICE COMPLICATION (General disorders) | 0 | 1
MEDICAL DEVICE PAIN (General disorders) | 1 | 0
MEDICAL DEVICE SITE REACTION (General disorders) | 1 | 0
METAPLASIA (General disorders) | 0 | 1
MULTI-ORGAN FAILURE (General disorders) | 0 | 1
NON-CARDIAC CHEST PAIN (General disorders) | 76 | 83
OEDEMA PERIPHERAL (General disorders) | 1 | 2
PAIN (General disorders) | 1 | 1
PYREXIA (General disorders) | 6 | 0
STENT-GRAFT ENDOLEAK (General disorders) | 0 | 1
SUDDEN CARDIAC DEATH (General disorders) | 0 | 1
SYSTEMIC INFLAMMATORY RESPONSE SYNDROME (General disorders) | 0 | 2
THROMBOSIS IN DEVICE (General disorders) | 12 | 13
ULCER (General disorders) | 0 | 1
ACUTE HEPATIC FAILURE (Hepatobiliary disorders) | 2 | 0
BILE DUCT OBSTRUCTION (Hepatobiliary disorders) | 1 | 0
BILE DUCT STONE (Hepatobiliary disorders) | 3 | 4
BILIARY COLIC (Hepatobiliary disorders) | 0 | 2
BILIARY DYSKINESIA (Hepatobiliary disorders) | 1 | 0
CHOLANGITIS (Hepatobiliary disorders) | 1 | 0
CHOLANGITIS ACUTE (Hepatobiliary disorders) | 1 | 1
CHOLECYSTITIS (Hepatobiliary disorders) | 3 | 3
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 3 | 3
CHOLECYSTITIS CHRONIC (Hepatobiliary disorders) | 0 | 2
CHOLELITHIASIS (Hepatobiliary disorders) | 9 | 4
CIRRHOSIS ALCOHOLIC (Hepatobiliary disorders) | 1 | 0
GALLBLADDER DISORDER (Hepatobiliary disorders) | 1 | 2
HEPATIC CIRRHOSIS (Hepatobiliary disorders) | 1 | 1
HEPATIC FAILURE (Hepatobiliary disorders) | 0 | 1
HEPATIC STEATOSIS (Hepatobiliary disorders) | 1 | 0
HEPATORENAL FAILURE (Hepatobiliary disorders) | 1 | 0
ISCHAEMIC HEPATITIS (Hepatobiliary disorders) | 1 | 0
JAUNDICE (Hepatobiliary disorders) | 1 | 0
JAUNDICE CHOLESTATIC (Hepatobiliary disorders) | 1 | 0
NON-ALCOHOLIC STEATOHEPATITIS (Hepatobiliary disorders) | 0 | 1
ALLERGY TO ARTHROPOD STING (Immune system disorders) | 0 | 1
AMYLOIDOSIS (Immune system disorders) | 0 | 1
ANAPHYLACTIC REACTION (Immune system disorders) | 1 | 0
DRUG HYPERSENSITIVITY (Immune system disorders) | 3 | 0
ABDOMINAL ABSCESS (Infections and infestations) | 0 | 2
ABDOMINAL SEPSIS (Infections and infestations) | 1 | 0
ABSCESS LIMB (Infections and infestations) | 2 | 1
ABSCESS NECK (Infections and infestations) | 1 | 0
ABSCESS OF SALIVARY GLAND (Infections and infestations) | 1 | 0
ABSCESS ORAL (Infections and infestations) | 0 | 1
APPENDICITIS (Infections and infestations) | 4 | 4
ARTERIOVENOUS GRAFT SITE INFECTION (Infections and infestations) | 0 | 1
ARTHRITIS INFECTIVE (Infections and infestations) | 1 | 0
BACTERAEMIA (Infections and infestations) | 1 | 0
BACTERIAL SEPSIS (Infections and infestations) | 0 | 1
BRONCHIOLITIS (Infections and infestations) | 1 | 0
BRONCHITIS (Infections and infestations) | 6 | 3
BRONCHITIS VIRAL (Infections and infestations) | 0 | 3
BRONCHOPNEUMONIA (Infections and infestations) | 0 | 1
BURSITIS INFECTIVE (Infections and infestations) | 0 | 1
CELLULITIS (Infections and infestations) | 8 | 8
CELLULITIS OF MALE EXTERNAL GENITAL ORGAN (Infections and infestations) | 1 | 0
CHOLECYSTITIS INFECTIVE (Infections and infestations) | 0 | 2
CLOSTRIDIAL INFECTION (Infections and infestations) | 1 | 3
CLOSTRIDIUM COLITIS (Infections and infestations) | 0 | 1
CLOSTRIDIUM DIFFICILE COLITIS (Infections and infestations) | 1 | 0
CORONA VIRUS INFECTION (Infections and infestations) | 7 | 1
CYSTITIS (Infections and infestations) | 1 | 1
DEVICE RELATED INFECTION (Infections and infestations) | 1 | 1
DIABETIC FOOT INFECTION (Infections and infestations) | 0 | 1
DIVERTICULITIS (Infections and infestations) | 9 | 9
EAR INFECTION (Infections and infestations) | 0 | 1
EMPYEMA (Infections and infestations) | 0 | 1
ENDOCARDITIS (Infections and infestations) | 1 | 0
ENTEROCOCCAL BACTERAEMIA (Infections and infestations) | 0 | 1
ENTEROCOLITIS INFECTIOUS (Infections and infestations) | 1 | 1
ESCHERICHIA BACTERAEMIA (Infections and infestations) | 1 | 0
ESCHERICHIA INFECTION (Infections and infestations) | 1 | 0
ESCHERICHIA SEPSIS (Infections and infestations) | 0 | 1
ESCHERICHIA URINARY TRACT INFECTION (Infections and infestations) | 0 | 1
EXTRADURAL ABSCESS (Infections and infestations) | 0 | 1
GANGRENE (Infections and infestations) | 3 | 1
GASTRIC INFECTION (Infections and infestations) | 0 | 1
GASTROENTERITIS (Infections and infestations) | 6 | 6
GASTROENTERITIS VIRAL (Infections and infestations) | 1 | 1
HEPATITIS C (Infections and infestations) | 1 | 0
HERPES ZOSTER (Infections and infestations) | 0 | 1
HERPES ZOSTER OTICUS (Infections and infestations) | 1 | 0
IMPLANT SITE INFECTION (Infections and infestations) | 0 | 1
INCISION SITE INFECTION (Infections and infestations) | 1 | 0
INFECTED DERMAL CYST (Infections and infestations) | 1 | 0
INFECTED SKIN ULCER (Infections and infestations) | 0 | 1
INFECTIOUS PLEURAL EFFUSION (Infections and infestations) | 1 | 0
INFLUENZA (Infections and infestations) | 5 | 5
KLEBSIELLA BACTERAEMIA (Infections and infestations) | 0 | 1
KLEBSIELLA SEPSIS (Infections and infestations) | 0 | 1
LABYRINTHITIS (Infections and infestations) | 0 | 1
LIVER ABSCESS (Infections and infestations) | 2 | 1
LOBAR PNEUMONIA (Infections and infestations) | 4 | 5
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 1
LUNG INFECTION (Infections and infestations) | 0 | 1
LUNG INFECTION PSEUDOMONAL (Infections and infestations) | 0 | 1
MUSCLE ABSCESS (Infections and infestations) | 1 | 0
NECROTISING FASCIITIS (Infections and infestations) | 0 | 1
OSTEOMYELITIS (Infections and infestations) | 0 | 5
OSTEOMYELITIS CHRONIC (Infections and infestations) | 0 | 1
PERIUMBILICAL ABSCESS (Infections and infestations) | 0 | 1
PHARYNGEAL ABSCESS (Infections and infestations) | 0 | 1
PHARYNGITIS (Infections and infestations) | 0 | 1
PLEURAL INFECTION (Infections and infestations) | 1 | 0
PNEUMONIA (Infections and infestations) | 37 | 34
PNEUMONIA KLEBSIELLA (Infections and infestations) | 0 | 1
PNEUMONIA STREPTOCOCCAL (Infections and infestations) | 0 | 1
PNEUMONIA VIRAL (Infections and infestations) | 1 | 4
POST PROCEDURAL CELLULITIS (Infections and infestations) | 0 | 1
POSTOPERATIVE ABSCESS (Infections and infestations) | 1 | 0
POSTOPERATIVE WOUND INFECTION (Infections and infestations) | 1 | 0
PYELONEPHRITIS (Infections and infestations) | 1 | 2
PYELONEPHRITIS ACUTE (Infections and infestations) | 1 | 1
RHINOVIRUS INFECTION (Infections and infestations) | 1 | 0
SCROTAL ABSCESS (Infections and infestations) | 2 | 0
SEPSIS (Infections and infestations) | 19 | 14
SEPSIS SYNDROME (Infections and infestations) | 0 | 1
SEPTIC ENCEPHALOPATHY (Infections and infestations) | 1 | 0
SEPTIC SHOCK (Infections and infestations) | 2 | 4
STAPHYLOCOCCAL BACTERAEMIA (Infections and infestations) | 1 | 1
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 0 | 1
STAPHYLOCOCCAL SEPSIS (Infections and infestations) | 1 | 1
SUBCUTANEOUS ABSCESS (Infections and infestations) | 1 | 0
TESTICULAR ABSCESS (Infections and infestations) | 1 | 0
TOOTH ABSCESS (Infections and infestations) | 0 | 1
TOOTH INFECTION (Infections and infestations) | 1 | 0
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 1
URETHRITIS (Infections and infestations) | 1 | 0
URINARY TRACT INFECTION (Infections and infestations) | 10 | 14
UROSEPSIS (Infections and infestations) | 5 | 1
VIRAL INFECTION (Infections and infestations) | 2 | 0
VIRAL LABYRINTHITIS (Infections and infestations) | 1 | 0
WEST NILE VIRAL INFECTION (Infections and infestations) | 1 | 0
WOUND INFECTION (Infections and infestations) | 2 | 1
WOUND INFECTION BACTERIAL (Infections and infestations) | 1 | 0
ACETABULUM FRACTURE (Injury, poisoning and procedural complications) | 2 | 0
ADRENAL GLAND INJURY (Injury, poisoning and procedural complications) | 0 | 1
ALCOHOL POISONING (Injury, poisoning and procedural complications) | 1 | 0
ANAEMIA POSTOPERATIVE (Injury, poisoning and procedural complications) | 1 | 1
ANASTOMOTIC LEAK (Injury, poisoning and procedural complications) | 0 | 1
ANASTOMOTIC ULCER HAEMORRHAGE (Injury, poisoning and procedural complications) | 1 | 0
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 2 | 8
ARTERIAL INJURY (Injury, poisoning and procedural complications) | 0 | 1
ARTHROPOD STING (Injury, poisoning and procedural complications) | 1 | 0
ASBESTOSIS (Injury, poisoning and procedural complications) | 1 | 0
BACK INJURY (Injury, poisoning and procedural complications) | 0 | 1
CARDIAC PROCEDURE COMPLICATION (Injury, poisoning and procedural complications) | 2 | 2
CATHETER SITE HAEMATOMA (Injury, poisoning and procedural complications) | 1 | 1
CERVICAL VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 1 | 2
COMMINUTED FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
CONCUSSION (Injury, poisoning and procedural complications) | 1 | 0
CONFUSION POSTOPERATIVE (Injury, poisoning and procedural complications) | 2 | 0
CONTUSION (Injury, poisoning and procedural complications) | 0 | 2
CORONARY ARTERY REOCCLUSION (Injury, poisoning and procedural complications) | 1 | 0
CORONARY ARTERY RESTENOSIS (Injury, poisoning and procedural complications) | 28 | 20
CRANIOCEREBRAL INJURY (Injury, poisoning and procedural complications) | 1 | 1
CYSTITIS RADIATION (Injury, poisoning and procedural complications) | 0 | 1
FACIAL BONES FRACTURE (Injury, poisoning and procedural complications) | 2 | 0
FALL (Injury, poisoning and procedural complications) | 6 | 4
FEMORAL NECK FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 3 | 1
FIBULA FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
FOOT FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
FOREARM FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
GASTROINTESTINAL STOMA COMPLICATION (Injury, poisoning and procedural complications) | 1 | 0
HAEMATURIA TRAUMATIC (Injury, poisoning and procedural complications) | 0 | 1
HAND FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
HEAT EXHAUSTION (Injury, poisoning and procedural complications) | 1 | 0
HEAT STROKE (Injury, poisoning and procedural complications) | 0 | 1
HIP FRACTURE (Injury, poisoning and procedural complications) | 2 | 2
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 2 | 1
IN-STENT ARTERIAL RESTENOSIS (Injury, poisoning and procedural complications) | 2 | 1
IN-STENT CORONARY ARTERY RESTENOSIS (Injury, poisoning and procedural complications) | 8 | 18
INCISIONAL HERNIA (Injury, poisoning and procedural complications) | 0 | 1
INJURY (Injury, poisoning and procedural complications) | 2 | 1
INTENTIONAL OVERDOSE (Injury, poisoning and procedural complications) | 1 | 0
JOINT DISLOCATION (Injury, poisoning and procedural complications) | 0 | 3
LACERATION (Injury, poisoning and procedural complications) | 3 | 0
LIGAMENT RUPTURE (Injury, poisoning and procedural complications) | 2 | 0
LIMB INJURY (Injury, poisoning and procedural complications) | 2 | 1
LUMBAR VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 2 | 1
MENISCUS LESION (Injury, poisoning and procedural complications) | 0 | 2
MULTIPLE FRACTURES (Injury, poisoning and procedural complications) | 1 | 0
MULTIPLE INJURIES (Injury, poisoning and procedural complications) | 1 | 0
OVERDOSE (Injury, poisoning and procedural complications) | 1 | 1
PATELLA FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
PELVIC FRACTURE (Injury, poisoning and procedural complications) | 0 | 3
PELVIC ORGAN INJURY (Injury, poisoning and procedural complications) | 0 | 1
PERIPROSTHETIC FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
PLAQUE SHIFT (Injury, poisoning and procedural complications) | 0 | 1
POISONING (Injury, poisoning and procedural complications) | 0 | 1
POISONING DELIBERATE (Injury, poisoning and procedural complications) | 0 | 1
POST LAMINECTOMY SYNDROME (Injury, poisoning and procedural complications) | 1 | 0
POST PROCEDURAL BILE LEAK (Injury, poisoning and procedural complications) | 1 | 1
POST PROCEDURAL COMPLICATION (Injury, poisoning and procedural complications) | 1 | 1
POST PROCEDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 1 | 0
POST PROCEDURAL MYOCARDIAL INFARCTION (Injury, poisoning and procedural complications) | 11 | 6
POST-TRAUMATIC PAIN (Injury, poisoning and procedural complications) | 0 | 3
POSTOPERATIVE ILEUS (Injury, poisoning and procedural complications) | 1 | 0
POSTOPERATIVE RESPIRATORY DISTRESS (Injury, poisoning and procedural complications) | 1 | 1
PROCEDURAL HYPERTENSION (Injury, poisoning and procedural complications) | 0 | 1
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 3 | 1
PROCEDURAL VOMITING (Injury, poisoning and procedural complications) | 1 | 0
RADIUS FRACTURE (Injury, poisoning and procedural complications) | 1 | 1
RIB FRACTURE (Injury, poisoning and procedural complications) | 3 | 1
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 1 | 1
SKULL FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
SPINAL COLUMN INJURY (Injury, poisoning and procedural complications) | 1 | 0
SPINAL COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 4 | 1
SPINAL FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
STAB WOUND (Injury, poisoning and procedural complications) | 0 | 1
STRESS ECHOCARDIOGRAM ABNORMAL (Injury, poisoning and procedural complications) | 1 | 0
SUBDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 1 | 3
SUBDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 1 | 0
TENDON RUPTURE (Injury, poisoning and procedural complications) | 2 | 3
THERMAL BURN (Injury, poisoning and procedural complications) | 1 | 1
THORACIC VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
TRAUMATIC ARTHRITIS (Injury, poisoning and procedural complications) | 0 | 1
TRAUMATIC HAEMATOMA (Injury, poisoning and procedural complications) | 0 | 1
TRAUMATIC HAEMORRHAGE (Injury, poisoning and procedural complications) | 1 | 0
TRAUMATIC INTRACRANIAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 1 | 0
TRAUMATIC LUNG INJURY (Injury, poisoning and procedural complications) | 0 | 1
ULNA FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
UPPER LIMB FRACTURE (Injury, poisoning and procedural complications) | 1 | 1
URINARY RETENTION POSTOPERATIVE (Injury, poisoning and procedural complications) | 0 | 1
VASCULAR GRAFT COMPLICATION (Injury, poisoning and procedural complications) | 0 | 1
VASCULAR GRAFT OCCLUSION (Injury, poisoning and procedural complications) | 0 | 2
VASCULAR PSEUDOANEURYSM (Injury, poisoning and procedural complications) | 4 | 5
WOUND DEHISCENCE (Injury, poisoning and procedural complications) | 1 | 1
WRIST FRACTURE (Injury, poisoning and procedural complications) | 0 | 3
ARTERIOGRAM CORONARY (Investigations) | 1 | 0
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 0 | 1
BLOOD CREATINE PHOSPHOKINASE MB INCREASED (Investigations) | 1 | 1
BLOOD GLUCOSE DECREASED (Investigations) | 0 | 1
BLOOD GLUCOSE INCREASED (Investigations) | 0 | 1
BLOOD PRESSURE INCREASED (Investigations) | 1 | 1
CARDIAC ENZYMES INCREASED (Investigations) | 4 | 4
CARDIAC STRESS TEST ABNORMAL (Investigations) | 0 | 1
CORONAVIRUS TEST POSITIVE (Investigations) | 0 | 1
EJECTION FRACTION DECREASED (Investigations) | 1 | 2
ELECTROCARDIOGRAM ABNORMAL (Investigations) | 2 | 0
GLYCOSYLATED HAEMOGLOBIN INCREASED (Investigations) | 0 | 1
N-TERMINAL PROHORMONE BRAIN NATRIURETIC PEPTIDE INCREASED (Investigations) | 0 | 1
TRANSAMINASES INCREASED (Investigations) | 0 | 1
TROPONIN INCREASED (Investigations) | 6 | 2
DEHYDRATION (Metabolism and nutrition disorders) | 6 | 4
DIABETES MELLITUS (Metabolism and nutrition disorders) | 1 | 2
DIABETES MELLITUS INADEQUATE CONTROL (Metabolism and nutrition disorders) | 4 | 0
DIABETIC KETOACIDOSIS (Metabolism and nutrition disorders) | 2 | 5
FAILURE TO THRIVE (Metabolism and nutrition disorders) | 2 | 0
FLUID OVERLOAD (Metabolism and nutrition disorders) | 0 | 1
GOUT (Metabolism and nutrition disorders) | 1 | 2
HYPERAMMONAEMIA (Metabolism and nutrition disorders) | 1 | 0
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 0 | 1
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 3 | 1
HYPERKALAEMIA (Metabolism and nutrition disorders) | 3 | 0
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 2 | 4
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 | 3
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 0 | 1
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 | 5
HYPOVOLAEMIA (Metabolism and nutrition disorders) | 2 | 0
KETOACIDOSIS (Metabolism and nutrition disorders) | 1 | 0
LACTIC ACIDOSIS (Metabolism and nutrition disorders) | 1 | 1
MALNUTRITION (Metabolism and nutrition disorders) | 1 | 0
METABOLIC ACIDOSIS (Metabolism and nutrition disorders) | 1 | 0
METABOLIC SYNDROME (Metabolism and nutrition disorders) | 1 | 0
OBESITY (Metabolism and nutrition disorders) | 1 | 4
TYPE 2 DIABETES MELLITUS (Metabolism and nutrition disorders) | 0 | 1
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 7 | 6
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 6 | 3
ARTHROPATHY (Musculoskeletal and connective tissue disorders) | 1 | 0
BACK PAIN (Musculoskeletal and connective tissue disorders) | 10 | 9
BURSITIS (Musculoskeletal and connective tissue disorders) | 0 | 1
CERVICAL SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 2 | 4
CHONDROCALCINOSIS PYROPHOSPHATE (Musculoskeletal and connective tissue disorders) | 0 | 1
COSTOCHONDRITIS (Musculoskeletal and connective tissue disorders) | 1 | 2
FACET JOINT SYNDROME (Musculoskeletal and connective tissue disorders) | 0 | 1
FEMOROACETABULAR IMPINGEMENT (Musculoskeletal and connective tissue disorders) | 1 | 0
FOOT DEFORMITY (Musculoskeletal and connective tissue disorders) | 2 | 0
INTERVERTEBRAL DISC DEGENERATION (Musculoskeletal and connective tissue disorders) | 2 | 1
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 2 | 1
JOINT SWELLING (Musculoskeletal and connective tissue disorders) | 1 | 0
LUMBAR SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 4 | 4
MUSCLE NECROSIS (Musculoskeletal and connective tissue disorders) | 0 | 1
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 1 | 1
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 2 | 2
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 1 | 5
MUSCULOSKELETAL DISCOMFORT (Musculoskeletal and connective tissue disorders) | 1 | 0
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 4 | 8
MYALGIA (Musculoskeletal and connective tissue disorders) | 0 | 2
MYOPATHY (Musculoskeletal and connective tissue disorders) | 0 | 1
NECK PAIN (Musculoskeletal and connective tissue disorders) | 3 | 1
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 29 | 24
OSTEOCHONDROSIS (Musculoskeletal and connective tissue disorders) | 1 | 1
OSTEONECROSIS (Musculoskeletal and connective tissue disorders) | 1 | 0
OSTEOPOROSIS (Musculoskeletal and connective tissue disorders) | 0 | 1
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 4 | 5
POLYMYALGIA RHEUMATICA (Musculoskeletal and connective tissue disorders) | 1 | 1
PSEUDARTHROSIS (Musculoskeletal and connective tissue disorders) | 1 | 0
RHABDOMYOLYSIS (Musculoskeletal and connective tissue disorders) | 3 | 0
RHEUMATOID ARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 2
ROTATOR CUFF SYNDROME (Musculoskeletal and connective tissue disorders) | 6 | 6
SPINAL COLUMN STENOSIS (Musculoskeletal and connective tissue disorders) | 3 | 3
SPINAL DISORDER (Musculoskeletal and connective tissue disorders) | 1 | 1
SPINAL OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 2 | 5
TENDONITIS (Musculoskeletal and connective tissue disorders) | 0 | 1
TENOSYNOVITIS STENOSANS (Musculoskeletal and connective tissue disorders) | 0 | 1
TRIGGER FINGER (Musculoskeletal and connective tissue disorders) | 0 | 3
VERTEBRAL FORAMINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 0 | 2
ACUTE MYELOID LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
ACUTE PROMYELOCYTIC LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
ADENOCARCINOMA PANCREAS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
B-CELL LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
B-CELL LYMPHOMA STAGE I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
B-CELL LYMPHOMA STAGE IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 6
BENIGN NEOPLASM OF BLADDER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
BENIGN SOFT TISSUE NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
BILE DUCT CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
BLADDER CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 4
BLADDER NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
BOWEN'S DISEASE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 5
BREAST CANCER IN SITU (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
BREAST CANCER STAGE II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
BRONCHIAL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
CHRONIC LYMPHOCYTIC LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
COLON ADENOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
COLON CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 5
ENDOMETRIAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
ENDOMETRIAL CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
GASTROINTESTINAL STROMAL TUMOUR (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
HEPATIC NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
HEPATIC NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
HEPATIC NEOPLASM MALIGNANT RECURRENT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
INTESTINAL ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
LARYNGEAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
LUNG ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
LUNG ADENOCARCINOMA METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
LUNG CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
LUNG CARCINOMA CELL TYPE UNSPECIFIED STAGE IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
LUNG NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
LUNG NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 4
LUNG SQUAMOUS CELL CARCINOMA STAGE UNSPECIFIED (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
MALIGNANT GLIOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
MALIGNANT MELANOMA IN SITU (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
MALIGNANT PLEURAL EFFUSION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
MANTLE CELL LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
MELANOCYTIC NAEVUS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
MENINGIOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
METASTASES TO CENTRAL NERVOUS SYSTEM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
METASTASES TO LIVER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
METASTATIC MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
METASTATIC NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
MUELLER'S MIXED TUMOUR (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
MULTIPLE MYELOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
MYELODYSPLASTIC SYNDROME (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
MYELOFIBROSIS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
NEOPLASM SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
NEUROENDOCRINE CARCINOMA METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
NON-HODGKIN'S LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
NON-SMALL CELL LUNG CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
OESOPHAGEAL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3
OROPHARYNGEAL CANCER STAGE UNSPECIFIED (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
OVARIAN CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
OVARIAN CANCER STAGE III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
OVARIAN NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
PANCREATIC CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
PANCREATIC CARCINOMA METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
PARATHYROID TUMOUR BENIGN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
PERITONEAL CARCINOMA METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
PLASMACYTOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
PLEURAL MESOTHELIOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
PLEURAL MESOTHELIOMA MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 | 6
PROSTATE CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
RECTAL ADENOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
RECTAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
RENAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
RENAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
SALIVARY GLAND CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
SALIVARY GLAND NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
SEBORRHOEIC KERATOSIS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
SKIN CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
SMALL CELL LUNG CANCER STAGE UNSPECIFIED (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
SQUAMOUS CELL CARCINOMA OF SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3
THYROID CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
TRACHEAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
TRANSITIONAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
URETERIC CANCER RECURRENT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
AMNESIA (Nervous system disorders) | 2 | 1
APHASIA (Nervous system disorders) | 0 | 2
BRAIN INJURY (Nervous system disorders) | 0 | 1
BRAIN MASS (Nervous system disorders) | 0 | 1
BRAIN STEM INFARCTION (Nervous system disorders) | 1 | 0
CAROTID ARTERY OCCLUSION (Nervous system disorders) | 1 | 0
CAROTID ARTERY STENOSIS (Nervous system disorders) | 11 | 8
CARPAL TUNNEL SYNDROME (Nervous system disorders) | 3 | 2
CENTRAL NERVOUS SYSTEM LESION (Nervous system disorders) | 1 | 0
CEREBELLAR INFARCTION (Nervous system disorders) | 0 | 2
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 2 | 3
CEREBRAL INFARCTION (Nervous system disorders) | 0 | 1
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 15 | 21
CEREBROVASCULAR DISORDER (Nervous system disorders) | 0 | 1
CERVICAL CORD COMPRESSION (Nervous system disorders) | 1 | 0
CERVICAL MYELOPATHY (Nervous system disorders) | 1 | 1
CERVICOBRACHIAL SYNDROME (Nervous system disorders) | 0 | 3
CHRONIC INFLAMMATORY DEMYELINATING POLYRADICULONEUROPATHY (Nervous system disorders) | 1 | 0
COMPLICATED MIGRAINE (Nervous system disorders) | 2 | 1
CONVULSION (Nervous system disorders) | 3 | 2
CRANIAL NERVE DISORDER (Nervous system disorders) | 1 | 0
CUBITAL TUNNEL SYNDROME (Nervous system disorders) | 0 | 1
DEMENTIA (Nervous system disorders) | 0 | 1
DEMENTIA ALZHEIMER'S TYPE (Nervous system disorders) | 1 | 1
DEPRESSED LEVEL OF CONSCIOUSNESS (Nervous system disorders) | 1 | 0
DIZZINESS (Nervous system disorders) | 4 | 7
DYSARTHRIA (Nervous system disorders) | 1 | 0
EMBOLIC CEREBRAL INFARCTION (Nervous system disorders) | 1 | 0
ENCEPHALOPATHY (Nervous system disorders) | 5 | 2
EPILEPSY (Nervous system disorders) | 0 | 1
GRAND MAL CONVULSION (Nervous system disorders) | 2 | 1
GUILLAIN-BARRE SYNDROME (Nervous system disorders) | 0 | 1
HAEMORRHAGE INTRACRANIAL (Nervous system disorders) | 1 | 3
HAEMORRHAGIC STROKE (Nervous system disorders) | 1 | 0
HEADACHE (Nervous system disorders) | 3 | 1
HYPOAESTHESIA (Nervous system disorders) | 1 | 0
IIIRD NERVE PARALYSIS (Nervous system disorders) | 1 | 0
INTRACRANIAL ANEURYSM (Nervous system disorders) | 0 | 1
INTRAVENTRICULAR HAEMORRHAGE (Nervous system disorders) | 1 | 0
ISCHAEMIC STROKE (Nervous system disorders) | 1 | 3
LUMBAR RADICULOPATHY (Nervous system disorders) | 0 | 1
METABOLIC ENCEPHALOPATHY (Nervous system disorders) | 6 | 1
MIGRAINE (Nervous system disorders) | 1 | 0
MIGRAINE WITH AURA (Nervous system disorders) | 1 | 0
MONONEURITIS (Nervous system disorders) | 1 | 0
MULTIPLE SCLEROSIS (Nervous system disorders) | 0 | 1
NEURODEGENERATIVE DISORDER (Nervous system disorders) | 1 | 0
PARKINSON'S DISEASE (Nervous system disorders) | 0 | 1
PARTIAL SEIZURES (Nervous system disorders) | 0 | 1
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 1 | 0
POSTERIOR REVERSIBLE ENCEPHALOPATHY SYNDROME (Nervous system disorders) | 0 | 1
PRESYNCOPE (Nervous system disorders) | 5 | 5
RADICULOPATHY (Nervous system disorders) | 1 | 0
SCIATICA (Nervous system disorders) | 3 | 3
SENSORY LOSS (Nervous system disorders) | 0 | 1
SUBARACHNOID HAEMORRHAGE (Nervous system disorders) | 0 | 4
SYNCOPE (Nervous system disorders) | 15 | 17
TOXIC ENCEPHALOPATHY (Nervous system disorders) | 0 | 1
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 14 | 11
TREMOR (Nervous system disorders) | 0 | 1
TRIGEMINAL NEURALGIA (Nervous system disorders) | 0 | 1
TYPICAL AURA WITHOUT HEADACHE (Nervous system disorders) | 1 | 0
ULNAR TUNNEL SYNDROME (Nervous system disorders) | 0 | 1
UNRESPONSIVE TO STIMULI (Nervous system disorders) | 1 | 0
VERTEBRAL ARTERY STENOSIS (Nervous system disorders) | 1 | 0
VIITH NERVE PARALYSIS (Nervous system disorders) | 0 | 1
ABORTION SPONTANEOUS (Pregnancy, puerperium and perinatal conditions) | 0 | 1
ALCOHOL WITHDRAWAL SYNDROME (Psychiatric disorders) | 1 | 0
ANXIETY (Psychiatric disorders) | 0 | 2
COMPLETED SUICIDE (Psychiatric disorders) | 1 | 0
CONFUSIONAL STATE (Psychiatric disorders) | 1 | 1
CONVERSION DISORDER (Psychiatric disorders) | 1 | 0
DELIRIUM (Psychiatric disorders) | 2 | 2
DEPRESSION (Psychiatric disorders) | 2 | 1
DEPRESSION SUICIDAL (Psychiatric disorders) | 0 | 1
IMPAIRED SELF-CARE (Psychiatric disorders) | 0 | 1
INTENTIONAL SELF-INJURY (Psychiatric disorders) | 0 | 1
MENTAL DISORDER DUE TO A GENERAL MEDICAL CONDITION (Psychiatric disorders) | 1 | 0
MENTAL STATUS CHANGES (Psychiatric disorders) | 5 | 5
POST-TRAUMATIC AMNESTIC DISORDER (Psychiatric disorders) | 0 | 1
PSYCHOGENIC PAIN DISORDER (Psychiatric disorders) | 1 | 0
SOMATOFORM DISORDER (Psychiatric disorders) | 0 | 1
SUICIDAL IDEATION (Psychiatric disorders) | 1 | 1
SUICIDE ATTEMPT (Psychiatric disorders) | 0 | 1
BLADDER NECK OBSTRUCTION (Renal and urinary disorders) | 1 | 0
BLADDER OBSTRUCTION (Renal and urinary disorders) | 0 | 1
BLADDER PERFORATION (Renal and urinary disorders) | 0 | 1
CALCULUS BLADDER (Renal and urinary disorders) | 1 | 0
CALCULUS URETERIC (Renal and urinary disorders) | 1 | 2
CYSTITIS HAEMORRHAGIC (Renal and urinary disorders) | 1 | 0
DYSURIA (Renal and urinary disorders) | 2 | 0
HAEMATURIA (Renal and urinary disorders) | 5 | 5
HYDRONEPHROSIS (Renal and urinary disorders) | 1 | 0
HYPERTONIC BLADDER (Renal and urinary disorders) | 0 | 1
NEPHROLITHIASIS (Renal and urinary disorders) | 7 | 7
OBSTRUCTIVE UROPATHY (Renal and urinary disorders) | 0 | 2
RENAL ARTERY STENOSIS (Renal and urinary disorders) | 2 | 3
RENAL FAILURE (Renal and urinary disorders) | 1 | 1
RENAL FAILURE ACUTE (Renal and urinary disorders) | 27 | 22
RENAL FAILURE CHRONIC (Renal and urinary disorders) | 1 | 4
RENAL HAEMORRHAGE (Renal and urinary disorders) | 0 | 1
RENAL IMPAIRMENT (Renal and urinary disorders) | 1 | 0
RENAL MASS (Renal and urinary disorders) | 1 | 1
URETERIC STENOSIS (Renal and urinary disorders) | 0 | 1
URINARY INCONTINENCE (Renal and urinary disorders) | 1 | 3
URINARY RETENTION (Renal and urinary disorders) | 0 | 2
ACQUIRED HYDROCELE (Reproductive system and breast disorders) | 1 | 0
BENIGN PROSTATIC HYPERPLASIA (Reproductive system and breast disorders) | 5 | 7
ENDOMETRIAL HYPERPLASIA (Reproductive system and breast disorders) | 1 | 0
EPIDIDYMITIS (Reproductive system and breast disorders) | 1 | 3
ERECTILE DYSFUNCTION (Reproductive system and breast disorders) | 0 | 2
GENITAL PAIN (Reproductive system and breast disorders) | 1 | 0
GYNAECOMASTIA (Reproductive system and breast disorders) | 0 | 1
MENORRHAGIA (Reproductive system and breast disorders) | 1 | 0
PELVIC PROLAPSE (Reproductive system and breast disorders) | 1 | 0
PROSTATITIS (Reproductive system and breast disorders) | 0 | 1
PROSTATOMEGALY (Reproductive system and breast disorders) | 0 | 1
UTERINE OBSTRUCTION (Reproductive system and breast disorders) | 0 | 1
UTERINE POLYP (Reproductive system and breast disorders) | 1 | 0
VAGINAL HAEMORRHAGE (Reproductive system and breast disorders) | 0 | 1
VAGINAL PROLAPSE (Reproductive system and breast disorders) | 1 | 1
VULVAR DYSPLASIA (Reproductive system and breast disorders) | 1 | 0
ACQUIRED DIAPHRAGMATIC EVENTRATION (Respiratory, thoracic and mediastinal disorders) | 1 | 0
ACUTE INTERSTITIAL PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
ACUTE PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 1 | 1
ACUTE RESPIRATORY DISTRESS SYNDROME (Respiratory, thoracic and mediastinal disorders) | 0 | 1
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 15 | 18
ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 1 | 0
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 3 | 1
ATELECTASIS (Respiratory, thoracic and mediastinal disorders) | 0 | 2
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 16 | 17
CHRONIC RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 | 0
DIAPHRAGMATIC PARALYSIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 21 | 24
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 9 | 10
EMPHYSEMA (Respiratory, thoracic and mediastinal disorders) | 1 | 0
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 2 | 1
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 0 | 1
HAEMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 | 1
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 1 | 1
INTERSTITIAL LUNG DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 | 0
LUNG INFILTRATION (Respiratory, thoracic and mediastinal disorders) | 0 | 1
NASAL SEPTUM DEVIATION (Respiratory, thoracic and mediastinal disorders) | 1 | 0
NASAL TURBINATE HYPERTROPHY (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PHARYNGEAL MASS (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 4 | 2
PLEURAL FIBROSIS (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PLEURITIC PAIN (Respiratory, thoracic and mediastinal disorders) | 1 | 2
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 2 | 1
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 3 | 2
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 8 | 5
PULMONARY FIBROSIS (Respiratory, thoracic and mediastinal disorders) | 2 | 0
PULMONARY HYPERTENSION (Respiratory, thoracic and mediastinal disorders) | 1 | 2
PULMONARY MASS (Respiratory, thoracic and mediastinal disorders) | 0 | 2
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 1 | 3
PULMONARY TOXICITY (Respiratory, thoracic and mediastinal disorders) | 1 | 0
RESPIRATORY ARREST (Respiratory, thoracic and mediastinal disorders) | 0 | 1
RESPIRATORY DISTRESS (Respiratory, thoracic and mediastinal disorders) | 3 | 1
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 12 | 5
SLEEP APNOEA SYNDROME (Respiratory, thoracic and mediastinal disorders) | 1 | 3
ANGIOEDEMA (Skin and subcutaneous tissue disorders) | 1 | 2
DECUBITUS ULCER (Skin and subcutaneous tissue disorders) | 1 | 0
DIGITAL ULCER (Skin and subcutaneous tissue disorders) | 0 | 1
DRUG ERUPTION (Skin and subcutaneous tissue disorders) | 0 | 1
DRY GANGRENE (Skin and subcutaneous tissue disorders) | 0 | 1
LEUKOCYTOCLASTIC VASCULITIS (Skin and subcutaneous tissue disorders) | 0 | 1
PRECANCEROUS SKIN LESION (Skin and subcutaneous tissue disorders) | 1 | 0
RASH (Skin and subcutaneous tissue disorders) | 0 | 1
SCAR PAIN (Skin and subcutaneous tissue disorders) | 0 | 1
SKIN ULCER (Skin and subcutaneous tissue disorders) | 1 | 3
AORTIC STENT INSERTION (Surgical and medical procedures) | 1 | 0
CORONARY ARTERIAL STENT INSERTION (Surgical and medical procedures) | 1 | 0
HERNIA REPAIR (Surgical and medical procedures) | 0 | 1
HIP ARTHROPLASTY (Surgical and medical procedures) | 1 | 1
HYSTERECTOMY (Surgical and medical procedures) | 1 | 0
IMPLANTABLE DEFIBRILLATOR INSERTION (Surgical and medical procedures) | 0 | 1
KNEE ARTHROPLASTY (Surgical and medical procedures) | 0 | 1
NASAL OPERATION (Surgical and medical procedures) | 1 | 0
NECK SURGERY (Surgical and medical procedures) | 0 | 1
PERCUTANEOUS CORONARY INTERVENTION (Surgical and medical procedures) | 1 | 0
ROTATOR CUFF REPAIR (Surgical and medical procedures) | 0 | 1
SURGERY (Surgical and medical procedures) | 0 | 1
ACCELERATED HYPERTENSION (Vascular disorders) | 1 | 1
ANEURYSM (Vascular disorders) | 0 | 1
AORTIC ANEURYSM (Vascular disorders) | 1 | 4
AORTIC DISSECTION (Vascular disorders) | 0 | 1
AORTIC STENOSIS (Vascular disorders) | 4 | 3
ARTERIAL DISORDER (Vascular disorders) | 1 | 0
ARTERIAL HAEMORRHAGE (Vascular disorders) | 0 | 1
ARTERIAL OCCLUSIVE DISEASE (Vascular disorders) | 1 | 0
ARTERIAL THROMBOSIS LIMB (Vascular disorders) | 0 | 1
ARTERIOSCLEROSIS (Vascular disorders) | 2 | 1
DEEP VEIN THROMBOSIS (Vascular disorders) | 4 | 4
EMBOLISM ARTERIAL (Vascular disorders) | 1 | 0
FEMORAL ARTERIAL STENOSIS (Vascular disorders) | 2 | 0
FEMORAL ARTERY ANEURYSM (Vascular disorders) | 1 | 0
FEMORAL ARTERY DISSECTION (Vascular disorders) | 1 | 0
FEMORAL ARTERY OCCLUSION (Vascular disorders) | 2 | 2
HAEMATOMA (Vascular disorders) | 1 | 2
HYPERTENSION (Vascular disorders) | 6 | 4
HYPERTENSIVE CRISIS (Vascular disorders) | 5 | 10
HYPERTENSIVE EMERGENCY (Vascular disorders) | 2 | 1
HYPOTENSION (Vascular disorders) | 5 | 5
HYPOVOLAEMIC SHOCK (Vascular disorders) | 0 | 1
ILIAC ARTERY STENOSIS (Vascular disorders) | 0 | 1
INTERMITTENT CLAUDICATION (Vascular disorders) | 8 | 3
LERICHE SYNDROME (Vascular disorders) | 0 | 1
MALIGNANT HYPERTENSION (Vascular disorders) | 1 | 0
ORTHOSTATIC HYPOTENSION (Vascular disorders) | 4 | 3
PELVIC VENOUS THROMBOSIS (Vascular disorders) | 1 | 0
PERIPHERAL ARTERIAL OCCLUSIVE DISEASE (Vascular disorders) | 7 | 15
PERIPHERAL ISCHAEMIA (Vascular disorders) | 0 | 2
PERIPHERAL VASCULAR DISORDER (Vascular disorders) | 5 | 5
SHOCK (Vascular disorders) | 1 | 0
THROMBOPHLEBITIS (Vascular disorders) | 0 | 1
THROMBOSIS (Vascular disorders) | 1 | 0
VARICOSE VEIN (Vascular disorders) | 1 | 0
VASCULAR STENOSIS (Vascular disorders) | 0 | 1
VENOUS RECANALISATION (Vascular disorders) | 1 | 0
VENOUS THROMBOSIS LIMB (Vascular disorders) | 1 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Absorb BVS (N=1296) | XIENCE (N=1308)
ANAEMIA (Blood and lymphatic system disorders) | 23 | 29
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 0 | 2
HAEMORRHAGIC ANAEMIA (Blood and lymphatic system disorders) | 3 | 2
HAEMORRHAGIC DIATHESIS (Blood and lymphatic system disorders) | 1 | 0
IRON DEFICIENCY ANAEMIA (Blood and lymphatic system disorders) | 7 | 9
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 0 | 5
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 2 | 1
NEUTROPENIA (Blood and lymphatic system disorders) | 0 | 1
NORMOCHROMIC NORMOCYTIC ANAEMIA (Blood and lymphatic system disorders) | 2 | 0
PANCYTOPENIA (Blood and lymphatic system disorders) | 0 | 1
SPLENIC GRANULOMA (Blood and lymphatic system disorders) | 0 | 1
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 2 | 1
ACCELERATED IDIOVENTRICULAR RHYTHM (Cardiac disorders) | 1 | 0
ACUTE CORONARY SYNDROME (Cardiac disorders) | 10 | 8
ACUTE LEFT VENTRICULAR FAILURE (Cardiac disorders) | 1 | 1
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 28 | 28
ANGINA PECTORIS (Cardiac disorders) | 342 | 332
ANGINA UNSTABLE (Cardiac disorders) | 61 | 70
AORTIC VALVE INCOMPETENCE (Cardiac disorders) | 2 | 0
AORTIC VALVE STENOSIS (Cardiac disorders) | 2 | 4
ARRHYTHMIA (Cardiac disorders) | 4 | 4
ARTERIOSCLEROSIS CORONARY ARTERY (Cardiac disorders) | 4 | 3
ARTERIOSPASM CORONARY (Cardiac disorders) | 0 | 3
ATRIAL FIBRILLATION (Cardiac disorders) | 78 | 57
ATRIAL FLUTTER (Cardiac disorders) | 4 | 6
ATRIAL TACHYCARDIA (Cardiac disorders) | 3 | 0
ATRIAL THROMBOSIS (Cardiac disorders) | 0 | 1
ATRIOVENTRICULAR BLOCK (Cardiac disorders) | 0 | 1
ATRIOVENTRICULAR BLOCK COMPLETE (Cardiac disorders) | 2 | 3
ATRIOVENTRICULAR BLOCK SECOND DEGREE (Cardiac disorders) | 1 | 0
BRADYCARDIA (Cardiac disorders) | 21 | 16
BUNDLE BRANCH BLOCK LEFT (Cardiac disorders) | 1 | 2
BUNDLE BRANCH BLOCK RIGHT (Cardiac disorders) | 0 | 1
CARDIAC ANEURYSM (Cardiac disorders) | 1 | 0
CARDIAC ARREST (Cardiac disorders) | 10 | 4
CARDIAC FAILURE (Cardiac disorders) | 16 | 5
CARDIAC FAILURE ACUTE (Cardiac disorders) | 6 | 6
CARDIAC FAILURE CHRONIC (Cardiac disorders) | 5 | 2
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 33 | 29
CARDIAC FLUTTER (Cardiac disorders) | 0 | 1
CARDIAC PERFORATION (Cardiac disorders) | 1 | 0
CARDIAC TAMPONADE (Cardiac disorders) | 1 | 0
CARDIAC VALVE DISEASE (Cardiac disorders) | 0 | 1
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 0 | 2
CARDIOGENIC SHOCK (Cardiac disorders) | 5 | 0
CARDIOMYOPATHY (Cardiac disorders) | 3 | 3
CARDIOPULMONARY FAILURE (Cardiac disorders) | 0 | 1
CARDIOVASCULAR DISORDER (Cardiac disorders) | 1 | 0
CHRONOTROPIC INCOMPETENCE (Cardiac disorders) | 1 | 1
CONGESTIVE CARDIOMYOPATHY (Cardiac disorders) | 0 | 1
COR PULMONALE (Cardiac disorders) | 1 | 0
CORONARY ARTERY ANEURYSM (Cardiac disorders) | 1 | 0
CORONARY ARTERY DISEASE (Cardiac disorders) | 49 | 47
CORONARY ARTERY DISSECTION (Cardiac disorders) | 92 | 63
CORONARY ARTERY EMBOLISM (Cardiac disorders) | 1 | 1
CORONARY ARTERY OCCLUSION (Cardiac disorders) | 8 | 4
CORONARY ARTERY PERFORATION (Cardiac disorders) | 2 | 1
CORONARY ARTERY STENOSIS (Cardiac disorders) | 16 | 17
CORONARY ARTERY THROMBOSIS (Cardiac disorders) | 2 | 1
CYANOSIS (Cardiac disorders) | 1 | 0
DIASTOLIC DYSFUNCTION (Cardiac disorders) | 0 | 1
EXTRASYSTOLES (Cardiac disorders) | 2 | 0
HEART VALVE INCOMPETENCE (Cardiac disorders) | 0 | 1
HYPERTENSIVE HEART DISEASE (Cardiac disorders) | 0 | 1
HYPERTROPHIC CARDIOMYOPATHY (Cardiac disorders) | 1 | 0
IN-STENT CORONARY ARTERY RESTENOSIS (Cardiac disorders) | 1 | 0
INTRACARDIAC THROMBUS (Cardiac disorders) | 1 | 1
INTRAPERICARDIAL THROMBOSIS (Cardiac disorders) | 1 | 0
ISCHAEMIC CARDIOMYOPATHY (Cardiac disorders) | 5 | 9
LEFT VENTRICULAR DYSFUNCTION (Cardiac disorders) | 2 | 1
LEFT VENTRICULAR HYPERTROPHY (Cardiac disorders) | 1 | 0
MICROVASCULAR ANGINA (Cardiac disorders) | 0 | 1
MITRAL VALVE INCOMPETENCE (Cardiac disorders) | 7 | 2
MITRAL VALVE PROLAPSE (Cardiac disorders) | 2 | 0
MITRAL VALVE STENOSIS (Cardiac disorders) | 1 | 0
MYOCARDIAL INFARCTION (Cardiac disorders) | 75 | 59
MYOCARDIAL ISCHAEMIA (Cardiac disorders) | 10 | 6
MYOCARDITIS (Cardiac disorders) | 0 | 1
MYOPERICARDITIS (Cardiac disorders) | 0 | 1
NODAL ARRHYTHMIA (Cardiac disorders) | 0 | 2
PALPITATIONS (Cardiac disorders) | 28 | 34
PERICARDIAL EFFUSION (Cardiac disorders) | 2 | 2
PERICARDIAL HAEMORRHAGE (Cardiac disorders) | 0 | 1
PERICARDITIS (Cardiac disorders) | 4 | 6
PRINZMETAL ANGINA (Cardiac disorders) | 2 | 1
PULSELESS ELECTRICAL ACTIVITY (Cardiac disorders) | 0 | 1
RESTRICTIVE CARDIOMYOPATHY (Cardiac disorders) | 0 | 1
SICK SINUS SYNDROME (Cardiac disorders) | 6 | 4
SINUS ARREST (Cardiac disorders) | 1 | 0
SINUS BRADYCARDIA (Cardiac disorders) | 4 | 3
SINUS TACHYCARDIA (Cardiac disorders) | 2 | 0
STRESS CARDIOMYOPATHY (Cardiac disorders) | 2 | 0
SUPRAVENTRICULAR EXTRASYSTOLES (Cardiac disorders) | 1 | 1
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 5 | 8
TACHYARRHYTHMIA (Cardiac disorders) | 1 | 0
TACHYCARDIA (Cardiac disorders) | 8 | 5
TRICUSPID VALVE INCOMPETENCE (Cardiac disorders) | 1 | 0
VENTRICULAR ARRHYTHMIA (Cardiac disorders) | 0 | 2
VENTRICULAR EXTRASYSTOLES (Cardiac disorders) | 6 | 4
VENTRICULAR FIBRILLATION (Cardiac disorders) | 6 | 1
VENTRICULAR TACHYCARDIA (Cardiac disorders) | 14 | 10
ARTERIOVENOUS MALFORMATION (Congenital, familial and genetic disorders) | 1 | 1
ATRIAL SEPTAL DEFECT (Congenital, familial and genetic disorders) | 2 | 0
CORNEAL DYSTROPHY (Congenital, familial and genetic disorders) | 1 | 0
GASTROINTESTINAL ARTERIOVENOUS MALFORMATION (Congenital, familial and genetic disorders) | 0 | 1
HYDROCELE (Congenital, familial and genetic disorders) | 2 | 1
PERONEAL MUSCULAR ATROPHY (Congenital, familial and genetic disorders) | 0 | 1
PHIMOSIS (Congenital, familial and genetic disorders) | 0 | 2
URACHAL ABNORMALITY (Congenital, familial and genetic disorders) | 0 | 1
CERUMEN IMPACTION (Ear and labyrinth disorders) | 1 | 3
DEAFNESS (Ear and labyrinth disorders) | 1 | 0
DEAFNESS UNILATERAL (Ear and labyrinth disorders) | 2 | 1
EAR CONGESTION (Ear and labyrinth disorders) | 1 | 0
EAR HAEMORRHAGE (Ear and labyrinth disorders) | 0 | 1
EAR PAIN (Ear and labyrinth disorders) | 1 | 1
EUSTACHIAN TUBE DYSFUNCTION (Ear and labyrinth disorders) | 0 | 1
NEUROSENSORY HYPOACUSIS (Ear and labyrinth disorders) | 1 | 0
TINNITUS (Ear and labyrinth disorders) | 1 | 1
TYMPANIC MEMBRANE PERFORATION (Ear and labyrinth disorders) | 1 | 0
VERTIGO (Ear and labyrinth disorders) | 8 | 14
VERTIGO POSITIONAL (Ear and labyrinth disorders) | 2 | 4
ADRENAL INSUFFICIENCY (Endocrine disorders) | 1 | 0
ADRENAL MASS (Endocrine disorders) | 0 | 1
CARCINOID SYNDROME (Endocrine disorders) | 0 | 1
GOITRE (Endocrine disorders) | 0 | 1
HYPERPARATHYROIDISM (Endocrine disorders) | 0 | 1
HYPERTHYROIDISM (Endocrine disorders) | 0 | 1
HYPOGONADISM (Endocrine disorders) | 1 | 0
HYPOTHYROIDIC GOITRE (Endocrine disorders) | 0 | 1
HYPOTHYROIDISM (Endocrine disorders) | 1 | 4
SECONDARY HYPOGONADISM (Endocrine disorders) | 1 | 0
THYROID MASS (Endocrine disorders) | 0 | 1
ABNORMAL SENSATION IN EYE (Eye disorders) | 0 | 1
AGE-RELATED MACULAR DEGENERATION (Eye disorders) | 0 | 1
AMAUROSIS FUGAX (Eye disorders) | 1 | 2
BLINDNESS (Eye disorders) | 0 | 1
BLINDNESS TRANSIENT (Eye disorders) | 0 | 1
CATARACT (Eye disorders) | 10 | 8
CONJUNCTIVAL HAEMORRHAGE (Eye disorders) | 0 | 2
CONJUNCTIVITIS (Eye disorders) | 0 | 1
DIABETIC RETINOPATHY (Eye disorders) | 0 | 1
DIPLOPIA (Eye disorders) | 1 | 3
DRY EYE (Eye disorders) | 0 | 1
EYE HAEMORRHAGE (Eye disorders) | 2 | 2
EYE PAIN (Eye disorders) | 1 | 0
GLAUCOMA (Eye disorders) | 1 | 1
LACRIMAL DISORDER (Eye disorders) | 1 | 0
MACULAR DEGENERATION (Eye disorders) | 0 | 1
MACULAR FIBROSIS (Eye disorders) | 0 | 1
MACULAR OEDEMA (Eye disorders) | 0 | 1
OCULAR HYPERAEMIA (Eye disorders) | 0 | 1
RETINAL ARTERY EMBOLISM (Eye disorders) | 0 | 1
RETINAL DETACHMENT (Eye disorders) | 0 | 3
RETINAL DISORDER (Eye disorders) | 0 | 1
RETINAL TEAR (Eye disorders) | 0 | 1
RETINOPATHY PROLIFERATIVE (Eye disorders) | 0 | 1
TOLOSA-HUNT SYNDROME (Eye disorders) | 0 | 1
VISION BLURRED (Eye disorders) | 2 | 5
VISUAL IMPAIRMENT (Eye disorders) | 0 | 1
VITREOUS DETACHMENT (Eye disorders) | 0 | 2
VITREOUS HAEMORRHAGE (Eye disorders) | 0 | 3
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 2 | 4
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 1 | 1
ABDOMINAL HERNIA (Gastrointestinal disorders) | 3 | 0
ABDOMINAL MASS (Gastrointestinal disorders) | 1 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 15 | 18
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 1 | 3
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 16 | 7
ANAL FISSURE (Gastrointestinal disorders) | 0 | 1
ANAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1
APPENDIX DISORDER (Gastrointestinal disorders) | 0 | 1
ASCITES (Gastrointestinal disorders) | 1 | 1
BARRETT'S OESOPHAGUS (Gastrointestinal disorders) | 0 | 2
BOWEL MOVEMENT IRREGULARITY (Gastrointestinal disorders) | 1 | 0
CHRONIC GASTROINTESTINAL BLEEDING (Gastrointestinal disorders) | 1 | 0
COLITIS (Gastrointestinal disorders) | 7 | 5
COLITIS ISCHAEMIC (Gastrointestinal disorders) | 0 | 2
COLITIS ULCERATIVE (Gastrointestinal disorders) | 1 | 0
COLONIC POLYP (Gastrointestinal disorders) | 5 | 8
CONSTIPATION (Gastrointestinal disorders) | 6 | 10
CROHN'S DISEASE (Gastrointestinal disorders) | 1 | 0
DENTAL CARIES (Gastrointestinal disorders) | 3 | 0
DIARRHOEA (Gastrointestinal disorders) | 18 | 20
DIVERTICULAR PERFORATION (Gastrointestinal disorders) | 0 | 1
DIVERTICULITIS INTESTINAL HAEMORRHAGIC (Gastrointestinal disorders) | 0 | 2
DIVERTICULUM (Gastrointestinal disorders) | 2 | 4
DIVERTICULUM INTESTINAL (Gastrointestinal disorders) | 2 | 7
DIVERTICULUM INTESTINAL HAEMORRHAGIC (Gastrointestinal disorders) | 1 | 0
DUODENAL PERFORATION (Gastrointestinal disorders) | 1 | 0
DUODENAL ULCER (Gastrointestinal disorders) | 0 | 1
DUODENAL ULCER PERFORATION (Gastrointestinal disorders) | 1 | 0
DUODENITIS (Gastrointestinal disorders) | 0 | 1
DYSPEPSIA (Gastrointestinal disorders) | 11 | 11
DYSPHAGIA (Gastrointestinal disorders) | 5 | 5
ENTERITIS (Gastrointestinal disorders) | 1 | 1
ENTEROCOLITIS HAEMORRHAGIC (Gastrointestinal disorders) | 1 | 1
ENTEROVESICAL FISTULA (Gastrointestinal disorders) | 0 | 1
EPIGASTRIC DISCOMFORT (Gastrointestinal disorders) | 0 | 1
EROSIVE OESOPHAGITIS (Gastrointestinal disorders) | 0 | 1
ERUCTATION (Gastrointestinal disorders) | 0 | 1
FAECALOMA (Gastrointestinal disorders) | 1 | 1
FAECES DISCOLOURED (Gastrointestinal disorders) | 2 | 1
FLATULENCE (Gastrointestinal disorders) | 0 | 2
FOOD POISONING (Gastrointestinal disorders) | 0 | 1
GASTRIC DISORDER (Gastrointestinal disorders) | 0 | 2
GASTRIC POLYPS (Gastrointestinal disorders) | 1 | 0
GASTRIC ULCER (Gastrointestinal disorders) | 1 | 2
GASTRIC ULCER HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1
GASTRITIS (Gastrointestinal disorders) | 7 | 10
GASTRITIS EROSIVE (Gastrointestinal disorders) | 1 | 2
GASTRITIS HAEMORRHAGIC (Gastrointestinal disorders) | 1 | 0
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 17 | 13
GASTROINTESTINAL MOTILITY DISORDER (Gastrointestinal disorders) | 0 | 1
GASTROINTESTINAL MUCOSAL DISORDER (Gastrointestinal disorders) | 0 | 1
GASTROINTESTINAL MUCOSAL EXFOLIATION (Gastrointestinal disorders) | 1 | 0
GASTROINTESTINAL ULCER HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 19 | 16
GINGIVAL BLEEDING (Gastrointestinal disorders) | 2 | 2
GINGIVAL DISORDER (Gastrointestinal disorders) | 1 | 0
HAEMATEMESIS (Gastrointestinal disorders) | 0 | 2
HAEMATOCHEZIA (Gastrointestinal disorders) | 6 | 4
HAEMORRHOIDAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 4
HAEMORRHOIDS (Gastrointestinal disorders) | 1 | 4
HIATUS HERNIA (Gastrointestinal disorders) | 5 | 3
ILEUS (Gastrointestinal disorders) | 1 | 2
IMPAIRED GASTRIC EMPTYING (Gastrointestinal disorders) | 1 | 1
INGUINAL HERNIA (Gastrointestinal disorders) | 14 | 8
INGUINAL HERNIA, OBSTRUCTIVE (Gastrointestinal disorders) | 1 | 0
INTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1
INTESTINAL ISCHAEMIA (Gastrointestinal disorders) | 1 | 1
INTESTINAL MASS (Gastrointestinal disorders) | 1 | 0
IRRITABLE BOWEL SYNDROME (Gastrointestinal disorders) | 1 | 0
LARGE INTESTINE PERFORATION (Gastrointestinal disorders) | 0 | 1
LIP HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0
LIP SWELLING (Gastrointestinal disorders) | 0 | 1
LOWER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 3 | 1
MALLORY-WEISS SYNDROME (Gastrointestinal disorders) | 0 | 1
MELAENA (Gastrointestinal disorders) | 3 | 3
MELANOSIS COLI (Gastrointestinal disorders) | 0 | 1
MESENTERIC HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0
MOUTH HAEMORRHAGE (Gastrointestinal disorders) | 1 | 1
MOUTH ULCERATION (Gastrointestinal disorders) | 1 | 0
NAUSEA (Gastrointestinal disorders) | 34 | 35
OBSTRUCTION GASTRIC (Gastrointestinal disorders) | 0 | 1
ODYNOPHAGIA (Gastrointestinal disorders) | 1 | 1
OESOPHAGEAL HYPOMOTILITY (Gastrointestinal disorders) | 1 | 0
OESOPHAGEAL SPASM (Gastrointestinal disorders) | 0 | 1
OESOPHAGEAL STENOSIS (Gastrointestinal disorders) | 1 | 0
OESOPHAGITIS (Gastrointestinal disorders) | 0 | 2
ORAL MUCOSAL DISCOLOURATION (Gastrointestinal disorders) | 0 | 1
PANCREATIC MASS (Gastrointestinal disorders) | 1 | 0
PANCREATITIS (Gastrointestinal disorders) | 1 | 6
PANCREATITIS ACUTE (Gastrointestinal disorders) | 1 | 5
PANCREATITIS CHRONIC (Gastrointestinal disorders) | 0 | 2
PARAESTHESIA ORAL (Gastrointestinal disorders) | 1 | 1
POLYP COLORECTAL (Gastrointestinal disorders) | 0 | 1
PROCTALGIA (Gastrointestinal disorders) | 0 | 1
PROCTITIS (Gastrointestinal disorders) | 1 | 1
PROCTITIS ULCERATIVE (Gastrointestinal disorders) | 1 | 1
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 8 | 11
RECTAL POLYP (Gastrointestinal disorders) | 1 | 2
RETROPERITONEAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 1
SALIVARY GLAND MASS (Gastrointestinal disorders) | 1 | 0
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 10 | 6
SPIGELIAN HERNIA (Gastrointestinal disorders) | 1 | 2
STOMACH MASS (Gastrointestinal disorders) | 1 | 0
STOMATITIS (Gastrointestinal disorders) | 1 | 1
SWOLLEN TONGUE (Gastrointestinal disorders) | 1 | 0
TOOTH DISORDER (Gastrointestinal disorders) | 0 | 2
TOOTH LOSS (Gastrointestinal disorders) | 1 | 0
TOOTHACHE (Gastrointestinal disorders) | 2 | 2
UMBILICAL HERNIA (Gastrointestinal disorders) | 3 | 4
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 7 | 2
VOLVULUS (Gastrointestinal disorders) | 1 | 0
VOMITING (Gastrointestinal disorders) | 5 | 6
ADVERSE DRUG REACTION (General disorders) | 78 | 75
ASTHENIA (General disorders) | 27 | 21
AXILLARY PAIN (General disorders) | 0 | 1
CARDIAC COMPLICATION ASSOCIATED WITH DEVICE (General disorders) | 3 | 0
CARDIAC DEATH (General disorders) | 1 | 0
CATHETER SITE HAEMATOMA (General disorders) | 26 | 32
CATHETER SITE HAEMORRHAGE (General disorders) | 8 | 16
CATHETER SITE NECROSIS (General disorders) | 0 | 1
CATHETER SITE PAIN (General disorders) | 9 | 21
CATHETER SITE RASH (General disorders) | 1 | 0
CATHETER SITE RELATED REACTION (General disorders) | 0 | 3
CATHETER SITE SWELLING (General disorders) | 2 | 1
CHEST DISCOMFORT (General disorders) | 60 | 65
CHEST PAIN (General disorders) | 105 | 110
CHILLS (General disorders) | 0 | 1
COMPLICATION OF DEVICE REMOVAL (General disorders) | 1 | 0
CYST (General disorders) | 0 | 6
DEATH (General disorders) | 7 | 11
DEVICE BREAKAGE (General disorders) | 1 | 1
DEVICE FAILURE (General disorders) | 0 | 2
DEVICE ISSUE (General disorders) | 1 | 1
DEVICE MALFUNCTION (General disorders) | 1 | 0
DEVICE MATERIAL ISSUE (General disorders) | 0 | 1
DEVICE OCCLUSION (General disorders) | 1 | 1
DISEASE PROGRESSION (General disorders) | 0 | 1
DRUG INTOLERANCE (General disorders) | 2 | 2
EARLY SATIETY (General disorders) | 0 | 1
EXERCISE TOLERANCE DECREASED (General disorders) | 1 | 0
FACIAL PAIN (General disorders) | 0 | 1
FATIGUE (General disorders) | 45 | 43
FEELING COLD (General disorders) | 1 | 0
FEELING HOT (General disorders) | 0 | 1
GAIT DISTURBANCE (General disorders) | 1 | 1
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 1 | 2
GENERALISED OEDEMA (General disorders) | 1 | 1
GRANULOMA (General disorders) | 2 | 0
HERNIA (General disorders) | 1 | 2
HYPERTHERMIA (General disorders) | 1 | 0
IMPAIRED HEALING (General disorders) | 1 | 2
INFLAMMATION (General disorders) | 1 | 0
INFLUENZA LIKE ILLNESS (General disorders) | 1 | 0
INFUSION SITE PAIN (General disorders) | 0 | 1
LOCAL SWELLING (General disorders) | 0 | 1
MALAISE (General disorders) | 9 | 10
MEDICAL DEVICE COMPLICATION (General disorders) | 0 | 1
MEDICAL DEVICE PAIN (General disorders) | 1 | 0
MEDICAL DEVICE SITE REACTION (General disorders) | 1 | 0
METAPLASIA (General disorders) | 0 | 1
MULTI-ORGAN FAILURE (General disorders) | 0 | 1
NON-CARDIAC CHEST PAIN (General disorders) | 230 | 274
OEDEMA (General disorders) | 1 | 3
OEDEMA PERIPHERAL (General disorders) | 27 | 22
PACEMAKER GENERATED ARRHYTHMIA (General disorders) | 1 | 0
PAIN (General disorders) | 2 | 9
PATIENT-DEVICE INCOMPATIBILITY (General disorders) | 1 | 0
PYREXIA (General disorders) | 9 | 3
SENSATION OF FOREIGN BODY (General disorders) | 1 | 1
SPINAL PAIN (General disorders) | 1 | 0
STENT-GRAFT ENDOLEAK (General disorders) | 0 | 1
SUDDEN CARDIAC DEATH (General disorders) | 0 | 1
SWELLING (General disorders) | 0 | 1
SYSTEMIC INFLAMMATORY RESPONSE SYNDROME (General disorders) | 0 | 2
THROMBOSIS IN DEVICE (General disorders) | 13 | 13
ULCER (General disorders) | 0 | 1
UNEVALUABLE EVENT (General disorders) | 1 | 0
VESSEL PUNCTURE SITE HAEMATOMA (General disorders) | 1 | 0
VESSEL PUNCTURE SITE THROMBOSIS (General disorders) | 0 | 1
ACUTE HEPATIC FAILURE (Hepatobiliary disorders) | 2 | 0
BILE DUCT OBSTRUCTION (Hepatobiliary disorders) | 1 | 0
BILE DUCT STONE (Hepatobiliary disorders) | 3 | 4
BILIARY COLIC (Hepatobiliary disorders) | 0 | 2
BILIARY DILATATION (Hepatobiliary disorders) | 0 | 1
BILIARY DYSKINESIA (Hepatobiliary disorders) | 1 | 0
CHOLANGITIS (Hepatobiliary disorders) | 2 | 0
CHOLANGITIS ACUTE (Hepatobiliary disorders) | 1 | 1
CHOLECYSTITIS (Hepatobiliary disorders) | 4 | 3
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 3 | 3
CHOLECYSTITIS CHRONIC (Hepatobiliary disorders) | 0 | 2
CHOLELITHIASIS (Hepatobiliary disorders) | 10 | 6
CIRRHOSIS ALCOHOLIC (Hepatobiliary disorders) | 1 | 0
GALLBLADDER DISORDER (Hepatobiliary disorders) | 1 | 2
GRANULOMATOUS LIVER DISEASE (Hepatobiliary disorders) | 0 | 1
HEPATIC CIRRHOSIS (Hepatobiliary disorders) | 1 | 1
HEPATIC CYST (Hepatobiliary disorders) | 1 | 2
HEPATIC FAILURE (Hepatobiliary disorders) | 0 | 1
HEPATIC FUNCTION ABNORMAL (Hepatobiliary disorders) | 2 | 0
HEPATIC LESION (Hepatobiliary disorders) | 0 | 1
HEPATIC PAIN (Hepatobiliary disorders) | 0 | 1
HEPATIC STEATOSIS (Hepatobiliary disorders) | 2 | 1
HEPATORENAL FAILURE (Hepatobiliary disorders) | 1 | 0
ISCHAEMIC HEPATITIS (Hepatobiliary disorders) | 1 | 0
JAUNDICE (Hepatobiliary disorders) | 2 | 0
JAUNDICE CHOLESTATIC (Hepatobiliary disorders) | 1 | 0
NON-ALCOHOLIC STEATOHEPATITIS (Hepatobiliary disorders) | 0 | 1
ALLERGY TO ARTHROPOD BITE (Immune system disorders) | 0 | 1
ALLERGY TO ARTHROPOD STING (Immune system disorders) | 1 | 1
AMYLOIDOSIS (Immune system disorders) | 0 | 1
ANAPHYLACTIC REACTION (Immune system disorders) | 1 | 0
CONTRAST MEDIA ALLERGY (Immune system disorders) | 1 | 1
DRUG HYPERSENSITIVITY (Immune system disorders) | 6 | 2
FOOD ALLERGY (Immune system disorders) | 0 | 1
HYPERSENSITIVITY (Immune system disorders) | 0 | 1
SARCOIDOSIS (Immune system disorders) | 0 | 1
SEASONAL ALLERGY (Immune system disorders) | 2 | 1
ABDOMINAL ABSCESS (Infections and infestations) | 0 | 2
ABDOMINAL SEPSIS (Infections and infestations) | 1 | 0
ABSCESS LIMB (Infections and infestations) | 2 | 3
ABSCESS NECK (Infections and infestations) | 1 | 0
ABSCESS OF SALIVARY GLAND (Infections and infestations) | 1 | 0
ABSCESS ORAL (Infections and infestations) | 0 | 1
ACARODERMATITIS (Infections and infestations) | 1 | 1
ACUTE SINUSITIS (Infections and infestations) | 5 | 5
APPENDICITIS (Infections and infestations) | 4 | 4
ARTERIOVENOUS GRAFT SITE INFECTION (Infections and infestations) | 0 | 1
ARTHRITIS INFECTIVE (Infections and infestations) | 1 | 0
BACTERAEMIA (Infections and infestations) | 1 | 1
BACTERIAL INFECTION (Infections and infestations) | 1 | 0
BACTERIAL SEPSIS (Infections and infestations) | 0 | 1
BODY TINEA (Infections and infestations) | 1 | 0
BRONCHIOLITIS (Infections and infestations) | 1 | 1
BRONCHITIS (Infections and infestations) | 23 | 20
BRONCHITIS VIRAL (Infections and infestations) | 0 | 3
BRONCHOPNEUMONIA (Infections and infestations) | 0 | 1
BURSITIS INFECTIVE (Infections and infestations) | 1 | 1
CAMPYLOBACTER INFECTION (Infections and infestations) | 0 | 1
CATHETER SITE ABSCESS (Infections and infestations) | 0 | 1
CATHETER SITE CELLULITIS (Infections and infestations) | 1 | 1
CELLULITIS (Infections and infestations) | 15 | 14
CELLULITIS OF MALE EXTERNAL GENITAL ORGAN (Infections and infestations) | 1 | 0
CHOLECYSTITIS INFECTIVE (Infections and infestations) | 0 | 2
CHRONIC SINUSITIS (Infections and infestations) | 0 | 2
CLOSTRIDIAL INFECTION (Infections and infestations) | 2 | 3
CLOSTRIDIUM COLITIS (Infections and infestations) | 0 | 1
CLOSTRIDIUM DIFFICILE COLITIS (Infections and infestations) | 1 | 0
CONJUNCTIVITIS BACTERIAL (Infections and infestations) | 1 | 0
CORONA VIRUS INFECTION (Infections and infestations) | 14 | 4
CYSTITIS (Infections and infestations) | 2 | 3
DEVICE RELATED INFECTION (Infections and infestations) | 1 | 1
DIABETIC FOOT INFECTION (Infections and infestations) | 0 | 1
DIVERTICULITIS (Infections and infestations) | 18 | 14
EAR INFECTION (Infections and infestations) | 1 | 2
EMPYEMA (Infections and infestations) | 0 | 1
ENDOCARDITIS (Infections and infestations) | 1 | 0
ENDOMETRITIS (Infections and infestations) | 1 | 0
ENTEROCOCCAL BACTERAEMIA (Infections and infestations) | 0 | 1
ENTEROCOLITIS INFECTIOUS (Infections and infestations) | 1 | 1
EPIDEMIC POLYARTHRITIS (Infections and infestations) | 1 | 0
ESCHERICHIA BACTERAEMIA (Infections and infestations) | 1 | 0
ESCHERICHIA INFECTION (Infections and infestations) | 1 | 0
ESCHERICHIA SEPSIS (Infections and infestations) | 0 | 1
ESCHERICHIA URINARY TRACT INFECTION (Infections and infestations) | 1 | 2
EXTRADURAL ABSCESS (Infections and infestations) | 0 | 1
FURUNCLE (Infections and infestations) | 0 | 1
GANGRENE (Infections and infestations) | 3 | 1
GASTRIC INFECTION (Infections and infestations) | 0 | 1
GASTRITIS VIRAL (Infections and infestations) | 1 | 0
GASTROENTERITIS (Infections and infestations) | 7 | 8
GASTROENTERITIS VIRAL (Infections and infestations) | 4 | 2
GASTROINTESTINAL INFECTION (Infections and infestations) | 1 | 0
GENITAL HERPES (Infections and infestations) | 1 | 1
HELICOBACTER GASTRITIS (Infections and infestations) | 1 | 0
HELICOBACTER INFECTION (Infections and infestations) | 1 | 2
HEPATITIS C (Infections and infestations) | 1 | 0
HERPES SIMPLEX (Infections and infestations) | 0 | 1
HERPES ZOSTER (Infections and infestations) | 6 | 8
HERPES ZOSTER OTICUS (Infections and infestations) | 1 | 0
IMPETIGO (Infections and infestations) | 0 | 1
IMPLANT SITE INFECTION (Infections and infestations) | 0 | 1
INCISION SITE INFECTION (Infections and infestations) | 1 | 0
INFECTED BITES (Infections and infestations) | 2 | 0
INFECTED CYST (Infections and infestations) | 0 | 1
INFECTED DERMAL CYST (Infections and infestations) | 1 | 0
INFECTED SKIN ULCER (Infections and infestations) | 0 | 1
INFECTIOUS PLEURAL EFFUSION (Infections and infestations) | 1 | 0
INFLUENZA (Infections and infestations) | 13 | 20
INTERTRIGO CANDIDA (Infections and infestations) | 0 | 1
KIDNEY INFECTION (Infections and infestations) | 0 | 1
KLEBSIELLA BACTERAEMIA (Infections and infestations) | 0 | 1
KLEBSIELLA SEPSIS (Infections and infestations) | 0 | 1
LABYRINTHITIS (Infections and infestations) | 0 | 1
LARYNGITIS (Infections and infestations) | 1 | 0
LIVER ABSCESS (Infections and infestations) | 2 | 1
LOBAR PNEUMONIA (Infections and infestations) | 6 | 5
LOCALISED INFECTION (Infections and infestations) | 2 | 0
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 3 | 4
LUNG INFECTION (Infections and infestations) | 0 | 1
LUNG INFECTION PSEUDOMONAL (Infections and infestations) | 0 | 1
LYME DISEASE (Infections and infestations) | 1 | 1
LYMPH GLAND INFECTION (Infections and infestations) | 1 | 0
MUSCLE ABSCESS (Infections and infestations) | 1 | 0
MYRINGITIS BULLOUS (Infections and infestations) | 1 | 0
NASOPHARYNGITIS (Infections and infestations) | 9 | 12
NECROTISING FASCIITIS (Infections and infestations) | 0 | 1
OESOPHAGEAL CANDIDIASIS (Infections and infestations) | 0 | 2
ORAL CANDIDIASIS (Infections and infestations) | 1 | 0
ORAL FUNGAL INFECTION (Infections and infestations) | 0 | 1
ORCHITIS (Infections and infestations) | 2 | 0
OSTEOMYELITIS (Infections and infestations) | 0 | 5
OSTEOMYELITIS CHRONIC (Infections and infestations) | 0 | 1
OTITIS EXTERNA (Infections and infestations) | 1 | 0
OTITIS MEDIA (Infections and infestations) | 1 | 1
OTITIS MEDIA ACUTE (Infections and infestations) | 1 | 0
OTITIS MEDIA CHRONIC (Infections and infestations) | 1 | 0
PELVIC INFECTION (Infections and infestations) | 1 | 0
PERIUMBILICAL ABSCESS (Infections and infestations) | 0 | 1
PHARYNGEAL ABSCESS (Infections and infestations) | 0 | 1
PHARYNGITIS (Infections and infestations) | 0 | 3
PHARYNGITIS BACTERIAL (Infections and infestations) | 1 | 0
PHARYNGITIS STREPTOCOCCAL (Infections and infestations) | 0 | 3
PLEURAL INFECTION (Infections and infestations) | 1 | 0
PNEUMONIA (Infections and infestations) | 42 | 42
PNEUMONIA ESCHERICHIA (Infections and infestations) | 1 | 0
PNEUMONIA KLEBSIELLA (Infections and infestations) | 0 | 1
PNEUMONIA STREPTOCOCCAL (Infections and infestations) | 0 | 1
PNEUMONIA VIRAL (Infections and infestations) | 1 | 4
POST PROCEDURAL CELLULITIS (Infections and infestations) | 0 | 1
POSTOPERATIVE ABSCESS (Infections and infestations) | 1 | 0
POSTOPERATIVE WOUND INFECTION (Infections and infestations) | 2 | 0
PYELONEPHRITIS (Infections and infestations) | 2 | 3
PYELONEPHRITIS ACUTE (Infections and infestations) | 1 | 1
RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 | 2
RESPIRATORY TRACT INFECTION VIRAL (Infections and infestations) | 1 | 1
RHINOVIRUS INFECTION (Infections and infestations) | 1 | 0
SCROTAL ABSCESS (Infections and infestations) | 3 | 0
SEPSIS (Infections and infestations) | 20 | 14
SEPSIS SYNDROME (Infections and infestations) | 0 | 1
SEPTIC ENCEPHALOPATHY (Infections and infestations) | 1 | 0
SEPTIC SHOCK (Infections and infestations) | 2 | 4
SIALOADENITIS (Infections and infestations) | 0 | 1
SINOBRONCHITIS (Infections and infestations) | 0 | 1
SINUSITIS (Infections and infestations) | 11 | 10
SINUSITIS BACTERIAL (Infections and infestations) | 2 | 0
SKIN INFECTION (Infections and infestations) | 0 | 1
STAPHYLOCOCCAL ABSCESS (Infections and infestations) | 0 | 1
STAPHYLOCOCCAL BACTERAEMIA (Infections and infestations) | 1 | 1
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 1 | 1
STAPHYLOCOCCAL SEPSIS (Infections and infestations) | 1 | 1
SUBCUTANEOUS ABSCESS (Infections and infestations) | 1 | 2
TESTICULAR ABSCESS (Infections and infestations) | 1 | 0
TINEA PEDIS (Infections and infestations) | 1 | 0
TOOTH ABSCESS (Infections and infestations) | 3 | 6
TOOTH INFECTION (Infections and infestations) | 3 | 5
TRICHOMONIASIS (Infections and infestations) | 1 | 0
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 20 | 24
UPPER RESPIRATORY TRACT INFECTION BACTERIAL (Infections and infestations) | 0 | 1
URETHRITIS (Infections and infestations) | 1 | 0
URINARY TRACT INFECTION (Infections and infestations) | 24 | 33
URINARY TRACT INFECTION BACTERIAL (Infections and infestations) | 1 | 0
UROSEPSIS (Infections and infestations) | 5 | 1
VAGINITIS BACTERIAL (Infections and infestations) | 1 | 1
VESTIBULAR NEURONITIS (Infections and infestations) | 1 | 0
VIRAL INFECTION (Infections and infestations) | 3 | 1
VIRAL LABYRINTHITIS (Infections and infestations) | 1 | 0
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 1
WEST NILE VIRAL INFECTION (Infections and infestations) | 1 | 0
WOUND INFECTION (Infections and infestations) | 2 | 3
WOUND INFECTION BACTERIAL (Infections and infestations) | 1 | 0
WOUND INFECTION STAPHYLOCOCCAL (Infections and infestations) | 0 | 1
ACCIDENTAL OVERDOSE (Injury, poisoning and procedural complications) | 1 | 2
ACETABULUM FRACTURE (Injury, poisoning and procedural complications) | 2 | 0
ADRENAL GLAND INJURY (Injury, poisoning and procedural complications) | 0 | 1
ALCOHOL POISONING (Injury, poisoning and procedural complications) | 1 | 1
ANAEMIA POSTOPERATIVE (Injury, poisoning and procedural complications) | 3 | 2
ANASTOMOTIC LEAK (Injury, poisoning and procedural complications) | 0 | 1
ANASTOMOTIC ULCER HAEMORRHAGE (Injury, poisoning and procedural complications) | 1 | 0
ANIMAL BITE (Injury, poisoning and procedural complications) | 0 | 4
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 3 | 10
ARTERIAL INJURY (Injury, poisoning and procedural complications) | 0 | 1
ARTHROPOD BITE (Injury, poisoning and procedural complications) | 2 | 1
ARTHROPOD STING (Injury, poisoning and procedural complications) | 1 | 1
ASBESTOSIS (Injury, poisoning and procedural complications) | 1 | 0
AXILLARY NERVE INJURY (Injury, poisoning and procedural complications) | 1 | 0
BACK INJURY (Injury, poisoning and procedural complications) | 1 | 1
CARDIAC PROCEDURE COMPLICATION (Injury, poisoning and procedural complications) | 7 | 3
CATHETER SITE HAEMATOMA (Injury, poisoning and procedural complications) | 3 | 6
CERVICAL VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 2 | 2
COMMINUTED FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
CONCUSSION (Injury, poisoning and procedural complications) | 2 | 0
CONFUSION POSTOPERATIVE (Injury, poisoning and procedural complications) | 2 | 0
CONTRAST MEDIA ALLERGY (Injury, poisoning and procedural complications) | 1 | 0
CONTUSION (Injury, poisoning and procedural complications) | 16 | 22
CORNEAL ABRASION (Injury, poisoning and procedural complications) | 1 | 0
CORONARY ARTERY REOCCLUSION (Injury, poisoning and procedural complications) | 1 | 0
CORONARY ARTERY RESTENOSIS (Injury, poisoning and procedural complications) | 30 | 21
CRANIOCEREBRAL INJURY (Injury, poisoning and procedural complications) | 3 | 2
CYSTITIS RADIATION (Injury, poisoning and procedural complications) | 0 | 2
DEPRESSION POSTOPERATIVE (Injury, poisoning and procedural complications) | 0 | 1
DRUG ADMINISTRATION ERROR (Injury, poisoning and procedural complications) | 0 | 1
EAR INJURY (Injury, poisoning and procedural complications) | 1 | 0
EPICONDYLITIS (Injury, poisoning and procedural complications) | 0 | 1
EXCORIATION (Injury, poisoning and procedural complications) | 0 | 2
EXPOSURE TO TOXIC AGENT (Injury, poisoning and procedural complications) | 0 | 1
EYE PENETRATION (Injury, poisoning and procedural complications) | 0 | 1
FACIAL BONES FRACTURE (Injury, poisoning and procedural complications) | 2 | 0
FALL (Injury, poisoning and procedural complications) | 17 | 21
FEMORAL NECK FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 3 | 1
FIBULA FRACTURE (Injury, poisoning and procedural complications) | 1 | 2
FOOT FRACTURE (Injury, poisoning and procedural complications) | 2 | 6
FOREARM FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
FOREIGN BODY IN EYE (Injury, poisoning and procedural complications) | 1 | 0
FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
GASTROINTESTINAL DISORDER POSTOPERATIVE (Injury, poisoning and procedural complications) | 0 | 1
GASTROINTESTINAL STOMA COMPLICATION (Injury, poisoning and procedural complications) | 1 | 0
HAEMATURIA TRAUMATIC (Injury, poisoning and procedural complications) | 0 | 1
HAND FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
HEAD INJURY (Injury, poisoning and procedural complications) | 1 | 1
HEAT EXHAUSTION (Injury, poisoning and procedural complications) | 1 | 0
HEAT STROKE (Injury, poisoning and procedural complications) | 0 | 1
HIP FRACTURE (Injury, poisoning and procedural complications) | 2 | 2
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 4 | 1
IN-STENT ARTERIAL RESTENOSIS (Injury, poisoning and procedural complications) | 2 | 1
IN-STENT CORONARY ARTERY RESTENOSIS (Injury, poisoning and procedural complications) | 8 | 19
INCISION SITE PAIN (Injury, poisoning and procedural complications) | 1 | 1
INCISIONAL HERNIA (Injury, poisoning and procedural complications) | 0 | 1
INCORRECT DOSE ADMINISTERED (Injury, poisoning and procedural complications) | 2 | 0
INJURY (Injury, poisoning and procedural complications) | 3 | 1
INTENTIONAL OVERDOSE (Injury, poisoning and procedural complications) | 1 | 0
JOINT DISLOCATION (Injury, poisoning and procedural complications) | 0 | 3
JOINT INJURY (Injury, poisoning and procedural complications) | 3 | 5
LACERATION (Injury, poisoning and procedural complications) | 11 | 11
LIGAMENT RUPTURE (Injury, poisoning and procedural complications) | 2 | 0
LIGAMENT SPRAIN (Injury, poisoning and procedural complications) | 6 | 6
LIMB INJURY (Injury, poisoning and procedural complications) | 3 | 4
LUMBAR VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 2 | 2
MENISCUS LESION (Injury, poisoning and procedural complications) | 1 | 2
MOUTH INJURY (Injury, poisoning and procedural complications) | 0 | 2
MULTIPLE FRACTURES (Injury, poisoning and procedural complications) | 1 | 0
MULTIPLE INJURIES (Injury, poisoning and procedural complications) | 1 | 0
MUSCLE RUPTURE (Injury, poisoning and procedural complications) | 2 | 0
MUSCLE STRAIN (Injury, poisoning and procedural complications) | 2 | 5
OVERDOSE (Injury, poisoning and procedural complications) | 1 | 1
PATELLA FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
PELVIC FRACTURE (Injury, poisoning and procedural complications) | 0 | 3
PELVIC ORGAN INJURY (Injury, poisoning and procedural complications) | 0 | 1
PERIPROSTHETIC FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
PLAQUE SHIFT (Injury, poisoning and procedural complications) | 3 | 4
POISONING (Injury, poisoning and procedural complications) | 0 | 1
POISONING DELIBERATE (Injury, poisoning and procedural complications) | 0 | 1
POST LAMINECTOMY SYNDROME (Injury, poisoning and procedural complications) | 1 | 0
POST PROCEDURAL BILE LEAK (Injury, poisoning and procedural complications) | 1 | 1
POST PROCEDURAL COMPLICATION (Injury, poisoning and procedural complications) | 2 | 1
POST PROCEDURAL DISCOMFORT (Injury, poisoning and procedural complications) | 1 | 1
POST PROCEDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 1 | 0
POST PROCEDURAL HAEMATURIA (Injury, poisoning and procedural complications) | 1 | 0
POST PROCEDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 1 | 0
POST PROCEDURAL MYOCARDIAL INFARCTION (Injury, poisoning and procedural complications) | 20 | 13
POST PROCEDURAL OEDEMA (Injury, poisoning and procedural complications) | 1 | 0
POST-TRAUMATIC PAIN (Injury, poisoning and procedural complications) | 8 | 7
POSTOPERATIVE FEVER (Injury, poisoning and procedural complications) | 2 | 1
POSTOPERATIVE HERNIA (Injury, poisoning and procedural complications) | 0 | 1
POSTOPERATIVE ILEUS (Injury, poisoning and procedural complications) | 1 | 0
POSTOPERATIVE RESPIRATORY DISTRESS (Injury, poisoning and procedural complications) | 1 | 1
PROCEDURAL COMPLICATION (Injury, poisoning and procedural complications) | 2 | 0
PROCEDURAL DIZZINESS (Injury, poisoning and procedural complications) | 2 | 0
PROCEDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 2 | 0
PROCEDURAL HEADACHE (Injury, poisoning and procedural complications) | 3 | 4
PROCEDURAL HYPERTENSION (Injury, poisoning and procedural complications) | 5 | 5
PROCEDURAL HYPOTENSION (Injury, poisoning and procedural complications) | 10 | 2
PROCEDURAL NAUSEA (Injury, poisoning and procedural complications) | 8 | 6
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 16 | 15
PROCEDURAL VOMITING (Injury, poisoning and procedural complications) | 1 | 3
RADIUS FRACTURE (Injury, poisoning and procedural complications) | 1 | 1
RIB FRACTURE (Injury, poisoning and procedural complications) | 7 | 3
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 6 | 6
SEROMA (Injury, poisoning and procedural complications) | 0 | 1
SKELETAL INJURY (Injury, poisoning and procedural complications) | 0 | 1
SKULL FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
SPINAL COLUMN INJURY (Injury, poisoning and procedural complications) | 1 | 0
SPINAL COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 5 | 1
SPINAL FRACTURE (Injury, poisoning and procedural complications) | 2 | 0
STAB WOUND (Injury, poisoning and procedural complications) | 0 | 1
SUBCUTANEOUS HAEMATOMA (Injury, poisoning and procedural complications) | 0 | 1
SUBDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 1 | 3
SUBDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 1 | 0
SUTURE RUPTURE (Injury, poisoning and procedural complications) | 0 | 1
TENDON RUPTURE (Injury, poisoning and procedural complications) | 2 | 3
THERMAL BURN (Injury, poisoning and procedural complications) | 3 | 1
THORACIC VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
TOOTH FRACTURE (Injury, poisoning and procedural complications) | 1 | 3
TRAUMATIC ARTHRITIS (Injury, poisoning and procedural complications) | 1 | 1
TRAUMATIC HAEMATOMA (Injury, poisoning and procedural complications) | 1 | 2
TRAUMATIC HAEMORRHAGE (Injury, poisoning and procedural complications) | 2 | 0
TRAUMATIC INTRACRANIAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 1 | 0
TRAUMATIC LUNG INJURY (Injury, poisoning and procedural complications) | 0 | 1
ULNA FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
UPPER LIMB FRACTURE (Injury, poisoning and procedural complications) | 1 | 3
URINARY RETENTION POSTOPERATIVE (Injury, poisoning and procedural complications) | 3 | 1
VASCULAR GRAFT COMPLICATION (Injury, poisoning and procedural complications) | 0 | 1
VASCULAR GRAFT OCCLUSION (Injury, poisoning and procedural complications) | 0 | 2
VASCULAR PSEUDOANEURYSM (Injury, poisoning and procedural complications) | 7 | 8
WOUND COMPLICATION (Injury, poisoning and procedural complications) | 1 | 1
WOUND DEHISCENCE (Injury, poisoning and procedural complications) | 1 | 1
WOUND HAEMORRHAGE (Injury, poisoning and procedural complications) | 0 | 1
WRIST FRACTURE (Injury, poisoning and procedural complications) | 1 | 5
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 | 1
ANGIOGRAM (Investigations) | 1 | 0
ARTERIAL BRUIT (Investigations) | 0 | 1
ARTERIOGRAM CORONARY (Investigations) | 2 | 0
ARTERIOGRAM CORONARY ABNORMAL (Investigations) | 1 | 4
BLOOD CHOLESTEROL DECREASED (Investigations) | 0 | 1
BLOOD CHOLESTEROL INCREASED (Investigations) | 0 | 1
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 18 | 20
BLOOD CREATINE PHOSPHOKINASE MB ABNORMAL (Investigations) | 1 | 0
BLOOD CREATINE PHOSPHOKINASE MB DECREASED (Investigations) | 0 | 1
BLOOD CREATINE PHOSPHOKINASE MB INCREASED (Investigations) | 68 | 59
BLOOD CREATININE INCREASED (Investigations) | 2 | 1
BLOOD GLUCOSE DECREASED (Investigations) | 0 | 1
BLOOD GLUCOSE INCREASED (Investigations) | 4 | 4
BLOOD LACTIC ACID INCREASED (Investigations) | 0 | 1
BLOOD MAGNESIUM DECREASED (Investigations) | 1 | 0
BLOOD POTASSIUM DECREASED (Investigations) | 0 | 1
BLOOD PRESSURE DECREASED (Investigations) | 1 | 0
BLOOD PRESSURE INCREASED (Investigations) | 12 | 6
BLOOD PRESSURE SYSTOLIC DECREASED (Investigations) | 0 | 1
BLOOD PRESSURE SYSTOLIC INCREASED (Investigations) | 2 | 0
BLOOD TESTOSTERONE DECREASED (Investigations) | 0 | 1
BLOOD TRIGLYCERIDES INCREASED (Investigations) | 0 | 1
BLOOD URIC ACID INCREASED (Investigations) | 0 | 1
BLOOD URINE PRESENT (Investigations) | 1 | 1
BODY TEMPERATURE INCREASED (Investigations) | 1 | 0
CARDIAC ENZYMES INCREASED (Investigations) | 149 | 150
CARDIAC IMAGING PROCEDURE ABNORMAL (Investigations) | 1 | 0
CARDIAC MURMUR (Investigations) | 0 | 1
CARDIAC STRESS TEST ABNORMAL (Investigations) | 3 | 5
CAROTID BRUIT (Investigations) | 0 | 1
CATHETERISATION CARDIAC (Investigations) | 1 | 0
COMPUTERISED TOMOGRAM THORAX ABNORMAL (Investigations) | 1 | 0
CORONAVIRUS TEST POSITIVE (Investigations) | 1 | 1
EJECTION FRACTION DECREASED (Investigations) | 4 | 3
ELECTROCARDIOGRAM ABNORMAL (Investigations) | 2 | 1
ELECTROCARDIOGRAM ST SEGMENT ELEVATION (Investigations) | 2 | 1
FEMORAL BRUIT (Investigations) | 1 | 0
FIBRIN D DIMER INCREASED (Investigations) | 0 | 1
GLYCOSYLATED HAEMOGLOBIN INCREASED (Investigations) | 0 | 3
HAEMOGLOBIN DECREASED (Investigations) | 1 | 0
HEART RATE DECREASED (Investigations) | 0 | 1
HEART RATE INCREASED (Investigations) | 2 | 2
HEART RATE IRREGULAR (Investigations) | 0 | 2
HEPATIC ENZYME INCREASED (Investigations) | 2 | 3
INFLUENZA A VIRUS TEST POSITIVE (Investigations) | 0 | 1
LEFT VENTRICULAR END-DIASTOLIC PRESSURE INCREASED (Investigations) | 1 | 2
LIVER FUNCTION TEST ABNORMAL (Investigations) | 3 | 3
LIVER SCAN ABNORMAL (Investigations) | 0 | 1
LOW DENSITY LIPOPROTEIN INCREASED (Investigations) | 1 | 0
LYMPHOCYTE COUNT INCREASED (Investigations) | 1 | 0
MEAN CELL VOLUME ABNORMAL (Investigations) | 0 | 1
N-TERMINAL PROHORMONE BRAIN NATRIURETIC PEPTIDE INCREASED (Investigations) | 0 | 1
OCCULT BLOOD POSITIVE (Investigations) | 1 | 0
OESOPHAGOGASTRODUODENOSCOPY ABNORMAL (Investigations) | 0 | 1
OXYGEN SATURATION DECREASED (Investigations) | 1 | 0
PLATELET COUNT DECREASED (Investigations) | 1 | 0
POSITRON EMISSION TOMOGRAM ABNORMAL (Investigations) | 0 | 1
PROSTATIC SPECIFIC ANTIGEN INCREASED (Investigations) | 1 | 3
SCAN MYOCARDIAL PERFUSION ABNORMAL (Investigations) | 1 | 0
STRESS ECHOCARDIOGRAM ABNORMAL (Investigations) | 2 | 0
TRANSAMINASES INCREASED (Investigations) | 0 | 1
TROPONIN I INCREASED (Investigations) | 8 | 14
TROPONIN INCREASED (Investigations) | 109 | 86
TROPONIN T INCREASED (Investigations) | 14 | 12
ULTRASOUND THYROID ABNORMAL (Investigations) | 0 | 1
WEIGHT DECREASED (Investigations) | 1 | 2
WEIGHT INCREASED (Investigations) | 2 | 2
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 1 | 0
CARBOHYDRATE INTOLERANCE (Metabolism and nutrition disorders) | 1 | 0
DECREASED APPETITE (Metabolism and nutrition disorders) | 2 | 0
DEHYDRATION (Metabolism and nutrition disorders) | 8 | 7
DIABETES MELLITUS (Metabolism and nutrition disorders) | 8 | 10
DIABETES MELLITUS INADEQUATE CONTROL (Metabolism and nutrition disorders) | 5 | 2
DIABETIC KETOACIDOSIS (Metabolism and nutrition disorders) | 2 | 5
FAILURE TO THRIVE (Metabolism and nutrition disorders) | 2 | 0
FLUID OVERLOAD (Metabolism and nutrition disorders) | 1 | 1
GLUCOSE TOLERANCE IMPAIRED (Metabolism and nutrition disorders) | 2 | 1
GOUT (Metabolism and nutrition disorders) | 10 | 7
HYPERAMMONAEMIA (Metabolism and nutrition disorders) | 1 | 0
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 0 | 1
HYPERCHOLESTEROLAEMIA (Metabolism and nutrition disorders) | 2 | 0
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 7 | 4
HYPERKALAEMIA (Metabolism and nutrition disorders) | 5 | 0
HYPERLIPIDAEMIA (Metabolism and nutrition disorders) | 2 | 4
HYPERTRIGLYCERIDAEMIA (Metabolism and nutrition disorders) | 3 | 1
HYPERURICAEMIA (Metabolism and nutrition disorders) | 1 | 0
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 7 | 8
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 | 4
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 1 | 3
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 | 6
HYPOVITAMINOSIS (Metabolism and nutrition disorders) | 0 | 1
HYPOVOLAEMIA (Metabolism and nutrition disorders) | 2 | 0
IMPAIRED FASTING GLUCOSE (Metabolism and nutrition disorders) | 0 | 1
IRON DEFICIENCY (Metabolism and nutrition disorders) | 1 | 0
KETOACIDOSIS (Metabolism and nutrition disorders) | 1 | 0
LACTIC ACIDOSIS (Metabolism and nutrition disorders) | 1 | 1
MALNUTRITION (Metabolism and nutrition disorders) | 1 | 1
METABOLIC ACIDOSIS (Metabolism and nutrition disorders) | 1 | 1
METABOLIC SYNDROME (Metabolism and nutrition disorders) | 1 | 0
OBESITY (Metabolism and nutrition disorders) | 1 | 5
TYPE 1 DIABETES MELLITUS (Metabolism and nutrition disorders) | 0 | 1
TYPE 2 DIABETES MELLITUS (Metabolism and nutrition disorders) | 5 | 5
VITAMIN B12 DEFICIENCY (Metabolism and nutrition disorders) | 1 | 0
VITAMIN D DEFICIENCY (Metabolism and nutrition disorders) | 2 | 2
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 37 | 26
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 10 | 7
ARTHROPATHY (Musculoskeletal and connective tissue disorders) | 1 | 0
BACK PAIN (Musculoskeletal and connective tissue disorders) | 35 | 40
BONE PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1
BURSITIS (Musculoskeletal and connective tissue disorders) | 3 | 2
CERVICAL SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 2 | 4
CHONDROCALCINOSIS PYROPHOSPHATE (Musculoskeletal and connective tissue disorders) | 0 | 1
CHONDROMALACIA (Musculoskeletal and connective tissue disorders) | 2 | 0
CHONDROSIS (Musculoskeletal and connective tissue disorders) | 0 | 1
COSTOCHONDRITIS (Musculoskeletal and connective tissue disorders) | 1 | 4
DUPUYTREN'S CONTRACTURE (Musculoskeletal and connective tissue disorders) | 0 | 1
EXOSTOSIS (Musculoskeletal and connective tissue disorders) | 0 | 1
FACET JOINT SYNDROME (Musculoskeletal and connective tissue disorders) | 0 | 1
FEMOROACETABULAR IMPINGEMENT (Musculoskeletal and connective tissue disorders) | 1 | 0
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 2 | 2
FOOT DEFORMITY (Musculoskeletal and connective tissue disorders) | 2 | 1
GOUTY ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 | 0
GROIN PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0
INTERVERTEBRAL DISC COMPRESSION (Musculoskeletal and connective tissue disorders) | 1 | 0
INTERVERTEBRAL DISC DEGENERATION (Musculoskeletal and connective tissue disorders) | 3 | 3
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 6 | 5
JOINT EFFUSION (Musculoskeletal and connective tissue disorders) | 1 | 1
JOINT STIFFNESS (Musculoskeletal and connective tissue disorders) | 0 | 2
JOINT SWELLING (Musculoskeletal and connective tissue disorders) | 6 | 4
LIMB DISCOMFORT (Musculoskeletal and connective tissue disorders) | 2 | 1
LUMBAR SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 4 | 5
MONARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 1
MUSCLE ATROPHY (Musculoskeletal and connective tissue disorders) | 0 | 1
MUSCLE NECROSIS (Musculoskeletal and connective tissue disorders) | 0 | 1
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 11 | 11
MUSCLE TIGHTNESS (Musculoskeletal and connective tissue disorders) | 0 | 2
MUSCLE TWITCHING (Musculoskeletal and connective tissue disorders) | 1 | 0
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 8 | 6
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 12 | 17
MUSCULOSKELETAL DISCOMFORT (Musculoskeletal and connective tissue disorders) | 3 | 4
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 26 | 27
MUSCULOSKELETAL STIFFNESS (Musculoskeletal and connective tissue disorders) | 0 | 2
MYALGIA (Musculoskeletal and connective tissue disorders) | 24 | 19
MYOPATHY (Musculoskeletal and connective tissue disorders) | 0 | 1
NECK PAIN (Musculoskeletal and connective tissue disorders) | 8 | 8
NEUROPATHIC ARTHROPATHY (Musculoskeletal and connective tissue disorders) | 0 | 2
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 35 | 31
OSTEOCHONDROSIS (Musculoskeletal and connective tissue disorders) | 1 | 1
OSTEONECROSIS (Musculoskeletal and connective tissue disorders) | 1 | 0
OSTEOPOROSIS (Musculoskeletal and connective tissue disorders) | 0 | 2
OSTEOSCLEROSIS (Musculoskeletal and connective tissue disorders) | 1 | 0
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 22 | 36
PAIN IN JAW (Musculoskeletal and connective tissue disorders) | 5 | 1
PERIARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 | 0
PLANTAR FASCIAL FIBROMATOSIS (Musculoskeletal and connective tissue disorders) | 1 | 0
PLANTAR FASCIITIS (Musculoskeletal and connective tissue disorders) | 0 | 1
POLYMYALGIA RHEUMATICA (Musculoskeletal and connective tissue disorders) | 2 | 2
PSEUDARTHROSIS (Musculoskeletal and connective tissue disorders) | 1 | 0
PSORIATIC ARTHROPATHY (Musculoskeletal and connective tissue disorders) | 1 | 0
RHABDOMYOLYSIS (Musculoskeletal and connective tissue disorders) | 3 | 0
RHEUMATOID ARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 4
ROTATOR CUFF SYNDROME (Musculoskeletal and connective tissue disorders) | 12 | 10
SACROILIITIS (Musculoskeletal and connective tissue disorders) | 0 | 1
SCLERODERMA (Musculoskeletal and connective tissue disorders) | 1 | 0
SENILE ANKYLOSING VERTEBRAL HYPEROSTOSIS (Musculoskeletal and connective tissue disorders) | 0 | 1
SPINAL COLUMN STENOSIS (Musculoskeletal and connective tissue disorders) | 3 | 3
SPINAL DISORDER (Musculoskeletal and connective tissue disorders) | 1 | 1
SPINAL OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 4 | 7
SPONDYLOLISTHESIS (Musculoskeletal and connective tissue disorders) | 2 | 0
SYNOVIAL CYST (Musculoskeletal and connective tissue disorders) | 3 | 1
TENDONITIS (Musculoskeletal and connective tissue disorders) | 1 | 1
TENOSYNOVITIS STENOSANS (Musculoskeletal and connective tissue disorders) | 0 | 1
TRIGGER FINGER (Musculoskeletal and connective tissue disorders) | 2 | 5
VERTEBRAL FORAMINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 0 | 2
ACUTE MYELOID LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
ACUTE PROMYELOCYTIC LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
ADENOCARCINOMA PANCREAS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
B-CELL LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
B-CELL LYMPHOMA STAGE I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
B-CELL LYMPHOMA STAGE IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 8
BENIGN BREAST NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
BENIGN NEOPLASM OF BLADDER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
BENIGN SOFT TISSUE NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
BILE DUCT CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
BLADDER CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 4
BLADDER NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
BOWEN'S DISEASE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 5
BREAST CANCER IN SITU (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
BREAST CANCER STAGE II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
BRONCHIAL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
CHRONIC LYMPHOCYTIC LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
COLON ADENOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 1
COLON CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 5
ENDOMETRIAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
ENDOMETRIAL CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
FIBROMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
GASTROINTESTINAL STROMAL TUMOUR (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
HEPATIC NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
HEPATIC NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
HEPATIC NEOPLASM MALIGNANT RECURRENT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
INTESTINAL ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
LARYNGEAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
LIPOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
LUNG ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
LUNG ADENOCARCINOMA METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
LUNG CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
LUNG CARCINOMA CELL TYPE UNSPECIFIED STAGE IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
LUNG NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 3
LUNG NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 | 4
LUNG SQUAMOUS CELL CARCINOMA STAGE UNSPECIFIED (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
MALIGNANT GLIOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
MALIGNANT MELANOMA IN SITU (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
MALIGNANT PLEURAL EFFUSION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
MANTLE CELL LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
MELANOCYTIC NAEVUS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
MENINGIOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
METASTASES TO CENTRAL NERVOUS SYSTEM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
METASTASES TO LIVER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
METASTATIC MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
METASTATIC NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
METASTATIC RENAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
MUELLER'S MIXED TUMOUR (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
MULTIPLE MYELOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
MYELODYSPLASTIC SYNDROME (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
MYELOFIBROSIS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
NEOPLASM OF APPENDIX (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
NEOPLASM SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
NEUROENDOCRINE CARCINOMA METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
NON-HODGKIN'S LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
NON-SMALL CELL LUNG CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
OESOPHAGEAL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3
OROPHARYNGEAL CANCER STAGE UNSPECIFIED (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
OVARIAN CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
OVARIAN CANCER STAGE III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
OVARIAN NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
PANCREATIC CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
PANCREATIC CARCINOMA METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
PANCREATIC NEUROENDOCRINE TUMOUR (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
PARATHYROID TUMOUR BENIGN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
PERITONEAL CARCINOMA METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
PHAEOCHROMOCYTOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
PITUITARY TUMOUR BENIGN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
PLASMACYTOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
PLEURAL MESOTHELIOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
PLEURAL MESOTHELIOMA MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 | 8
PROSTATE CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
RECTAL ADENOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
RECTAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
RENAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
RENAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
SALIVARY GLAND CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
SALIVARY GLAND NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
SEBORRHOEIC KERATOSIS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
SKIN CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
SMALL CELL LUNG CANCER STAGE UNSPECIFIED (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3
SQUAMOUS CELL CARCINOMA OF SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 4
THYROID CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
THYROID NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3
TRACHEAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
TRANSITIONAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
URETERIC CANCER RECURRENT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
AMNESIA (Nervous system disorders) | 2 | 1
APHASIA (Nervous system disorders) | 1 | 3
BASAL GANGLIA INFARCTION (Nervous system disorders) | 0 | 1
BASILAR ARTERY STENOSIS (Nervous system disorders) | 0 | 1
BRAIN INJURY (Nervous system disorders) | 0 | 1
BRAIN MASS (Nervous system disorders) | 0 | 2
BRAIN STEM INFARCTION (Nervous system disorders) | 1 | 0
CAROTID ARTERIOSCLEROSIS (Nervous system disorders) | 1 | 1
CAROTID ARTERY DISEASE (Nervous system disorders) | 0 | 1
CAROTID ARTERY OCCLUSION (Nervous system disorders) | 1 | 0
CAROTID ARTERY STENOSIS (Nervous system disorders) | 12 | 10
CARPAL TUNNEL SYNDROME (Nervous system disorders) | 8 | 9
CENTRAL NERVOUS SYSTEM LESION (Nervous system disorders) | 1 | 0
CEREBELLAR ATROPHY (Nervous system disorders) | 1 | 0
CEREBELLAR INFARCTION (Nervous system disorders) | 0 | 2
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 2 | 3
CEREBRAL INFARCTION (Nervous system disorders) | 0 | 1
CEREBRAL SMALL VESSEL ISCHAEMIC DISEASE (Nervous system disorders) | 0 | 1
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 15 | 23
CEREBROVASCULAR DISORDER (Nervous system disorders) | 0 | 1
CERVICAL CORD COMPRESSION (Nervous system disorders) | 1 | 0
CERVICAL MYELOPATHY (Nervous system disorders) | 1 | 1
CERVICOBRACHIAL SYNDROME (Nervous system disorders) | 3 | 3
CHRONIC INFLAMMATORY DEMYELINATING POLYRADICULONEUROPATHY (Nervous system disorders) | 1 | 0
COGNITIVE DISORDER (Nervous system disorders) | 0 | 1
COMPLICATED MIGRAINE (Nervous system disorders) | 2 | 1
CONVULSION (Nervous system disorders) | 4 | 2
CRANIAL NERVE DISORDER (Nervous system disorders) | 1 | 0
CUBITAL TUNNEL SYNDROME (Nervous system disorders) | 0 | 1
DEMENTIA (Nervous system disorders) | 2 | 2
DEMENTIA ALZHEIMER'S TYPE (Nervous system disorders) | 2 | 1
DEPRESSED LEVEL OF CONSCIOUSNESS (Nervous system disorders) | 1 | 0
DIABETIC NEUROPATHY (Nervous system disorders) | 1 | 1
DIZZINESS (Nervous system disorders) | 74 | 72
DIZZINESS EXERTIONAL (Nervous system disorders) | 1 | 0
DIZZINESS POSTURAL (Nervous system disorders) | 14 | 6
DRUG WITHDRAWAL HEADACHE (Nervous system disorders) | 1 | 0
DYSARTHRIA (Nervous system disorders) | 1 | 3
DYSGEUSIA (Nervous system disorders) | 1 | 0
EMBOLIC CEREBRAL INFARCTION (Nervous system disorders) | 1 | 0
ENCEPHALOPATHY (Nervous system disorders) | 7 | 2
EPILEPSY (Nervous system disorders) | 0 | 1
ESSENTIAL TREMOR (Nervous system disorders) | 1 | 0
FACIAL PARESIS (Nervous system disorders) | 0 | 1
GRAND MAL CONVULSION (Nervous system disorders) | 2 | 1
GUILLAIN-BARRE SYNDROME (Nervous system disorders) | 0 | 1
HAEMORRHAGE INTRACRANIAL (Nervous system disorders) | 1 | 3
HAEMORRHAGIC STROKE (Nervous system disorders) | 1 | 0
HEAD DISCOMFORT (Nervous system disorders) | 1 | 0
HEAD TITUBATION (Nervous system disorders) | 0 | 1
HEADACHE (Nervous system disorders) | 23 | 28
HEMIPARESIS (Nervous system disorders) | 0 | 1
HYPERTONIA (Nervous system disorders) | 0 | 1
HYPOAESTHESIA (Nervous system disorders) | 27 | 18
IIIRD NERVE PARALYSIS (Nervous system disorders) | 1 | 0
INTERCOSTAL NEURALGIA (Nervous system disorders) | 1 | 0
INTRACRANIAL ANEURYSM (Nervous system disorders) | 0 | 1
INTRAVENTRICULAR HAEMORRHAGE (Nervous system disorders) | 1 | 0
ISCHAEMIC STROKE (Nervous system disorders) | 1 | 3
LACUNAR INFARCTION (Nervous system disorders) | 2 | 0
LETHARGY (Nervous system disorders) | 0 | 2
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 1 | 0
LUMBAR RADICULOPATHY (Nervous system disorders) | 0 | 3
MEMORY IMPAIRMENT (Nervous system disorders) | 0 | 1
METABOLIC ENCEPHALOPATHY (Nervous system disorders) | 6 | 1
MIGRAINE (Nervous system disorders) | 5 | 3
MIGRAINE WITH AURA (Nervous system disorders) | 1 | 1
MONONEURITIS (Nervous system disorders) | 1 | 0
MULTIPLE SCLEROSIS (Nervous system disorders) | 0 | 1
MUSCLE CONTRACTIONS INVOLUNTARY (Nervous system disorders) | 0 | 1
NERVE COMPRESSION (Nervous system disorders) | 2 | 2
NEURALGIA (Nervous system disorders) | 3 | 1
NEURODEGENERATIVE DISORDER (Nervous system disorders) | 1 | 0
NEUROPATHY PERIPHERAL (Nervous system disorders) | 3 | 5
PARAESTHESIA (Nervous system disorders) | 28 | 24
PARKINSON'S DISEASE (Nervous system disorders) | 0 | 2
PARTIAL SEIZURES (Nervous system disorders) | 0 | 1
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 1 | 0
POSTERIOR REVERSIBLE ENCEPHALOPATHY SYNDROME (Nervous system disorders) | 0 | 1
PRESYNCOPE (Nervous system disorders) | 13 | 10
RADIAL NERVE COMPRESSION (Nervous system disorders) | 0 | 1
RADICULOPATHY (Nervous system disorders) | 2 | 0
RESTLESS LEGS SYNDROME (Nervous system disorders) | 2 | 1
SCIATICA (Nervous system disorders) | 7 | 8
SENSORY LOSS (Nervous system disorders) | 0 | 1
SOMNOLENCE (Nervous system disorders) | 2 | 2
SUBARACHNOID HAEMORRHAGE (Nervous system disorders) | 0 | 4
SYNCOPE (Nervous system disorders) | 27 | 36
TENSION HEADACHE (Nervous system disorders) | 0 | 1
TOXIC ENCEPHALOPATHY (Nervous system disorders) | 0 | 1
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 16 | 14
TREMOR (Nervous system disorders) | 2 | 1
TRIGEMINAL NEURALGIA (Nervous system disorders) | 0 | 1
TYPICAL AURA WITHOUT HEADACHE (Nervous system disorders) | 1 | 0
ULNAR TUNNEL SYNDROME (Nervous system disorders) | 0 | 1
UNRESPONSIVE TO STIMULI (Nervous system disorders) | 1 | 0
VERTEBRAL ARTERY STENOSIS (Nervous system disorders) | 1 | 0
VIITH NERVE PARALYSIS (Nervous system disorders) | 2 | 1
ABORTION SPONTANEOUS (Pregnancy, puerperium and perinatal conditions) | 0 | 1
ALCOHOL WITHDRAWAL SYNDROME (Psychiatric disorders) | 1 | 0
ANORGASMIA (Psychiatric disorders) | 0 | 1
ANXIETY (Psychiatric disorders) | 20 | 18
ANXIETY DISORDER DUE TO A GENERAL MEDICAL CONDITION (Psychiatric disorders) | 1 | 0
COMPLETED SUICIDE (Psychiatric disorders) | 1 | 0
CONFUSIONAL STATE (Psychiatric disorders) | 1 | 4
CONVERSION DISORDER (Psychiatric disorders) | 1 | 0
DELIRIUM (Psychiatric disorders) | 3 | 2
DEPRESSION (Psychiatric disorders) | 8 | 12
DEPRESSION SUICIDAL (Psychiatric disorders) | 0 | 2
DISORIENTATION (Psychiatric disorders) | 1 | 0
IMPAIRED SELF-CARE (Psychiatric disorders) | 0 | 1
INSOMNIA (Psychiatric disorders) | 7 | 7
INTENTIONAL SELF-INJURY (Psychiatric disorders) | 0 | 2
MENTAL DISORDER DUE TO A GENERAL MEDICAL CONDITION (Psychiatric disorders) | 1 | 0
MENTAL STATUS CHANGES (Psychiatric disorders) | 7 | 6
PANIC ATTACK (Psychiatric disorders) | 2 | 4
PANIC DISORDER (Psychiatric disorders) | 1 | 0
PERSONALITY DISORDER (Psychiatric disorders) | 1 | 0
POST-TRAUMATIC AMNESTIC DISORDER (Psychiatric disorders) | 0 | 1
PSYCHOGENIC PAIN DISORDER (Psychiatric disorders) | 1 | 0
SLEEP DISORDER (Psychiatric disorders) | 0 | 1
SOMATOFORM DISORDER (Psychiatric disorders) | 0 | 1
STRESS (Psychiatric disorders) | 1 | 2
SUICIDAL IDEATION (Psychiatric disorders) | 1 | 1
SUICIDE ATTEMPT (Psychiatric disorders) | 0 | 1
WITHDRAWAL SYNDROME (Psychiatric disorders) | 0 | 1
AZOTAEMIA (Renal and urinary disorders) | 0 | 1
BLADDER NECK OBSTRUCTION (Renal and urinary disorders) | 1 | 1
BLADDER OBSTRUCTION (Renal and urinary disorders) | 0 | 1
BLADDER PERFORATION (Renal and urinary disorders) | 0 | 1
BLADDER PROLAPSE (Renal and urinary disorders) | 1 | 0
CALCULUS BLADDER (Renal and urinary disorders) | 2 | 0
CALCULUS URETERIC (Renal and urinary disorders) | 1 | 3
CALCULUS URINARY (Renal and urinary disorders) | 1 | 1
CYSTITIS HAEMORRHAGIC (Renal and urinary disorders) | 1 | 0
DYSURIA (Renal and urinary disorders) | 5 | 3
HAEMATURIA (Renal and urinary disorders) | 11 | 18
HYDRONEPHROSIS (Renal and urinary disorders) | 1 | 1
HYPERTONIC BLADDER (Renal and urinary disorders) | 0 | 2
NEPHROLITHIASIS (Renal and urinary disorders) | 14 | 15
NOCTURIA (Renal and urinary disorders) | 2 | 0
OBSTRUCTIVE UROPATHY (Renal and urinary disorders) | 0 | 2
POLLAKIURIA (Renal and urinary disorders) | 2 | 0
POLYURIA (Renal and urinary disorders) | 2 | 0
PROTEINURIA (Renal and urinary disorders) | 0 | 1
RENAL ARTERY STENOSIS (Renal and urinary disorders) | 2 | 4
RENAL COLIC (Renal and urinary disorders) | 1 | 0
RENAL CYST (Renal and urinary disorders) | 3 | 2
RENAL FAILURE (Renal and urinary disorders) | 2 | 3
RENAL FAILURE ACUTE (Renal and urinary disorders) | 32 | 29
RENAL FAILURE CHRONIC (Renal and urinary disorders) | 1 | 5
RENAL HAEMORRHAGE (Renal and urinary disorders) | 0 | 1
RENAL IMPAIRMENT (Renal and urinary disorders) | 2 | 3
RENAL MASS (Renal and urinary disorders) | 3 | 1
RENAL PAIN (Renal and urinary disorders) | 1 | 0
URETERIC STENOSIS (Renal and urinary disorders) | 0 | 1
URETHRAL MEATUS STENOSIS (Renal and urinary disorders) | 0 | 1
URINARY BLADDER POLYP (Renal and urinary disorders) | 0 | 1
URINARY HESITATION (Renal and urinary disorders) | 0 | 1
URINARY INCONTINENCE (Renal and urinary disorders) | 2 | 4
URINARY RETENTION (Renal and urinary disorders) | 3 | 3
URINARY TRACT OBSTRUCTION (Renal and urinary disorders) | 1 | 0
URINE FLOW DECREASED (Renal and urinary disorders) | 1 | 0
ACQUIRED HYDROCELE (Reproductive system and breast disorders) | 2 | 0
ADNEXA UTERI MASS (Reproductive system and breast disorders) | 1 | 0
ATROPHIC VULVOVAGINITIS (Reproductive system and breast disorders) | 0 | 1
BENIGN PROSTATIC HYPERPLASIA (Reproductive system and breast disorders) | 9 | 11
BREAST PAIN (Reproductive system and breast disorders) | 2 | 0
CYSTOCELE (Reproductive system and breast disorders) | 0 | 1
ENDOMETRIAL HYPERPLASIA (Reproductive system and breast disorders) | 1 | 0
EPIDIDYMITIS (Reproductive system and breast disorders) | 2 | 4
ERECTILE DYSFUNCTION (Reproductive system and breast disorders) | 7 | 2
GENITAL PAIN (Reproductive system and breast disorders) | 1 | 0
GENITAL SWELLING (Reproductive system and breast disorders) | 0 | 1
GYNAECOMASTIA (Reproductive system and breast disorders) | 0 | 1
MENORRHAGIA (Reproductive system and breast disorders) | 1 | 1
PELVIC PROLAPSE (Reproductive system and breast disorders) | 1 | 0
PENILE PAIN (Reproductive system and breast disorders) | 0 | 2
PEYRONIE'S DISEASE (Reproductive system and breast disorders) | 0 | 1
PROSTATITIS (Reproductive system and breast disorders) | 0 | 2
PROSTATOMEGALY (Reproductive system and breast disorders) | 1 | 2
SCROTAL CYST (Reproductive system and breast disorders) | 0 | 1
UTERINE OBSTRUCTION (Reproductive system and breast disorders) | 0 | 1
UTERINE POLYP (Reproductive system and breast disorders) | 1 | 0
VAGINAL HAEMATOMA (Reproductive system and breast disorders) | 1 | 0
VAGINAL HAEMORRHAGE (Reproductive system and breast disorders) | 0 | 4
VAGINAL PROLAPSE (Reproductive system and breast disorders) | 1 | 1
VULVAR DYSPLASIA (Reproductive system and breast disorders) | 1 | 0
ACQUIRED DIAPHRAGMATIC EVENTRATION (Respiratory, thoracic and mediastinal disorders) | 1 | 0
ACUTE INTERSTITIAL PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
ACUTE PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 1 | 1
ACUTE RESPIRATORY DISTRESS SYNDROME (Respiratory, thoracic and mediastinal disorders) | 0 | 1
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 15 | 18
ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 1 | 0
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 10 | 4
ATELECTASIS (Respiratory, thoracic and mediastinal disorders) | 3 | 6
BRONCHITIS CHRONIC (Respiratory, thoracic and mediastinal disorders) | 0 | 1
BRONCHOSPASM (Respiratory, thoracic and mediastinal disorders) | 0 | 1
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 27 | 22
CHRONIC RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 | 0
COUGH (Respiratory, thoracic and mediastinal disorders) | 18 | 32
DIAPHRAGMATIC PARALYSIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 159 | 167
DYSPNOEA AT REST (Respiratory, thoracic and mediastinal disorders) | 1 | 0
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 58 | 66
EMPHYSEMA (Respiratory, thoracic and mediastinal disorders) | 4 | 0
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 21 | 16
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 2 | 3
HAEMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 | 1
HICCUPS (Respiratory, thoracic and mediastinal disorders) | 0 | 1
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 2 | 1
INTERSTITIAL LUNG DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 | 0
LUNG DISORDER (Respiratory, thoracic and mediastinal disorders) | 1 | 0
LUNG INFILTRATION (Respiratory, thoracic and mediastinal disorders) | 0 | 1
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 | 1
NASAL SEPTUM DEVIATION (Respiratory, thoracic and mediastinal disorders) | 2 | 0
NASAL TURBINATE HYPERTROPHY (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OBSTRUCTIVE AIRWAYS DISORDER (Respiratory, thoracic and mediastinal disorders) | 1 | 1
OROPHARYNGEAL DISCOMFORT (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 1 | 1
PHARYNGEAL HYPERTROPHY (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PHARYNGEAL MASS (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 7 | 3
PLEURAL FIBROSIS (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PLEURITIC PAIN (Respiratory, thoracic and mediastinal disorders) | 3 | 4
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 3 | 2
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 0 | 2
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 3 | 2
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 1 | 2
PULMONARY CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 | 3
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 10 | 6
PULMONARY FIBROSIS (Respiratory, thoracic and mediastinal disorders) | 2 | 2
PULMONARY HYPERTENSION (Respiratory, thoracic and mediastinal disorders) | 4 | 3
PULMONARY MASS (Respiratory, thoracic and mediastinal disorders) | 1 | 3
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 1 | 5
PULMONARY TOXICITY (Respiratory, thoracic and mediastinal disorders) | 1 | 0
REFLUX LARYNGITIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
RESPIRATORY ALKALOSIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
RESPIRATORY ARREST (Respiratory, thoracic and mediastinal disorders) | 0 | 1
RESPIRATORY DISTRESS (Respiratory, thoracic and mediastinal disorders) | 3 | 1
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 12 | 5
RESTRICTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 | 2
RHINITIS ALLERGIC (Respiratory, thoracic and mediastinal disorders) | 2 | 2
SINUS CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 | 0
SLEEP APNOEA SYNDROME (Respiratory, thoracic and mediastinal disorders) | 6 | 13
THROAT IRRITATION (Respiratory, thoracic and mediastinal disorders) | 2 | 0
THROAT TIGHTNESS (Respiratory, thoracic and mediastinal disorders) | 2 | 0
UPPER RESPIRATORY TRACT CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 | 0
VOCAL CORD POLYP (Respiratory, thoracic and mediastinal disorders) | 0 | 1
WHEEZING (Respiratory, thoracic and mediastinal disorders) | 1 | 2
ACNE (Skin and subcutaneous tissue disorders) | 0 | 1
ACTINIC KERATOSIS (Skin and subcutaneous tissue disorders) | 2 | 1
ALOPECIA (Skin and subcutaneous tissue disorders) | 1 | 0
ANGIOEDEMA (Skin and subcutaneous tissue disorders) | 1 | 2
COLD SWEAT (Skin and subcutaneous tissue disorders) | 1 | 0
DECUBITUS ULCER (Skin and subcutaneous tissue disorders) | 1 | 0
DERMAL CYST (Skin and subcutaneous tissue disorders) | 0 | 1
DERMATITIS (Skin and subcutaneous tissue disorders) | 2 | 2
DERMATITIS CONTACT (Skin and subcutaneous tissue disorders) | 2 | 1
DIGITAL ULCER (Skin and subcutaneous tissue disorders) | 0 | 1
DRUG ERUPTION (Skin and subcutaneous tissue disorders) | 10 | 6
DRY GANGRENE (Skin and subcutaneous tissue disorders) | 0 | 1
ECCHYMOSIS (Skin and subcutaneous tissue disorders) | 1 | 4
ERYTHEMA (Skin and subcutaneous tissue disorders) | 1 | 1
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 21 | 23
INCREASED TENDENCY TO BRUISE (Skin and subcutaneous tissue disorders) | 4 | 6
INGROWING NAIL (Skin and subcutaneous tissue disorders) | 1 | 0
LEUKOCYTOCLASTIC VASCULITIS (Skin and subcutaneous tissue disorders) | 0 | 1
LICHEN SCLEROSUS (Skin and subcutaneous tissue disorders) | 0 | 1
LIVEDO RETICULARIS (Skin and subcutaneous tissue disorders) | 0 | 1
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 3 | 5
PETECHIAE (Skin and subcutaneous tissue disorders) | 1 | 0
PRECANCEROUS SKIN LESION (Skin and subcutaneous tissue disorders) | 1 | 0
PRURITUS (Skin and subcutaneous tissue disorders) | 4 | 2
PRURITUS ALLERGIC (Skin and subcutaneous tissue disorders) | 0 | 2
PSORIASIS (Skin and subcutaneous tissue disorders) | 0 | 1
RASH (Skin and subcutaneous tissue disorders) | 13 | 5
RASH GENERALISED (Skin and subcutaneous tissue disorders) | 0 | 2
RASH MACULAR (Skin and subcutaneous tissue disorders) | 1 | 0
RASH PRURITIC (Skin and subcutaneous tissue disorders) | 4 | 2
SCAR PAIN (Skin and subcutaneous tissue disorders) | 0 | 1
SKIN DISCOLOURATION (Skin and subcutaneous tissue disorders) | 0 | 1
SKIN FISSURES (Skin and subcutaneous tissue disorders) | 0 | 1
SKIN LESION (Skin and subcutaneous tissue disorders) | 2 | 3
SKIN ULCER (Skin and subcutaneous tissue disorders) | 3 | 4
SWELLING FACE (Skin and subcutaneous tissue disorders) | 1 | 1
SYSTEMIC LUPUS ERYTHEMATOSUS RASH (Skin and subcutaneous tissue disorders) | 1 | 0
URTICARIA (Skin and subcutaneous tissue disorders) | 5 | 2
MENOPAUSE (Social circumstances) | 1 | 0
PHYSICAL ASSAULT (Social circumstances) | 0 | 1
TREATMENT NONCOMPLIANCE (Social circumstances) | 0 | 1
ABSCESS DRAINAGE (Surgical and medical procedures) | 0 | 1
AORTIC STENT INSERTION (Surgical and medical procedures) | 1 | 0
BAKER'S CYST EXCISION (Surgical and medical procedures) | 1 | 0
CARDIAC PACEMAKER BATTERY REPLACEMENT (Surgical and medical procedures) | 0 | 2
CATARACT OPERATION (Surgical and medical procedures) | 1 | 0
CORONARY ARTERIAL STENT INSERTION (Surgical and medical procedures) | 1 | 0
FRACTURE REDUCTION (Surgical and medical procedures) | 0 | 1
HERNIA REPAIR (Surgical and medical procedures) | 0 | 1
HIP ARTHROPLASTY (Surgical and medical procedures) | 1 | 1
HYSTERECTOMY (Surgical and medical procedures) | 1 | 0
IMPLANTABLE DEFIBRILLATOR INSERTION (Surgical and medical procedures) | 0 | 1
KNEE ARTHROPLASTY (Surgical and medical procedures) | 0 | 1
NASAL OPERATION (Surgical and medical procedures) | 1 | 0
NECK SURGERY (Surgical and medical procedures) | 0 | 1
PERCUTANEOUS CORONARY INTERVENTION (Surgical and medical procedures) | 1 | 0
ROTATOR CUFF REPAIR (Surgical and medical procedures) | 1 | 1
SURGERY (Surgical and medical procedures) | 0 | 1
ACCELERATED HYPERTENSION (Vascular disorders) | 1 | 1
ANEURYSM (Vascular disorders) | 1 | 1
AORTIC ANEURYSM (Vascular disorders) | 2 | 4
AORTIC DISSECTION (Vascular disorders) | 0 | 1
AORTIC INTRAMURAL HAEMATOMA (Vascular disorders) | 1 | 1
AORTIC STENOSIS (Vascular disorders) | 4 | 4
ARTERIAL DISORDER (Vascular disorders) | 1 | 0
ARTERIAL HAEMORRHAGE (Vascular disorders) | 0 | 1
ARTERIAL OCCLUSIVE DISEASE (Vascular disorders) | 1 | 1
ARTERIAL SPASM (Vascular disorders) | 1 | 2
ARTERIAL THROMBOSIS LIMB (Vascular disorders) | 0 | 1
ARTERIOSCLEROSIS (Vascular disorders) | 2 | 1
ARTERIOVENOUS FISTULA (Vascular disorders) | 1 | 2
DEEP VEIN THROMBOSIS (Vascular disorders) | 7 | 6
EMBOLISM ARTERIAL (Vascular disorders) | 1 | 0
ESSENTIAL HYOERTENSION (Vascular disorders) | 1 | 0
FEMORAL ARTERIAL STENOSIS (Vascular disorders) | 2 | 1
FEMORAL ARTERY ANEURYSM (Vascular disorders) | 1 | 0
FEMORAL ARTERY DISSECTION (Vascular disorders) | 2 | 0
FEMORAL ARTERY OCCLUSION (Vascular disorders) | 2 | 2
HAEMATOMA (Vascular disorders) | 8 | 12
HAEMORRHAGE (Vascular disorders) | 0 | 1
HOT FLUSH (Vascular disorders) | 2 | 1
HYPERTENSION (Vascular disorders) | 55 | 69
HYPERTENSIVE CRISIS (Vascular disorders) | 13 | 11
HYPERTENSIVE EMERGENCY (Vascular disorders) | 2 | 2
HYPOTENSION (Vascular disorders) | 38 | 29
HYPOVOLAEMIC SHOCK (Vascular disorders) | 0 | 1
ILIAC ARTERY OCCLUSION (Vascular disorders) | 0 | 1
ILIAC ARTERY STENOSIS (Vascular disorders) | 0 | 1
INTERMITTENT CLAUDICATION (Vascular disorders) | 10 | 6
INTRA-ABDOMINAL HAEMATOMA (Vascular disorders) | 0 | 1
ISCHAEMIC LIMB PAIN (Vascular disorders) | 0 | 1
LERICHE SYNDROME (Vascular disorders) | 0 | 1
LYMPHOEDEMA (Vascular disorders) | 0 | 1
MACROANGIOPATHY (Vascular disorders) | 0 | 1
MALIGNANT HYPERTENSION (Vascular disorders) | 2 | 0
ORTHOSTATIC HYPOTENSION (Vascular disorders) | 8 | 7
PELVIC VENOUS THROMBOSIS (Vascular disorders) | 1 | 0
PERIPHERAL ARTERIAL OCCLUSIVE DISEASE (Vascular disorders) | 9 | 16
PERIPHERAL COLDNESS (Vascular disorders) | 0 | 1
PERIPHERAL ISCHAEMIA (Vascular disorders) | 0 | 2
PERIPHERAL VASCULAR DISORDER (Vascular disorders) | 5 | 6
REPERFUSION INJURY (Vascular disorders) | 2 | 2
SHOCK (Vascular disorders) | 1 | 0
THROMBOPHLEBITIS (Vascular disorders) | 0 | 2
THROMBOPHLEBITIS SUPERFICIAL (Vascular disorders) | 0 | 3
THROMBOSIS (Vascular disorders) | 2 | 0
VARICOSE VEIN (Vascular disorders) | 2 | 0
VASCULAR STENOSIS (Vascular disorders) | 0 | 1
VASOSPASM (Vascular disorders) | 2 | 1
VENOUS INSUFFICIENCY (Vascular disorders) | 2 | 2
VENOUS RECANALISATION (Vascular disorders) | 1 | 0
VENOUS THROMBOSIS LIMB (Vascular disorders) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2018-08-16): https://cdn.clinicaltrials.gov/large-docs/79/NCT02173379/Prot_003.pdf
  • Statistical Analysis Plan (2018-08-16): https://cdn.clinicaltrials.gov/large-docs/79/NCT02173379/SAP_004.pdf